## VERSION HISTORY

# **Bond Avillion 2 Development LP**

**Clinical Study Protocol** 

Version 3.0, Amendment 2 sion of such application

Of July 2020

Of July 2020 Drug Substance

Study Code

**EudraCT Number** 

Version

Date

A 12-week, Randomized, Double-blind, Placebo-controlled, Multicenter, Parallel Group, Phase III Study Evaluating the Efficacy and Safety of PT027 Compared to PT008 and PT007 Administered QID in Adults and Children 4 Years of Age or Older with Asthma (DENALI)

Sponsor: Bond Avillion 2 Development LP,

Version 3.0, Amendment 2, 06

Global Protocol Amendment

Version 2.0, Amendment 1, 11 February 2019

Global Protocol

7 December 2018 FINAL/APPROVED

This Clinical Study Protocol has been subject to a peer review according to Bond Avillion 2 Development LP Standard procedures. The Clinical Study Protocol is publicly registered and the results are disclosed and/or published according to the Bond Avillion 2 Development LP Global Policy on Bioethics and in compliance with prevailing laws and regulations.

The decorate trade and the based to support out make the last.

## CLINICAL STUDY PROTOCOL SYNOPSIS

PT027 Compared to PT008 and PT007 Administered QID in Adults and Children 4 Years of Age or Older with Asthma (DENALI)



Approximately 100 study sites are anticipated to randomize 1000 adult and adolescent subjects (≥12 years of age) with asthma. Subjects will be randomized 1:1:1:1:1 to 1 of 5 treatment groups. Approximately 200 subjects per group: budesonide/albuterol metered-dose inhaler (BDA MDI) 200 180 µg 4 times daily (QID), BDA MDI 160/180 µg QID, budesonide metered-dose inhaler (BD MDI) 160 μg QID, albuterol sulfate metered-dose inhaler (AS MDI) 180 μg (AD, or placebo MDI. In addition, up to 30 child subjects (aged 4 to 11 years) with asthme will be enrolled but will not receive high dose inhaled corticosteroid (ICS) and will be condomized 1:1:1 to receive low-dose BDA MDI 80/180  $\mu g$  QID, AS MDI 180  $\mu g$ Studential QIDeor placebo MDI. Approximately 2000 subjects will need to be screened, assuming an estimated screen failure rate of 50% prior to randomization. This Phase III study is planned to

This is a 12-week, randomized, double-blind, placebo-controlled, multicenter, parallel group, Phase III study. The purpose of this study is to compare 2 dose levels of BDA MDI compared to its constitute components BD MDI and AS MDI on improvement in lung function and asthma symptoms after 12 weeks of treatment in adults, adolescents, and child subjects, aged 4 years and older, with symptomatic asthma currently being treated with short/rapid-acting β2-

Subjects meeting all entry criteria at the screening visit (Visit 1) will enter a 14 to 28-day screening (run-in) period. Only Sponsor-provided investigational product (IP) and Sponsor provided Ventolin to be used in response to asthma symptoms are allowed during the study.

No other asthma medications are allowed during the study.

No other asthma medications are allowed during the study.

During the screening (run-in) period, subjects will self-administer single-blind placebo MDI OID and Ventalin are forced. QID and Ventolin prn for asthma symptoms only. Subjects will be trained and instructed in the use of an electronic diary (eDiary) and peak flow meter at Visit 1 to record protocol required data into the eDiary twice daily. Eligible subjects will be randomized at Visit 2. or ari

## **Objectives**

| Primary objective: Primary endpoint: | |
|---|---|
| To demonstrate the contribution of budesonide and albuterol in BDA MDI 80/180 μg and 160/180 μg administered QID by comparing with mono-components (BD MDI 160 μg, AS MDI 180 μg) and placebo on lung function | Dual Strimator endpoints: Change from baseline in FEV <sub>1</sub> AUC <sub>0-6 hours</sub> over 12 weeks Change from baseline in trough FEV <sub>1</sub> at Week 12 |
| Secondary objective: | Secondary endpoint: |
| To characterize the effect of BDA MDI 804180 µg and 160/180 µg administered QID or bronchodilation and asthma symptoms compared to the mono-components (BD MDI 160 µg, AS MDI 180 µg) and placebo | <ul> <li>The time to onset (defined as 15% increase in FEV₁ over the pre-treatment value on Day 1), and duration of response on Day 1</li> <li>Number (%) of subjects who have an Asthma Control Questionnaire-7 (ACQ-7) score of ≥1.5 at baseline who achieve a clinically meaningful improvement (a decrease of at least 0.5 units from baseline) in ACQ-7 at Week 12</li> <li>Trough FEV₁ at Week 1</li> </ul> |
| Safety objective: | Safety endpoints: |
| To caluate the safety and tolerability of BDA MDI 80/180 μg and 160/180 μg administered QID compared to BD MDI (160 μg) and AS MDI (180 μg) | <ul> <li>AE/SAEs</li> <li>Vital signs (ie, heart rate, blood pressure only)</li> <li>Clinical chemistry and hematology parameters</li> <li>Electrocardiogram (ECG)</li> </ul> |

| Exploratory objective: | Exploratory endpoints: |
|---|---|
| To characterize the effect of BDA MDI 80/180 µg and 160/180 µg administered QID on bronchodilation and asthma symptoms compared to the mono-components (BD MDI 160 µg, AS MDI 180 µg) and placebo | <ul> <li>Deteriorations of asthma</li> <li>Incidence of severe exacerbations</li> <li>Change from baseline in: <ul> <li>Trough FEV<sub>1</sub> at individual time points</li> <li>FEV<sub>1</sub> AUC<sub>0-6</sub> hours at individual time points</li> <li>Peak change from baseline FEV<sub>1</sub> at Day 1 and Day 7</li> <li>Morning and evening peak expiratory flow (PEF)</li> <li>Use of Ventolin therapy in response to asthma symptoms</li> <li>Asthma daytime/night-time symptoms</li> <li>Asthma Control Questionaire-5 (ACQ-5) and responder analysis at Week 12</li> <li>Asthma Quality of Life Questionnaire +12 for 12 years and older (AQLQ+12)/Pediatric Asthma Quality of Life Questionnaire (PAQLQ) change from baseline at Week 12</li> </ul> </li> </ul> |

Target Subject Population

Male and female subjects ≥4 years of age where approved, ≥18 years of age for all other countries, with a diagnosis of asthma (GINA) criteria with pre-bronchodilator FEV of ≥50 to <85% predicted normal value (subjects ≥18 years of age) and ≥50% predicted normal value for subjects 4 to 17 years of age, where approved, with demonstrate in-clinic FEV1 reversibility to Sponsor-provided SABA will be included.

Subjects must be taking a stable dosing of asthma therapies (only prn SABA or stable low-dose ICS in addition to prn SABA) for at least the last 30 days prior to Visit 1 may be eligible for this study.

• A screening/run-:• A 12

- A screening/run-in period (14 to 28 days).

A safety follow-up period: where a safety follow-up telephone contact (TC) will occur 2 weeks (±4 days) after the subject's last dose of treatment (end-of-treatment [EOT]) or premature discontinuation visit (PDV).

Investigational Product, Dosage, and Mode of Administration

BDA MDI is formulated as both micronized budesonide and micronized albuteroff co-suspended with spray-dried porous particles in a hydrofluoroalkane propertient co-suspension formulation ensures that subjects receive a consistent deliverable actuation of the MDI.

Only Sponsor-provided IP adminimized budesonide in response deliverable and micronized albuteroff co-suspension formulation ensures that subjects receive a consistent deliverable actuation of the MDI.

medications are allowed during the study.

At randomization (Visit 2), adult (≥18 years of age) and adolescent subjects (aged 12 - 17 years, where approved) who meet the eligibility criteria will be randomly assigned to 1 of the following 5 treatment groups in a 1:1:1:1:1 ratio:

- BDA MDI 80/180 μg QID (given \$2 actuations of BDA MDI 40/90 μg per puff)
- BDA MDI 160/180 μg QID (given as 2 actuations of BDA MDI 80/90 μg per puff)
- BD MDI 160 μg QID (given as 2 actuations of BD MDI 80 μg per puff)
- AS MDI 180 µg QID (given as 2 actuations of AS MDI 90 µg per puff)
- Placebo MDI QID (given as 2 actuations)

The maximum daily dosage of IP should not exceed 12 puffs per day.

Subjects All be recommended not to take more than 8 puffs of Ventolin per day and advised to contact the investigator if their symptoms necessitate more than 8 puffs of Ventolin in a

## **Statistical Methods**

## **Sample Size Calculation**

A preliminary sample size calculation was based on historical trial data. A sample size of 600 subjects was initially proposed to provide 93% power to detect a difference in change

from baseline in trough FEV<sub>1</sub> at week 12 of 100 mL for comparisons of BD MDI versus placebo MDI, BDA MDI versus placebo MDI, or BDA MDI versus AS MDI. This calculation was based on a standard deviation of 210 mL obtained from the placebo MDI group of Study

because the assumed variability from the lung function data has a large impact on the estimated sample size necessary to achieve a stated power, a blinded estimate of the variability of pre-dose trough FEV<sub>1</sub> at Week 12 was calculated. The review was performed once 440× subjects had completed Week 12, and prior to the 600<sup>th</sup> subject had completed Week 12, and prior to the 600<sup>th</sup> subject had completed Week 12.

Decisions following the blinded sample size re-estimation

The blinded sample size re-estimation was performed once 44% of subjects had completed Week 12. Based on the blinded estimate of variability, approximately 1000 subjects are required in order to demonstrate 90% power. Consequently, the total number of randomized adult and adolescent subjects has been increased by 400 to 1,000.

Randomization of approximately 200 subjects to each treatment group will provide 90% probability to detect a 100 mL difference in the change from baseline in trough FEV<sub>1</sub> at Week 12 for comparison of BD MDI versus placebo MDO BDA MDI versus placebo MDI, or BDA MDI versus AS MDI. This calculation is based on a standard deviation of 290 mL obtained from the blinded sample size re-estimation performed after 44% of subjects completed week 12 and an estimated overall dropout rate of 11% prior to Week 12.

The sample size of 200 subjects per treatment group will also provide >99% probability to detect a 130 mL difference in FEV<sub>1</sub> AUC<sub>0-6 hours</sub> over 12 weeks for comparison of BDA MDI versus BD MDI (effect sizes for AS MDI or BDA MDI versus placebo MDI should be considerably larger). This calculation assumes 2% dropout prior to Week 1 and an effective standard deviation of 300 mL obtained from the blinded sample size re-estimation performed after 44% of subjects completed Week 12.

Approximately 1000 adults (≥18 years of age) and adolescent subjects (12 - 17 years of age, where approved) with asthma will be randomized 1:1:1:1:1 to 1 of 5 treatment groups (approximately 200 subjects per group: BDA MDI 80/180 μg QID, BDA MDI 160/180 μg QEO, BD MDI 160 µg QID, AS MDI 180 µg QID, or placebo MDI). In addition, where approved, up to 30 child subjects (aged 4 to 11 years) with asthma will be enrolled but will not receive high dose ICS and will be randomized 1:1:1 to receive low-dose BDA MDI 80/180 μg QID, AS MDI 180 µg QID, or placebo MDI. Approximately 2000 subjects will need to be screened, assuming an estimated screen failure rate of approximately 50% prior to randomization. This Phase III study is planned to be conducted globally.

A second blinded sample size re-estimation will be performed once approximately 65% of the revised sample has completed 12 weeks and prior to the last subject being randomized. This will allow the re-assessment of variability in a larger sample and at a point where any impact

The potential increase in sample size will be capped at 1300, a 30% increase above the revised number of 1000 subjects.

Primary Efficacy Analysis

The first and second dual-primary variables, change from baseline in FEV<sub>1</sub> At C<sub>0-6</sub> hours, and change from baseline in trough FEV<sub>1</sub> will each be analyzed using a repeated measures (RM) linear model to compare treatment groups. The model will include back to Ventolin, and age as continuous by-visit interaction and by-visit interaction, and prior ICS use (Yes/No) as categorical covariates. Baseline will be defined as the average of the pre-dose assessments collected on randomization (Visit 2).

An unstructured variance-covariance matrix will a implemented. If this model fails to converge, a heterogeneous Toeplitz (TOEPH) will be fit.

## **Secondary Efficacy Analyses**

The median time to onset (defined as 15% increase in FEV<sub>1</sub>) over the pre-treatment value at randomization (Visit 2) will be compared among treatment groups using a Wilcoxon rank sum test. Confidence intervals for the median treatment difference will be calculated using the Hodges-Lehmann method. Descriptive statistics for duration of response will be reported by treatment group. Only the subjects who achieve the 15% increase in FEV<sub>1</sub> within 30 minutes post-dose will be included in these calculations.

The treatment effect for change from baseline in ACQ-7 will be estimated using a mixed model RM (NEMRM) analysis. All data up to Week 12 will be included in the model, with terms for age, treatment, visit, treatment\* visit, prior ICS use (Yes/No), baseline ACQ-7 score and baseline post-dose percent predicted FEV<sub>1</sub>. Visit will be fitted as a categorical variable, and the variance-covariance matrix will be assumed to be unstructured. If the procedure does not converge, then a heterogeneous Toeplitz (TOEPH) will be used instead. This model will be used to give an overall assessment of the treatment effect as well as 95% confidence intervals.

## **Estimands**

The primary estimand of interest is the efficacy estimand, defined as the effect of the The second estimand of interest is the attributable estimand, defined as the effect of treatment in subjects attributable to the randomized treatment. For this estimand, discontinuation randomized treatment for reasons such as tolerability or lack of efficience negative outcome. This estimand is a mixture of defined in the draft ICH EO

. disco.
. icacy is coi
. hypothetical st,
hypothetical st,
of any painting

of any painting

of any painting

this document must not be used to support any marketing att.

This document must not be used to support any marketing att.


# **TABLE OF CONTENTS**

| TITLE PA | GE | 1 |
|---|---|---|
| VERSION | HISTORY | 1 |
| CLINICAI | L STUDY PROTOCOL SYNOPSIS | 3 |
| TABLE O | F CONTENTS | 10 |
| LIST OF A | ABBREVIATIONS AND DEFINITION OF TERMS | 16\$\ |
| 1 | INTRODUCTION Background Rationale for study design, doses, and control groups Benefit/risk and ethical assessment Study design Study governance and oversight Independent data monitoring committee STUDY OBJECTIVES Primary objectives Secondary objectives Exploratory objectives EXPLICATION ENDOLLMENT DANDOMIZATION | :018 |
| 1.1 | Background | .el18 |
| 1.2 | Rationale for study design, doses, and control groups. | 19 |
| 1.3 | Benefit/risk and ethical assessment. | 20 |
| 1.4 | Study design | 21 |
| 1.5 | Study governance and oversight | 23 |
| 1.5.1 | Independent data monitoring committee | 23 |
| 2 | STUDY OBJECTIVES | 24 |
| 2.1 | Primary objectives | 24 |
| 2.2 | Secondary objectives | 24 |
| 2.3 | Safety objectives | 24 |
| 2.4 | Exploratory objectives | 25 |
| 3 | RESTRICTIONS TREATMENTODISCONTINUATION AND STUDY | |
| 3.1 | TERMINATION Inclusion criteria Exclusion criteria | 25 |
| 3.2 | Exclusion criteria | 27 |
| 3.3 | Subject enrollment and randomization | 30 |
| 3.4 | Procedures for bandling incorrectly enrolled or randomized subjects | 30 |
| 3.5 | Methods for ssigning treatment groups | |
| 3.6 | Methods for ensuring blinding | 31 |
| 3.7 | Methods for unblinding | 31 |
| 3.8 | Restrictions | 32 |
| 3.9 | Treatment discontinuation by subject and/or Sponsor | 33 |
| 3.10 Jist . | Study termination | 33 |
| 3. N. | Screen failures | 34 |
| \$ <sup>0</sup> , | Methods for ensuring blinding Methods for unblinding Restrictions Treatment discontinuation by subject and/or Sponsor Study termination Screen failures STUDY PLAN AND TIMING OF PROCEDURES | 35 |
| 4.1 | Screening and enrollment period | |
| 4.2 | Randomization/treatment period | 42 |
| 4.3 | Treatment discontinuation visit | 43 |
| 4.4 | Unscheduled visit | 44 |

| 4.5 | Safety Follow-up period4 | |
|---|---|---|
| 5 | STUDY ASSESSMENTS | 44 |
| 5.1 | Efficacy assessments | 44 |
| 5.1.1 | Lung function measurement by spirometry | |
| 5.1.1.1 | Reversibility test | |
| 5.1.1.2 | COVID-19 and Pulmonary Function Testing | |
| 5.1.2 | Asthma Control Questionnaire-5 | |
| 5.1.3 | Asthma Control Questionnaire-7 | 48% |
| 5.1.4 | Asthma Control Questionnaire-Interviewer-Administered | 480 |
| 5.1.5 | Asthma Control Questionnaire-Interviewer-Administered | fe si <sup>ON</sup> |
| | Questionnaire | .e48 |
| 5.1.5.1 | Asthma Quality of Life Questionnaire+12 | 48 |
| 5.1.5.2 | Pediatric Asthma Quality of Life Questionnaire | 48 |
| 5.1.6 | eDiary | 49 |
| 5.1.6.1 | Peak expiratory flow | 49 |
| 5.1.6.2 | Asthma Quality of Life Questionnaire+12/Pediatric Asthma Quality of Life Questionnaire Asthma Quality of Life Questionnaire+12 Pediatric Asthma Quality of Life Questionnaire eDiary Peak expiratory flow eDiary investigational product use eDiary Ventolin therapy use eDiary recording of symptoms and alerts Deterioration of asthma | 49 |
| 5.1.6.3 | eDiary Ventolin therapy use | 49 |
| 5.1.6.4 | eDiary recording of symptoms and alerts | 49 |
| 5.1.7 | Deterioration of asthma | 50 |
| 5.1.8 | Definition of asthma symptom worsening Signature Signatu | 51 |
| 5.1.8.1 | Definition of asthma symptom worsening | 51 |
| 5.1.8.2 | Investigator justified asthma exacerbations Severe asthma exacerbations | 51 |
| 5.1.8.3 | | |
| 5.1.8.4 | Treatment for severe asthma exacerbations | 52 |
| 5.1.8.5 | Onset and duration of asthma exacerbations | 52 |
| 5.1.8.6 | Approach for capturing asthma exacerbations | 53 |
| 5.2 | Safety assessments | 53 |
| 5.2.1 | Laboratory safety assessments | 53 |
| 5.2.2 | Resting 12-lead electrocardiogram | 54 |
| 5.2.3 | Vital sign measurements | 55 |
| 5.2.4 | Adverse event assessments | |
| 5.3 | Other assessments | 55 |
| 5.3.1 | Physical examination | 55 |
| 5.3.2 | Concooltant medications | 55 |
| 5.4 | Phaonacokinetics | 56 |
| 5.5 | Pharmacodynamics | 56 |
| 5.6 | Genetics | 56 |
| 5.7 MUS | Biomarker analysis | 56 |
| ent | Other assessments Physical examination Concopitant medications Pharmacokinetics Pharmacodynamics Genetics Biomarker analysis SAFETY REPORTING AND MEDICAL MANAGEMENT Definition of adverse events | 56 |
| 6.1 | Definition of adverse events | 56 |
| 6.2 | Definitions of serious adverse event | 56 |
| 6.3 | Recording of adverse events | 57 |
| 6.3.1 | Period for collection of adverse events | |

| 6.3.2 | Follow-up of unresolved adverse events | 57 |
|---|---|---|
| 6.3.3 | Variables | 57 |
| 6.3.4 | Causality collection | 58 |
| 6.3.5 | Adverse events based on signs and symptoms | 58 |
| 6.3.6 | Adverse events based on examinations and tests | |
| 6.3.7 | Hy's Law | 59 |
| 6.3.8 | COVID-19 adverse events | 59 |
| 6.4 | Reporting of serious adverse events | 60, |
| 6.5 | Overdose | 6O |
| 6.6 | Pregnancy | <b>.</b> 61 |
| 6.6.1 | Maternal exposure | 61 |
| 6.6.2 | Paternal exposure | 62 |
| 6.7 | Medication error | 62 |
| 6.8 | Overdose Pregnancy Maternal exposure Paternal exposure Medication error Management of investigational product–related toxicities INVESTIGATIONAL PRODUCT AND OTHER TREATMENTS | 63 |
| 7 | INVESTIGATIONAL PRODUCT AND OTHER TREATMENTS | 63 |
| 7.1 | Identity of investigational product(s) Dose and treatment regimens Labelling Storage Compliance Accountability | 63 |
| 7.2 | Dose and treatment regimens | 64 |
| 7.3 | Labelling | 65 |
| 7.4 | Storage | 66 |
| 7.5 | Compliance | 66 |
| 7.6 | Accountability | 66 |
| 7.7 | Metered-dose inhaler: handling and cleaning | 67 |
| 7.8 | Concomitant medications and other treatments | 67 |
| 7.8.1 | Investigational product and Ventolin therapies | 67 |
| 7.8.2 | Medications that may affective versibility and FEV <sub>1</sub> testing | 67 |
| 7.8.3 | Prohibited medications | 67 |
| 8 | STATISTICAL ANALYSES | 68 |
| 8.1 | Statistical considerations | 68 |
| 8.1.1 | Estimands Sample size estimate | 68 |
| 8.2 | Sample size estimate | 68 |
| 8.2.1 | Initial assumptions and estimates | 68 |
| 8.2.2 | Blinged sample size re-estimation | 69 |
| 8.3 | Definitions of analysis sets | 70 |
| 8.3.1 | Full analysis set | 70 |
| 8.3.2 | Safety analysis set | 70 |
| 8.4. | Initial assumptions and estimates Blinged sample size re-estimation Definitions of analysis sets Full analysis set Safety analysis set Violations and deviations Outcome measures for analyses | 70 |
| 84.5 | Outcome measures for analyses | 71 |
| 8.5.1 | Primary efficacy analysis | / I |
| 8.5.1.1 | Dual-primary efficacy endpoints | |
| 8.5.2 | Secondary efficacy analyses | |
| 8.5.2.1 | Derivation for time to onset (15% increase in FEV <sub>1</sub> ) on Day 1 and duration of | |
| | effect on Day 1 | 71 |

| 8.5.2.2 | Derivation of Asthma Control Questionnaire-7 variables | |
|---|---|---|
| 8.5.3 | Exploratory efficacy analyses | |
| 8.5.3.1 | Derivation of severe exacerbation endpoints | 72 |
| 8.5.3.2 | Derivation of deterioration of asthma variables | 73 |
| 8.5.3.3 | Derivation of peak FEV <sub>1</sub> | 73 |
| 8.5.3.4 | Derivation of peak expiratory flow | 73 |
| 8.5.3.5 | Derivation of Asthma Control Questionnaire-5 variables | |
| 8.5.3.6 | Derivation of Asthma Quality of Life Questionnaire +12 and Pediatric Astl | |
| 8.5.3.7 | Derivation of Ventolin therapy variables | <i>\$</i> 74 |
| 8.5.3.8 | Derivation of other eDiary variables | |
| 8.6 | Quality of Life Questionnaire variables Derivation of Ventolin therapy variables Derivation of other eDiary variables Methods for statistical analyses Analysis of the dual-primary variable Analysis of the secondary efficacy variables Median time to onset (15% increase in FEV <sub>1</sub> ) and duration of effect Asthma Control Questionnaire-7 Analysis of safety variables Adverse events Vital signs Clinical chemistry and hematology Electrocardiogram Concomitant medication Analysis of exploratory variables | وم<br>74 |
| 8.6.1 | Analysis of the dual-primary variable | 74 |
| 8.6.2 | Analysis of the secondary efficacy variables | 76 |
| 8.6.2.1 | Median time to onset (15% increase in FEV <sub>1</sub> ) and duration of effect | 76 |
| 8.6.2.2 | Asthma Control Ouestionnaire-7 | 76 |
| 8.6.3 | Analysis of safety variables | 77 |
| 8.6.3.1 | Adverse events | 77 |
| 8.6.3.2 | Vital signs | 77 |
| 8.6.3.3 | Clinical chemistry and hematology | 77 |
| 8.6.3.4 | Electrocardiogram | 77 |
| 8.6.3.5 | Concomitant medication. | 78 |
| 8.6.4 | Analysis of exploratory variables | 78 |
| 8.6.4.1 | Severe exacerbations | /8 |
| 8.6.4.2 | Deterioration of asthma | 78 |
| 8.6.4.3 | Deterioration of asthma. Peak FEV1 Peak expiratory flow | 78 |
| 8.6.4.4 | Peak expiratory flow | 78 |
| 8.6.4.5 | Asthma Control Questionnare-5 variables | 78 |
| 8.6.4.6 | Asthma Quality of Life Questionnaire +12 and Pediatric Asthma Quality of Questionnaire | f Life |
| | Questionnaire | 79 |
| 8.6.4.7 | Ventolin therapy, 2 | 79 |
| 8.6.4.8 | Other eDiary variables | 79 |
| 8.6.5 | Subgroup analysis | 80 |
| 8.6.6 | Interim analysis | 80 |
| 8.6.7 | Sensitivity analysis | 80 |
| 8.6.7.1 | Tipping point analysis | 80 |
| 8.6.7.2 | Addributable estimand | 80 |
| 8.6.7.3 | CCOVID-19 pandemic impacts | 81 |
| 9 Milest | Interim analysis Sensitivity analysis Tipping point analysis Anributable estimand COVID-19 pandemic impacts STUDY AND DATA MANAGEMENT Training of study site staff Monitoring of the study | 81 |
| 9.1 | Training of study site staff | 81 |
| 9.2 | Monitoring of the study | 81 |
| 9.2.1 | Source data | 82 |
| 9.2.2 | Study agreements | 82 |
| 9.2.3 | Archiving of study documents | 82 |
| 9.3 | Study timetable and end-of-study | 83 |

| 9.4 | Data management | 83 |
|---|---|---|
| 10 | ETHICAL AND REGULATORY REQUIREMENTS | 84 |
| 10.1 | Ethical conduct of the study | 84 |
| 10.2 | Subject data protection | 84 |
| 10.3 | Ethics and regulatory review | 84 |
| 10.4 | Informed consent/assent | 85 |
| 10.5 | Changes to the clinical study protocol and informed consent/assent form | 85 ج |
| 10.6 | Audits and inspections | 86 |
| 11 | SUMMARY OF CHANGES | 86 |
| 11.1 | Changes to protocol amendment 2 (Version 3.0) | 86 |
| 11.2 | Changes to protocol amendment 1 (Version 2.0) | 93 |
| 12 | LIST OF REFERENCES | 95 |
| APPEND | Changes to the clinical study protocol and informed consent/assent form | 97 |
| APPEND | DIX B, PRIMARY INVESTIGATOR SIGNATURE PAGE | 98 |
| APPEND | DIX C, GLOBAL INITIATIVE FOR ASTHMA (GINA) 2018) | 99 |
| APPEND | DIX D, ADDITIONAL SAFETY INFORMATION (CO.) | 101 |
| APPEND | DIX E, HY'S LAW | 103 |
| APPEND | DIX F, ASTHMA QUALITY OF LIFE 12 QUESTIONNAIRE | 108 |
| | DIX G, PEDIATRIC ASTHMA QUALITY OF LIFE QUESTIONNAIRE | |
| APPEND | DIX H, ASTHMA CONTROISOUESTIONNAIRE | 119 |
| APPEND | OIX I, ASTHMA CONTROL GOESTIONNAIRE-INTERVIEWER-<br>ADMINISTERED | |
| APPEND | DIX J, METERED-DOSE INHALER HANDLING AND CLEANING | |
| APPEND | DIX K, SPIROMET&Y ASSESSMENT CRITERIA | 138 |
| | DIX L, COVID SEMERGENCY MEASURES PERMITTED TO ENSURE SUBJECT SAFETY | 140 |
| LIST O | Study assessments and procedures Timed assessments at Visit 2 through Visit 6 and Premature Discontinuation Visit | |
| Table | Study assessments and procedures | 37 |
| Table 2 | Timed assessments at Visit 2 through Visit 6 and Premature | |
| Up | Discontinuation Visit | 40 |
| Table 3 | Schedule of FEV <sub>1</sub> measurements at standard visits | 46 |
| Table 4 | Laboratory Safety Variables | 54 |
| Table 5 | Investigational Product Strength and Dosage Form | 64 |

The dather rust rate leads to append on the rest of the state of the s


# LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

The following abbreviations and special terms are used in this Clinical Study Protocol.

| Abbreviation or special term | Explanation |
|---|---|
| ACQ-5 | Asthma Control Questionnaire-5 |
| ACQ-7 | Asthma Control Questionnaire-7 |
| ACQ-IA | Asthma Control Questionnaire-Interviewer-Administered |
| AE | Asthma Control Questionnaire-5 Asthma Control Questionnaire-Interviewer-Administered adverse event allergy immunotherapy alanine aminotransferase Asthma Quality of Life Questionnaire for 12 years and older albuterol sulfate metered-dose inhaler aspartate aminotransferase American Thoracic Society/European Respiratory Society area under the concentration curve from Quot 6 hours |
| AIT | allergy immunotherapy |
| ALT | alanine aminotransferase |
| AQLQ+12 | Asthma Quality of Life Questionnaire for 12 years and older |
| AS MDI (PT007) | albuterol sulfate metered-dose inhaler |
| AST | aspartate aminotransferase |
| ATS/ERS | American Thoracic Society/European Respiratory Society |
| AUC <sub>0-6 hours</sub> | area under the concentration curve from 0 6 hours |
| BD MDI (PT008) | budesonide metered-dose inhales |
| BDA MDI (PT027) | budesonide/albuterol meterod-dose inhaler |
| β-hCG | β-human chorionic gonadotropin |
| BMI | body mass index |
| CFC | chlorofluorocaroon propellant |
| EC | Ethics Committee synonymous to Institutional Review Board (IRB) and Independent thics Committee (IEC) |
| ECG | electrocardiogram |
| eCRF | electionic case report form |
| eDiary | ectronic diary |
| EOT S | end-of-treatment |
| ePRO ed | electronic patient reported outcome |
| FEV <sub>1</sub> | forced expiratory volume in 1 second |
| FVC X | forced vital capacity |
| GCP AT | Good Clinical Practice |
| eCRF eDiary EOT ePRO FEV1 FVC GCP GRA GMP HL | Global Initiative for Asthma |
| <b>C</b> GMP | Good Manufacturing Practice |
| HL | Hy's Law |
| ICF | informed consent form |
| ICH | International Conference on Harmonization |
| ICS | inhaled corticosteroid |

| | Abbreviation or special term | Explanation |
|---|---|---|
| | IDMC | Independent Data Monitoring Committee |
| | International Coordinating investigator | If a study is conducted in several countries, the International Coordinating investigator is the investigator coordinating the investigators and/or activities internationally. |
| | IP | investigational product |
| | IWRS | Interactive Web Response System |
| | LABA | long-acting β2-agonist |
| | MDI | metered-dose inhaler |
| | MID | minimal important difference |
| | MMRM | mixed model repeated measures |
| | PAQLQ | Pediatric Asthma Quality of Life Questionnaire |
| | PDV | premature discontinuation visit |
| | PEF | peak expiratory flow |
| | PFT | Interactive Web Response System long-acting β2-agonist metered-dose inhaler minimal important difference mixed model repeated measures Pediatric Asthma Quality of Life Questionnaire premature discontinuation visit peak expiratory flow pulmonary function test |
| | PHL | potential Hy's Law |
| | prn | pulmonary function test potential Hy's Law as needed OF OF |
| | QID | four times daily |
| | RM | repeated measures |
| | SABA | short/rapid-acting β2-adrenoreceptor agonist |
| | SAE | serious adverse events |
| | SAP | Statistical Analysis Plan |
| | SCS | |
| | SMART | budeson de/formoterol (Symbicort); approved for maintenance and reliever therapy |
| | TBL | Sotal bilirubin |
| | TC 5 | telephone contact |
| | ULN ed | upper limit of normal |
| | WBDC VS | Web Based Data Capture |
| This docut | SCS SMART TBL TC ULN WBDC WBDC TENTIFICATION TO SERVICE OF SERVI | |

#### INTRODUCTION 1

#### 1.1 **Background**

metered-dose inhaler [BDA MDI]) pressurized inhalation suspension in adults and children 4 years of age or older with asthma. Please refer to the current Investigator Brochure for additional of information.

Albuterol is a short/rapid-acting β2-adrenoreceptor agonist (SABA), inducing airway smooth muscle relaxation and reducing or preventing bronchoconstriction.

clinical practice, albuterol is used as an as needed (prn) reliever therapy (Global Initiative for Asthma [GINA] 2018). Albuterol is approved in many countries as salbutation in multiple formulations for the treatment or prevention of bronchoconstriction.

Budesonide is a well-established anti-inflammatory corticosteroid that exhibits potent glucocorticoid and weak mineralocorticoid activity and is approved worldwide in orally inhaled formulations for the treatment of asthma and chronic obstructive pulmonary disease both as a mono-product and in combination with a long/rapid-acting \beta2-agonist (LABA, formoterol).

In vitro studies have demonstrated that inhaled corticosteroid (ICS) agents potentiate the effects of SABAs in reducing airway smooth muscle tone (Mendes 2008) and can reverse adrenergic receptor tolerance and desensitization (Cooper and Panettieri 2008). Clinically, similar functional potentiation with combined ICSs and allower old has been observed in patients with asthma for functional measures of airway smooth muscle and airway blood flow (Mendes 2015). An analysis of 425 asthma exacerbations in patients from the Formoterol and Corticosteroids Establishing Therapy International Study Group study (Tattersfield 1999) revealed that asthma symptoms use were noted. Wer several days before the start of an asthma exacerbation; increased reliever therapy (ie, albuterol) followed a similar pattern, providing rapid bronchodilation to treat the symptoms. Combining albuterol with budesonide in the proposed BDA MDI combination product should not only provide rapid bronchodilation, but also treat worsening airway inflammation by the addition of the budesonide component. Per current treatment guidelines (GINA 2008), ICS/formoterol maintenance and reliever can be used in patients with asthma. Studies of budesonide and a rapid-acting LABA (formoterol) as reliever therapy have demonstrated enhanced protection from severe exacerbations in patients already receiving Ombination therapy for maintenance without an increase in adverse effects (Rabe 2006; O'Byrne 2005). In addition, budesonide/formoterol as maintenance and reliever therapy or 'SMART' (available commercially as the Symbicort Turbuhaler [Symbicort] in the European Union and other markets) significantly reduced severe exacerbation risk in pediatric patients (O'Byrne 2007).

With SMART application, patients with asthma use Symbicort as maintenance inhalation medication and also prn in response to symptoms. The simultaneous administration of budesonide with formoterol when symptoms occur ensures that patients with asthma receive both a rapid-acting bronchodilator for symptom relief and anti-inflammatory medication to treat their persistent airway inflammation. BDA MDI would have added effect on improvement of lung function and achieving asthma improvement beyond what is seen with albuterol and budesonide alone. Current treatment guidelines (GINA 2018) recommend considering addition of low-dose ICS to SABA used as reliever medication as early as in GINA step 1 asthma (previously treated with SABA prn alone), broadening the range of asthma severity grades that would be treated by both ICS and β2-adrenoreceptor agonist. Anti-inflammatory and bronchodilation component in combination is expected to result with superior control and decreased risk of experiencing asthma symptoms.

# 1.2 Rationale for study design, doses, and control groups

This is a 12-week, randomized, double-blind, placebo-controlled, multicenter, parallel group, Phase III study in adults, adolescents, and child subjects, aged 4 years and older, with symptomatic asthma currently being treated with SABA prn alone or with low-dose ICS maintenance therapy plus SABA prn.

This 12-week Phase III study is a pivotal efficacy and safety study for approval of BDA MDI fixed dose combination product. This study is designed to investigate the benefit of 2 dose levels of BDA MDI compared to its constituent components budesonide metered-dose inhaler (BD MDI [PT008]) and albuterol sulfate metered-dose inhaler (AS MDI [PT007]) based on improvement in lung function and asthmat symptoms after 12 weeks of treatment. This study will demonstrate the combination rule regarded by the Food and Drug Administration according to the 21 Code of Federal Regulation 300.50.

Two dosage levels, of BDA MDI administered 4 times daily (QID), 80/180 µg (given as 2 actuations of BDA MDI 40/90 µg per puff) and 160/180 µg (given as 2 actuations of BDA MDI 80/90 µg per puff), are included in this study to support final dose selection for approval. Children aged 4 to 91 years will only be randomized to the lower dosage level of BDA MDI (80/180 µg QID) or AS MDI [180 µg QID], or placebo MDI).

The treatment duration of 12 weeks for each subject, is considered to be an appropriate duration to evaluate lung function benefit in asthma subjects. This is supported by a 12-week standard treatment duration being assessed in Symbicort® (budesonide/formoterol fumarate dihydrate), Breo Ellipta (fluticasone/furoate and vilanterol), and Advair® (fluticasone/propionate/salmeterol) lung function studies (Symbicort [Corren 2007 and Noonan 2006], Breo [Kerwin 2017], Advair [Kavuru 2000]).

Two dose levels of BDA MDI will be used to evaluate the dual-primary efficacy measures versus the mono-components BD MDI 160 ug OID and AS MDI 180 ug OID as active control groups in order to demonstrate the combination rule and to compare efficacy outcomes.

Dual-primary efficacy measures have been selected to demonstrate the therapeutic contribution of each component of the combination to the overall bronchodilator efficacy:

## 1.3

Change from baseline in forced expiratory volume in 1 second (FEV<sub>1</sub>) area under the curve such application from 0 to 6 hours (AUC<sub>0-6 hours</sub>) over 12 weeks

Change from baseline in trough FEV<sub>1</sub> at Week 12

Benefit/risk and ethical assessment

study consists of 12 weeks of treatment and 2 weeks of safety follow-unixonian in the effect of BDA MDI on asthma symptoms and all design for lung function. This study consists of 12 weeks of treatment and 2 weeks of safety follow-up designed to evaluate the effect of BDA MDI on asthma symptoms and lung function. This study with its typical design for lung function studies is complementary to the AV003\MANDALA study evaluating the effect of BDA MDI on the occurrence of severe asthma exacerbations and is part of the regulatory requirements for US registration of BDA MDI for an asthma indication. This study has 2 active control groups (BD MDI and AS MDI), and a placebo MDI control group, designed. SABA (Ventolin®) will also be provided to each subject prn in response to asthma symptoms.

It should be noted that as part of this study design, some of the subjects who have not received ICS before may be assigned to treatmen with BD MDI or BDA MDI. In addition, some subjects who have been receiving low-dose ICS may be randomized to either placebo MDI or AS MDI (ie, they will no longer be receiving ICS treatment).

To mitigate potential risks, all subjects will be closely monitored to ensure subject safety throughout the study through a range of mechanisms including:

- Frequently evaluated by investigator during clinic visits at Weeks 1, 4, 8, and 12.
- Subjects will provide information to the electronic diary (eDiary) including; asthma symptoms segre, use of Ventolin prn in response to asthma symptoms, dosing of Sponsorprovided investigational product (IP, captured in eDiary in evenings only), and peak expiratory flow (PEF) twice daily. In the situation where the subject's symptoms and/or Ventolin prn use has increased and/or PEF decreased over 2 days, an eDiary alert is created and sent to the subject, the investigator site, and the Sponsor's medical monitoring team. This alert should initiate contact between the subject and the investigator site to determine the well-being of the subject.
- The eDiary will be programmed to alert both the subject and study center to assess the wellbeing of the subject and any possible asthma exacerbation.
- An Independent Data Monitoring Committee (IDMC) will be established to assess the ongoing safety of the study.

The Sponsor's medical team will have medical oversight of blinded data for continuous subject safety evaluations.

The Sponsor considers the risk and benefit profile of Study AV004-DENALI to be acceptable when considering and assessing all non-clinical and clinical data available for study treatments.

## COVID-19

Recent information from the American Academy of Allery Asthma and Immunology (AAAA) published on their website (https://www.aaaai.org/) on June 4, 2020 indicates that currently there is no evidence of increased infection rates in subjects with asthma and that it is best to get and keep their asthma under control." In the DENALI study, subjects are provided Vestolin for as needed use and have their asthma symptoms closely monitored through daily. Wiary symptom alerts provided to the investigator and medical monitors. The Sponsor believes that the benefitrisk assessment for trial participants to enroll and continue in the study remains positive. of an

1.4 Study design

This is a 12-week, randomized, double-blind, placebo convolled, multicenter, parallel group, Phase III study. The purpose of this study is to compare 2 dose levels of BDA MDI compared to its constitute components BD MDI and AS MDY on improvement in lung function and asthma symptoms after 12 weeks of treatment (Section 5.1.1) in adults, adolescents, and child subjects, aged 4 years and older, with symptomatic astoma currently being treated with SABA prn alone or with low-dose ICS maintenance therap plus SABA prn.

Subjects meeting all entry criteria atthe screening visit (Visit 1) will enter a 14 to 28-day screening (run-in) period.

Only Sponsor-provided IP diministered 4 times per day (QID) and Sponsor-provided Ventolin to be used in response to asthma symptoms are allowed during the study. No other asthma medications are allowed during the study.

During the screening (run-in) period, subjects will self-administer single-blind placebo MDI QID and Ventokin prn to be used in response to asthma symptoms only. Subjects will be trained and instructed in the use of an eDiary and peak flow meter at Visit 1 to record protocol required data into the eDiary twice daily (Section 5.1.6).

Eligible subjects will be randomized at Visit 2.

At randomization (Visit 2), adult and adolescent subjects (age ≥12 years) who meet the eligibility criteria will be randomly assigned to 1 of the following 5 treatment groups in a 1:1:1:1:1 ratio:

- BDA MDI 80/180 µg QID (given as 2 actuations of BDA MDI 40/90 µg per puff)
- BDA MDI 160/180 µg QID (given as 2 actuations of BDA MDI 80/90 µg per puff)
- BD MDI 160 µg QID (given as 2 actuations of BD MDI 80 µg per puff)

Children aged 4 to 11 will be randomized in a 1:1:1 ratio only to the lower BDA MDI QID of cauch additional dosage, AS MDI QID, or placebo MDI QID.

Ventolin will be provided to all subjects for prn use in response to asthma symptoms with a daily dosing recommendation not to exceed 8 puffs per day. See Figure 1 for a graphical presentation of the study schema and Table 1 for a list of study assessments and Table 2 fax 3 assessments at Visit 2 through Visit 6.

The study will

The study will consist of 3 periods:

- A screening/run-in period (14 to 28 days).
- A 12-week treatment period.

A safety follow-up period: where a safety fellow-up TC will occur 2 weeks (±4 days) after the subject's last dose of treatment (end-of-treatment [EOT]) or premature discontinuation visit (PDV).

The study will be completed when the study will be completed when telephone contact. Subjects who discontinue IP prior to the end of the 12-week treatment period will be withdrawn from the study and will be asked to complete a PDV, and adverse events This document must not be used to support (AEs)/serious AEs (SAEs) will be followed up if medically indicated.

Figure 1 Study design



Abbreviations: AS MDI=albuterol metered-dose inhaler; BD MDI=budesonide metered-dose inhaler; BDA MDI=budesonide/albuterol metered-dose inhaler; N=humber; placebo MDI=placebo metered-dose inhaler; PRN=as needed; QID=four time daily; R=randomization; SV=screening visit; W=week.

#### 1.5 Study governance and oversight

#### 1.5.1 Independent data monitoring committee

An IDMC will be established to assess the ongoing safety of the study. The IDMC will review blinded data (open session) and unblinded safety data (closed session) to assess any safety related reasons why the tudy should continue, be modified, or stopped. Closed sessions will be supported by the anblinded statistician and responsibilities of the IDMC will be clarified within a charter before initiation of the study.

The IDMC chair and all committee members will be independent investigators/specialists separate from the study team or contract research organization.

documen recommendation made to the Sponsor. decisions made by the IDMC will be documented within written records of meetings and

# 2 STUDY OBJECTIVES

# 2.1 Primary objectives

| Primary objective: | Primary endpoints: |
|---|---|
| To demonstrate the contribution of budesonide | Dual-primary endpoints: |
| and albuterol in BDA MDI 80/180 µg and | • Change from baseline in FEV <sub>1</sub> AUC <sub>0-6 hours</sub> over |
| 160/180 μg administered QID by comparing with | 12 weeks |
| mono-components (BD MDI 160 µg, AS MDI 180 | • Change from baseline in trough FEV $_1$ at |
| μg) and placebo on lung function | Week 12 |

# 2.2 Secondary objectives

| Secondary objective: | Secondary endpoints: |
|---|---|
| To characterize the effect of BDA MDI 80/180 μg and 160/180 μg administered QID on bronchodilation and asthma symptoms compared to the mono-components (BD MDI 160 μg, AS MDI 180 μg) and placebo | <ul> <li>The time to onset (defined as 15% increase in FEV1 over the predicatment value on Day 1), and duration of response on Day 1</li> <li>Number (%) of subjects who have an Asthma Control Questionnaire-7 (ACQ-7) score of ≥1.5 at baseline who achieve a clinically meaningful improvement (a decrease of at least 0.5 units</li> <li>from baseline) in ACQ-7 at Week 12</li> <li>Trough FEV1 at Week 1</li> </ul> |

# 2.3 Safety objectives

| Safety objective: | Safety endpoints: |
|---|---|
| To evaluate the safety and tolerability of BDA | • AE/SAEs |
| MDI 80/180 μg and 160/180 to administered QID | • Vital signs (ie, heart rate, blood pressure only) |
| compared to BD MDI (1600g) and AS MDI (180 µg) | Clinical chemistry and hematology parameters |
| , x0 3 | • Electrocardiogram (ECG) |
| This document must not be used to | |

# 2.4 Exploratory objectives

| Exploratory objective: | Exploratory endpoints: |
|---|---|
| To characterize the effect of BDA MDI 80/180 μg and 160/180 μg administered QID on bronchodilation and asthma symptoms compared to the mono-components (BD MDI 160 μg, AS MDI 180 μg) and placebo | <ul> <li>Deteriorations of asthma</li> <li>Incidence of severe exacerbations</li> <li>Change from baseline in: <ul> <li>Trough FEV<sub>1</sub> at individual time points</li> <li>FEV<sub>1</sub> AUC<sub>0-6 hours</sub> at individual time points</li> <li>Peak change from baseline FEV<sub>1</sub> at David and Day 7</li> <li>Morning and evening PEF</li> <li>Use of Ventolin therapy in response to asthma symptoms</li> <li>Asthma daytime/night time symptoms</li> <li>Asthma Control Questionaire-5 (ACQ-5) and responder analysis at Week 12</li> <li>Asthma Quality of Life Questionnaire +12 for 12 years and older (AQLQ+12)/Pediatric</li> <li>Asthma Quality of Life Questionnaire (PAQLQ) change from baseline at Week 12</li> </ul> </li> </ul> |

# 3 SUBJECT SELECTION, ENROLLMENT, RANDOMIZATION, RESTRICTIONS, TREATMENT DISCONTINUATION, AND STUDY TERMINATION

Each subject must meet all of the inclusion criteria and none of the exclusion criteria for this study.

No study-related procedures may be performed before the subject has signed the Ethics Committee (EC) approved Informed Consent Form (ICF)/assent form.

# 3.1 Miclusion criteria

For inclosion in the study, subjects must fulfill the following criteria within the screening period:

Able and willing to provide written informed consent or sign age-appropriate forms; subjects below legal age of consent must have parent(s) or guardian sign the ICF before participation

2 Female or male aged ≥4 years at the time of informed consent. In the Czech Republic, Germany, Serbia, Slovakia, and Ukraine only subjects ≥18 years will be included.

- Diagnosis of asthma as defined by GINA criteria with a documented history of the last 6 months prior to Visit 1
- of such application Receiving 1 of the following inhaled asthma medications with stable dosing for at least 30 days prior to Visit 1:
  - (a) Only SABA used prn
  - (b) Stable low-dose ICS (Appendix C, GINA 2018) in addition to prn use of SABA The following defines the minimally acceptable documentation required to support inclusion criterion 4:
    - Signed and dated notes from a referring physician, including name, doss, and duration of the SABA or SABA with low-dose ICS (or names and doses, if used as separate inhalers), if applicable, and/or
    - Evidence of prescriptions for SABA or SABA with low-dosoiCS, if applicable, medications that demonstrate coverage for the duration specified in inclusion criteria
- Pre-bronchodilator FEV₁ of ≥50 to <85% predicted normal value for adults (≥18 years of age) and ≥50% predicted normal value for subjects aged 4 to 17 years after withholding SABA ≥6 hours at Visit 1. If subject took SABA or viry bronchodilator in the morning of Visit 1, either the entire visit must be rescheduled 8r just PFT assessment rescheduled. Subjects 4 to 17 years of age who previously: wiled inclusion criteria 5 due to the upper FEV<sub>1</sub> limit will be permitted to re-screen once and will be required to meet all eligibility criteria upon re-screening.
- Demonstrate reversibility of airflow limitation defined as a  $\geq 15\%$  increase in FEV<sub>1</sub> relative to baseline after administration of Sponsor-provided SABA (Ventolin) at either Visit 1 or Visit 1a. One re-test for reversibility testing is allowed within the screening period prior to Visit 2
- period prior to Visit 2

  Demonstrate acceptable spirometry performance (ie, meet American Thoracic Society/European Respiratory Society [ATS/ERS]) acceptability/repeatability criteria (Appendix K, Spirometry Assessment Criteria). Subjects 4 to 11 years will be eligible if they provide 2 acceptable / repeatable measurements.
- 8 Taken Wentolin on  $\geq 2$  days out of 7 days prior to Visit 2
- Willing and, in the opinion of the investigator, able to adjust current asthma therapy, as squired by the protocol
  - Demonstrate acceptable metered-dose-inhaler (MDI) administration technique as assessed by the investigator. Note: spacer use is not allowed throughout the screening and randomized treatment periods
- 11 Able to perform acceptable and reproducible PEF measurements as assessed by the investigator
- 12 Body mass index (BMI) <40 kg/m<sup>2</sup>

- 13 Willing to remain at the study site as required per protocol and complete all visit assessments
- 14 Negative pregnancy test (serum at Visit 1) for female subjects of childbearing potential
- 15 Women of childbearing potential and sexually active in heterosexual relationships must agree to 1 of the following options to prevent pregnancy:
  - (a) Practice complete abstinence defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. Periodic abstinence is not acceptable. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and esual lifestyle of the subject. Therefore, complete abstinence is an acceptable method of contraception only if it is consistent with the preferred and usual lifestyle of the subject.
  - (b) If a female of childbearing potential agrees to prevent pregnancial following effective methods of birth control from the date the ICF is signed until 2 weeks after the final dose of IP is taken:
    - Hormonal contraception (eg, oral contraceptive, contraceptive implant, or injectable hormonal contraceptive)
    - Double-barrier birth control (eg, a combination of male condom with either ii. cap, diaphragm, or sponge with spermicide)
    - iii. Maintenance of a monogamous sexual relationship with a male partner who has been surgically sterilized by vasectomy
  - (c) Note: Women are considered to be of nonchildbearing potential if they are physiologically incapable of becoming pregnant, including any female who is 2 years postmenopausal, or surgically sterile, defined as having a bilateral oophorectomy, hysterectomy, tubal ligation, or other permanent birth control measures. For purposes of this protocol, menopausal women are defined as women that are amenorrheic for 12 consecutive months or more after cessation of all exogenous hormonal treatment. Adolescent specific recommendations: if subject is female and has reached menarche or has reached Tanner stage 3 breast developments (even if not having reached
- sterile or agree to use a double-barrier effective method of contraception (condom with subjects must not donate sperm during their study participation period.

  3.2 Exclusion criteria

  Subjects must not enter the the subjects must not enter the subjects

the screening period:


- Chronic obstructive pulmonary disease or other significant lung disease (eg, chronic bronchitis, emphysema, bronchiectasis with the need of treatment, cystic fibrosis, or bronchopulmonary dysplasia)

- Received any marketed (eg, omalizumab, mepolizumab, reslizumab, benralizumab, dupilumab) or investigational biologic within 3 months or 5 half-lives before Visit 1, whichever is longer, or any other prohibited medication

  Current smokers, former smokers with >10 pack-years history, or former smokers topped smoking <6 months before Visit 1 (including all for [vaping], and marijuana)

  Life-threatening
- Life-threatening asthma defined as any history of significant asthma episode(s) requiring admission to an intensive care unit, intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma-related syncopal episode(s) within 5 years of Visit 1
- Completed treatment for lower respiratory infection within 6 weeks prior to Visit 1
- Upper respiratory infection involving antibiotic treatment not resolved within 7 days prior to Visit 1
- Hospitalizations due to asthma within 6 prior to Visit 1
- 10 Have taken ≥12 actuations per day of Sponsor-provided Ventolin during the run-in period prior to Visit 2 according to the below criteria:
  - (a)  $\geq 2$  days out of 14 days of runcing
  - (b)  $\geq$ 3 days out of 15 to 21 days of run-in
  - (c) ≥4 days out of 22 or more days of run-in
- 11 Unable to comply with study procedures including non-compliance with diary completion (ie, <70% subject completion of diary assessments in the last 7 days preceding Visit 2 or QID dosing, < 80% compliance during the placebo run-in period)
- 12 Clinically significant laboratory abnormalities, in the opinion of the investigator, or having any of the following results at Visit 1:
  - (a) Serum creatinine value >1.5 times the upper limit of the reference range
  - a serum total bilirubin value (TBL) >1.5 times the upper limit of the reference range
  - (c) a serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >2.5 times the upper limit of the reference range

Note: Laboratory tests may be repeated once: if laboratory tests have to be repeated, the results must be available for review before Visit 2 (randomization).

13 Any of the following results at Visit 1:

- (a) an abnormal electrocardiogram (ECG) that is, in the investigator's opinion, clinically significant
- (b) a QTC<sub>F</sub> interval >480 ms (subjects aged  $\geq$ 12 years)/ $\geq$ 460 ms (subjects aged 4 to 11 years, based on the Fridericia correction where QT<sub>c</sub>F=QT/RR<sup>0.33</sup>)
- Historical or current evidence of a clinically significant disease including, but not limited to: cardiovascular (eg, congestive heart failure, known aortic aneurysm, clinically significant cardiac arrhythmia, coronary heart disease), hepatic, renal, hematological, neuropsychological, endocrine (eg, uncontrolled diabetes mellitus, uncontrolled thyrold disorder, Addison's disease, Cushing's syndrome), or gastrointestinal (eg, poorly controlled peptic ulcer, gastroesophageal reflux disease) disorders. Significant defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through study participation, or that could affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
- 15 Cancer not in complete remission for at least 5 years before Visit 1 Note: Subjects with squamous cell carcinoma of the skin, basal cell carcinoma of the skin, in situ carcinoma of the cervix, or localized prostate cancer are eligible, if in the opinion of the investigator, the condition has been clinically controlled and the subject's participation in the study would not represent safety concern.
- 16 Hospitalization for psychiatric disorder or attempted suicide within 1 year of Visit 1
- 17 History of psychiatric disease, intellectual deficiency, poor motivation, or other conditions if their magnitude is maintain informed consent validity
- 18 Significant abuse of alcohol or drugs, in the opinion of the investigator
- 19 A known or suspected hypersensitivity to albuterol/salbutamol, or budesonide and/or their excipients
- 20 A scheduled/planned hapitalization during the study
- 21 Inability to abstain from protocol-defined prohibited medications during the study
- 22 Using any herbar products by inhalation or nebulizer within 2 weeks of Visit 1 and not agreeing to cop during the study duration
- 23 Receive a live attenuated vaccination within 7 days of Visit 1
- 24 Currently pregnant or breastfeeding
- 25 Study investigators, sub investigators, coordinators, and their employees or immediate family members, or employees of the Sponsor
- Treatment with any investigational treatment or device in another clinical study within the last 30 days (or 5 half-lives, whichever is longer) of Visit 1
- 27 Currently participating in any interventional study
- 28 Previously been randomized in this study or any other PT007 or PT027 clinical study. For pediatrics, see inclusion criterion 4.

This do

Procedures for withdrawal of incorrectly enrolled subjects are described in Section 3.4.

and adolescent subjects (≥12 years of age) with asthma will be and adolescent subjects (≥12 years of age) with asthma will be and adolescent subjects (≥12 years of age) with asthma will be MDI 80/180 µg QID, BDA MDI 160/180 µg QID, BD MDI 160 µg QID, or AS MDI 180 µg QID or placebo MDI). In addition, up to 30 child subjects (4 to 11 years of age) with asthma will be enrolled but will not receive high dose ICS and will be low-dose BDA MDI 80/180 µg QID and Q 2000 subjects will need to be screened, assuming an estimated screen failure rate of 50% prior to randomization. This Phase III study is planned to be conducted globally.

The investigator(s) and/or study personnel will:

- Obtain signed informed consent/assent (as applicable) from the potential subject and/or their guardian/legal representative before any study specific procedures are performed
- Enter the subject data into the enrollment module in Rave Web Based Data Capture (WBDC) electronic case report form (eCRF) to enable the allocation of subject identification (Ecode)
- Determine subject eligibility (Sections 3.1 and 3.2)
- Enter the information required to enable the Interactive Web Response System (IWRS) to initiate randomization and generate the randomization code

Randomization codes will be assigned through IWRS strictly sequentially to subjects eligible for randomization. If a subject worldraws from participation in the study, then his/her randomization code cannot be eused.

# Procedures for handling incorrectly enrolled or randomized 3.4

Subjects who call to meet the eligibility criteria should not, under any circumstances, be randomize for receive IP. There can be no waivers granted from the Sponsor for any subject not meeting inclusion or exclusion criteria.

Sincorrectly started on-treatment, the investigator should inform the medical monitor assigned to the project immediately, and a discussion should occur between the medical monitor assigned to the project and the investigator regarding with subject from treatment. subject from treatment. The Sponsor's medical monitor assigned to the project must ensure all decisions and protocol deviations, if any, are appropriately documented.

#### 3.5 Methods for assigning treatment groups

A randomization schedule will be generated by a designated statistical representative of such application performing statistical support for the study. This schedule will be prepared before the start of the treatment period. The designated statistical representative will follow their established standard operating procedures regarding generation, security, and distribution of the randomization schedule. Randomization will be centralized.

Randomization for adults and adolescents will be centralized and stratified by pre-study background therapy consisting of either ICS or non-ICS (subjects not previously treated with ICS), by Asthma Control Questionnaire-7 (ACQ-7;  $\leq 1.5$ ,  $\geq 1.5$ ), and by age ( $\geq 12$  to  $\langle 07, \geq 18 \rangle$ ). Children aged 4 to 11 years will not be stratified.

Upon enrollment, subjects will be assigned a unique subject identification code (Ecode) which is automatically generated by the electronic data capture system (Rave BDC) based on the order of entry. Once it has been determined that a subject meets all engibility criteria, the subject information will be integrated into the IWRS (Randomization and Trial Supply Management) for randomization.

# 3.6

Methods for ensuring blinding P plication blind is to be made in the manner of the man The study blind is to be maintained until all subjects have completed the treatment period and until after the database has been locked. The study site receives documentation of subject study identification and kit allocation through the IWRS. The randomization code will not be available, with the exception of unblinding procedures described in Section 3.7, to the study team, study center personnel, Sponsor monitors, Sponsor project statisticians, or any other personnel employed or affiliated with the Sponsor, as well as investigators and subjects until after the database has been locked.

The 5 different kit types of study IP are visually identical, protecting the blind through their similarity in appearance

#### Methods for unblinding 3.7

The treatment blind should not be broken except in medical emergencies and based on the investigator's clinical judgement when the appropriate management and welfare of the subject requires knowledge of the treatment allocation. Individual treatment details, for each subject, will be available to the investigator(s) or pharmacists from the IWRS, if needed. If unblinding occurs, the investigator must notify the Sponsor as soon as possible, but without revealing the treatment assignment of the unblinded subject. Routines for this will be described in the IWRS user manual that will be provided to each center. The IWRS provides unblinding procedures, if needed.

The designated representative retains the right to break the code for SAEs that are unexpected and are suspected to be causally related to an IP and that potentially require expedited reporting to regulatory authorities. Treatment codes will not be broken for the planned analyses of data until all decisions on the evaluability of the data from each individual subject have been made and documented.

With the exception of emergency unblinding as described above, all members of the study team, investigators, and site staff will be blinded. The only individuals who will have access to unblinded information during the conduct of the study in advance of the primary outcome database lock will be the unblinded statistician supporting the IDMC closed session review which will be performed in accordance with the IDMC charter.

## 3.8 Restrictions

Subjects should be advised that marketed (eg, omalizumab, mepolizumab, reslizumab, benralizumab) or investigational biologic treatments are not allowed during the treatment period. Subjects requiring chronic SCS are excluded.

Only Sponsor-provided IP and Sponsor-provided Ventoling be used in response to asthma symptoms are allowed during the study. No other atthred medications are allowed during the study. Restrictions regarding concomitant medications are described in Section 7.8.

Subjects should not take Sponsor-provided Ventolin ≤6 hours before a study visit (if Ventolin is needed in the morning of a study visit, either the entire visit must be rescheduled or just PFT assessment rescheduled).

Subjects should avoid strenuous exercise for at least 30 minutes prior to a study visit.

Subjects should avoid having a large meal at least 2 hours prior to a study visit.

Subjects must not inger xanthine and/or xanthine analogue (caffeine)-containing foods and beverages for at least 6 hours prior to and for the duration of each in-clinic study visit. Examples of such products include coffee, tea, chocolate, and cola. Decaffeinated beverages are acceptable.

Illicit crugs or drugs of abuse will not be allowed from Visit 1 to the end of the follow-up telephone contact or to whenever the subject withdraws from the study. If any illicit drugs or trugs of abuse are used by the subject during the study, the dates of use and the amount will be documented, and the subject will be discontinued at the discretion of the Investigator. Medical marijuana is not an exclusionary drug if used for medical purposes, and there is no change in the dose or frequency of consumption.

#### 3.9 Treatment discontinuation by subject and/or Sponsor

Subjects may be withdrawn from the study at any time at their own request, upon request of and AE considered to jeopardize the safety of a subject participating in the study
Subjects who suffer 1 severe exacerbation should be considered for discontinuation if of Sponsor and the investigator decide that it is in the best interest of the subject to discontinue randomized treatment and withdraw from the study

In the opinion of the investigator, the subject to Protocol (eg. post the investigator, or by the Sponsor at any time or for any reason. The subject or his/her parent/legal representative is free to discontinue treatment at any time, without prejudice to further treatment. Other reasons for IP discontinuation may include:

- or is lost to follow-up and no alternative contact information is available (this implies that at least 2 documented attempts have been made to contact the subject)
- If female subject becomes pregnant, the subject will automatically be discontinued from
- In subjects who have elevated liver enzymes AST and or ALT ≥3 times the upper limit of normal (×ULN) and total bilirubin ≥2×ULN (e, meeting the criteria of at least potential Hy's Law), IP will be suspended until the Divertest values return to the normal range. If the AST, ALT, or total bilirubin reach these elevated levels again, after recommencement of IP, the subject will be discontinued from IP and withdrawn from the study.

Subjects who discontinue IP prior to the end of the 12-week treatment period will be withdrawn from the study and will be sked to complete a PDV, and AEs/SAEs will be followed up if medically indicated

A subject that decides to discontinue IP will always be asked about the reason(s) and the presence of any AEs. If wassible, they will be seen and assessed by an investigator(s). AEs and SAEs will be followed up (Section 6); eDiary and all IPs should be returned by the subject.

#### Study termination 3.10

If the Sporsor, investigator, study monitor, IDMC, or regulatory officials discover conditions arising during the study that indicate that the subject's safety and/or scientific value of the stude and/or quality of the IPs have been compromised, the study may be halted or the study center's participation may be terminated. Ongoing subjects will be discontinued from the study and assigned to receive treatment as per local standard of care.

Conditions that may warrant termination of the study include, but are not limited to, the following list:

- The study may be stopped if, in the judgement of the Sponsor, study subjects are placed at undue risk because of findings that:
  - are considered significant
- are not considered to be consistent with continuation of the study

  The discovery of an unexpected, serious, or unacceptable risk to the subjects enrolled in the study

  A decision on the part of the Sponsor to suspend or discontinue testing, evaluation of development of the IP for any reason

  ditions that may warrant termination of a study ted to, the follow:

Conditions that may warrant termination of a study center's participation include, but are not limited to, the following list:

- Failure of the investigator to enroll subjects into the study at an acceptable rate or within an agreed timeline
- Failure of the investigator to comply with pertinent governing body regulations
- Submission of knowingly false information from the research facility to the Sponsor, study monitor, medical officer, or regulatory official
- Insufficient adherence to protocol requirements

Regardless of the reason for termination, all data available for the subject at the time of discontinuation of follow-up must be recorded in the eCRF. All reasons for discontinuation of treatment must be documented.

In terminating the study, the Sponsor will ensure that adequate consideration is given to the protection of the subjects' interests.

Study termination and follow-up will be performed in compliance with applicable governing body regulations

## Screen failures 3.11

Screening failures are subjects who do not fulfill the eligibility criteria for the study, and therefore must not be randomized. These subjects, who have a reason for not enrolling to the stady, should be recorded as 'Screen failure'. Subjects who are screen failures will not be re-Screened with the exception of children and adolescents who screen-failed because they did not meet the now obsolete upper FEV1 % predicted limit. Children and adolescents who previously failed to meet the upper FEV1 % predicted threshold, but who met all other eligibility requirements, may re-screen once. Upon re-screening, these subjects must meet all eligibility requirements in order to be randomized.

#### 4 STUDY PLAN AND TIMING OF PROCEDURES

Table 1 presents study assessments and procedures and Table 2 presents timed assessments at Visit 2 through Visit 6. Repeat assessments, if needed, will be captured in unscheduled visits.

#### **General Considerations**

- For subjects who inadvertently took IP, SABA, or any bronchodilator in the morning of any study visit, either the entire visit must be rescheduled or just PFT assessment and beverages for at least 6 hor study visit. study visit. Examples of such products include coffee, tea, chocolate, and cola. Decaffeinated beverages are acceptable.
- Subjects should avoid having a large meal at least 2 hours prior a study visit.
- Subjects will be required to return to the clinic at approximately the same time at Visit 2 for all treatment visits (±2 hours) and dosing time should not exceed 10:00 AM and pulmonary function tests (PFTs) should be completed within  $\pm 1$  hour of Visit 2. Subjects will be required to remain at clinic until completion of all protocol-defined assessments. In order to minimize diurnal variance, sites should make every effort to assess subjects at the same time throughout the study.
- IP should be taken in the morning upon waking, and then distributed equally throughout the day with the final dose taken before going to sleep. The evening before clinic visits, subjects should be advised to take the last dose at  $22:00 \pm 2$  hours.
- To ensure dosing time standardization, it is recommended that sites encourage subjects to maintain a dosing schedule consistent with their in-clinic dosing time and that sites call the subjects on the day before a scheduled visit to remind the subject of the following:
  - To take their last dose the evening before the scheduled visit
  - To withhold a Rinhaled medications (oral and intranasal) for at least 6 hours prior to **PFTs**
  - To bring their study medications and eDiary with them to the clinic

Site personnel will instruct subjects not to take any inhaled medications, without site Should take every precaution to prevent subject use of and Ventolin prior to the visit start before performing any study procedures and return the IP and Ventolin to the subject at the end of the visit when all study procedures are completed, and the Subjects will be asked to abstain wherever possible for a subject is experience. personnel permission, during a visit until all study procedures have been completed, and the arthma medications during the test day. Site personnel may request the subject to surrender all IP and Ventolin to the subject at the end of the visit when all study procedures are completed. Subjects will be asked to abstain wherever possible from using Ventolin during study visits. If symptoms at any time during a test day, site personnel must note the time and justification of

The decorate trade and the based to support out make the last.
Table 1 Study assessments and procedures

| | Screening (run-in) <sup>b</sup> | | Double-i | blind Treatme | ent Period | | PDV <sup>d</sup> (if applicable) | Safety Follow-up TC (2 weeks [±4 days] after treatment discontinuation) |
|---|---|---|---|---|---|---|---|---|
| Visit <sup>a</sup> | 1 (1/1a) | 2 | 3 | 4 | 5 | 6 <sup>c</sup> | of | (2 weeks [±4 days] after |
| Week | -4 to -2 | 0 | 1 | 4 | 8 | 12 | rion | treatment discontinuation) |
| Day | -28 to -14 | 1 | 7±2 | 28±2 | 56±2 | | ailat | |
| Informed consent | X | | | | | of any | | |
| Eligibility criteria | X | X | | | × | 6<br>0, | | |
| Routine clinical procedures | | | • | | of jico | • | | |
| Medical/surgical history<br>(including any on-study<br>medical/surgical procedures) <sup>e</sup> | X | X | X | | p x | X | X | |
| Demography | X | | | | | | | |
| Physical examination <sup>f</sup> | X | | QK. | alit | | X | X | |
| Concomitant medications | X | X | nakeino | X | X | X | X | Х |
| SABA reversibility test <sup>g</sup> | X | .6 | Wa | | | | | |
| Safety measurements | | X.O | | | | | | |
| Vital signs (HR and BP only) | X | 106x | X | X | X | X | X | |
| 12-lead ECG | X xO | o X | | | | X | X | |
| Adverse events | x edic | X | X | X | X | X | X | X |
| Pregnancy test <sup>h</sup> | XUSE | X | X | X | X | X | X | |
| Safety laboratory assessments (clinical chemistry, hematology) | X X X X X X X X X X X X X X X X X X X | | | | | X | X | |

| | Screening (run-in) <sup>b</sup> | | Double-i | blind Treatme | ent Period | | PDV <sup>d</sup> (if applicable) | Safety Follow-up TC |
|---|---|---|---|---|---|---|---|---|
| Visit a | 1 (1/1a) | 2 | 3 | 4 | 5 | 6 <sup>c</sup> | | (2 weeks [±4 days] after |
| Week | -4 to -2 | 0 | 1 | 4 | 8 | 12 | | Di treatment atscontinuation) |
| Day | -28 to -14 | 1 | 7±2 | 28±2 | 56±2 | 84±2 | ationor | |
| Efficacy measurements | | | | | | | alle | |
| Spirometry (FEV <sub>1</sub> ) <sup>i</sup> | X | X | X | X | X | $X^{\mathcal{A}}$ | X | |
| ACQ-5 | X | X | X | X | X | orany | X | |
| ACQ-7 | X | X | X | X | RY phical | o x | X | |
| AQLQ+12/PAQLQ | | X | | х | 84 aplice | X | X | |
| Review of PEF, use of Ventolin<br>therapy, asthma daytime/night-<br>time symptoms, night-time<br>awakenings due to asthma<br>symptoms <sup>j</sup> | | X | x Reting | | p<br>X | X | X | |
| Dispense/collect eDiary (AM3+) | X | | 5.0 | S. | | X | X | |
| Review compliance with eDiary | | X | or Metil. | X | X | X | X | |
| Investigational product administ | tration | | Wel. | | | | | |
| IP compliance | | X of | X | X | X | X | X | |
| Randomization | | OPR | | | | | | |
| IP (dispense/collect) <sup>k</sup> | d vO | c/dk | c/d | c/d | c/d | c/d <sup>n</sup> | c/d <sup>n</sup> | |
| Ventolin (collect/dispense) | disedie | $c/d^l$ | c/d <sup>l</sup> | c/d <sup>l</sup> | c/dl | С | c | |
| Ventolin administration<br>(recorded in MasterScope) | tration d d d d d S T D X | | | | | | | |
| IP administration (recorded in MasterScope) <sup>m</sup> | \$``<br> | X | X | X | X | X | X | |

Abbreviations: ACQ-5=Asthma Control Questionnaire-5; ACQ-7=Asthma Control Questionnaire-7; AQLQ+12= Asthma Quality of Life Questionnaire-3 12 years and older; β-hCG=β-human chorionic gonadotropin: RP=blood pressure: a= collect. d=discusses RP.  $\beta$ -hCG=  $\beta$ -human chorionic gonadotropin; BP=blood pressure; c= collect; d=dispense; eDiary=electronic diary; ECG=electrocardiogram; FEV<sub>1</sub>- $\beta$ -orced expiratory volume in I second; HR=heart rate; IP=investigational product; PAQLQ=Pediatric Asthma Quality of Life Questionnaire; PDV= premature discontinuation visit; PEF= peak expiratory flow; OID=4 times daily; SABA=short/rapid-acting β2-adrenoreceptor agonist; TC=telephone contact; V=visit

- Screening (run-in) Period may be 14 to 28 days. Visit 1 may be split (used for repeated assessments, if needed) for the repeat assessment of SABA reversibility test, if cable.

  Planned end-of-treatment (EOT) will occur at Visit 6. applicable.
- Subjects who prematurely withdraw (withdraw pre-week 12) from study treatment will undergo a PDV.
- Details of any surgical procedures occurring during randomization and the treatment period will be also recorded.
- Includes evaluation of height, body mass index, and weight at Visit 1 and weight only for Visit 6 or PDV. Demonstrate reversibility at Visit 1, with an increase in FEV $_1 \ge 15\%$  relative to baseline after administration of Sponsor-provided Ventolin via central spirometry at either Visit 1 (reversibility must be demonstrated at either Visit 1 or Visit 1a); Visit 1a will be used for re-testing, if needed; with only 1 reversibility re-test permitted prior to randomization (Visit 2).
- Mization (+ isit 2).
  A serum pregnancy test (β-hCG) will be performed at Visits 1 and treatment discontinuation (EOT) or PDV? urine β-hCG test will be performed at all other visits (for women of childbearing potential only).
- Pre-bronchodilator (Visit 1/Visit 1a)/Pre-dose (Visit 2 onwards) FEV1 will be measured in the morning between 06:00 and 10:00 AM at the designated visits in Table 1, and within 1 hour of FEV1 measured at Visit 2. Pre-bronchodilator FEV1 of  $\geq$ 50 to <85% predicted formal value for adults ( $\geq$ 18 years of age) and  $\geq$ 50% predicted normal value for subjects aged 4 to 17 years after withholding SABA ≥6 hours (at Visit 1 or Visit 1a, if applicate). If Sobject took SABA within 6 hours in the morning of Visit 1, either the entire visit must be rescheduled or just PFT assessment rescheduled. At Visit 1, pre- and post- dose will be with respect to administration of Sponsor-provided bronchodilator (Ventolin). From Visit 2 onwards, pre- and post- dose measurements will be with respect to administration IP.
- The eDiary (AM3+) will be dispensed at screening.
- All subjects will be assigned placebo during the run-in period for dosing QID. Compliance to dosing should be reviewed prior to randomization.
- Ventolin usage to be reviewed at each collection/dispensing visit using eDiary. Replacement kit dispensed as required. The actuator should be cleaned once per week if used in the last 7 days according to instruction summarized in Appendix J, Meter Hosen haler Handling and Cleaning.
- IP should be taken in the morning upon waking, and then distributed equal by throughout the day with the final dose taken before going to sleep. The evening before clinic visits, subjects should be advised to take the last dose at 22:00 (10:00 PM) ±2 dours. For all on-treatment visits, IP should be administered before 10:00 AM in the clinic using newly dispensed IP. The actuator should be cleaned once per week if used in the last 7 days according to instruction summarized in Appendix J, Metered-dose Inhaler Handling and Cleaning.
- IP will be dispensed at Visit 6 and PDV for performance of FEV measurements only, this will not be taken home by the subjects. IP dispensed at these visits will be retained at the site following the visit and reconciled for IP accountability

Table 2 Timed assessments at Visit 2 through Visit 6 and Premature Discontinuation Visit

| Clinical Variable | Pre-Dose | | IP<br>Dose | Post-Dose 5 min 15 min 30 min 45 min 60 min 120 100 240 300 360 min min min min min | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -60<br>min | -30<br>min | 0 min | 5 min | 15 min | 30 min | 45 min | 60 min | 120<br>min | ASO<br>min | 240<br>min | 300<br>min | 360<br>min |
| IP Collection <sup>h</sup> | Xª | | | | | | | | ariation | | | | |
| IP Dispensing <sup>i</sup> | Xa | | | | | | | | ailai | | | | |
| IP Dosing <sup>i</sup> | | | X | | | | | N | 70 | | | | |
| Questionnaires<br>ACQ-5<br>ACQ-7<br>AQLQ+12/PAQLQ | $X^{a,b}$ | | | | | R | Palication | or and | | | | | |
| Review of Electronic Diary | Xª | | | | | 0, | 64 | | | | | | |
| Vital Signs <sup>c</sup> | $X^{a,d}$ | | | | 4 | 60 410 | | | | | | | |
| 12-Lead ECG | X <sup>a,e</sup> | | | | | | | | | | | | |
| Clinical Laboratory<br>Testing | $X^{a,f}$ | | | | RE OUT | | | | | | | | |
| Spirometry (FEV <sub>1</sub> ) <sup>g</sup> | X | X | | X | e <sup>til</sup> X | X | X | X | X | X | X | X | X |

Abbreviations: ACQ-7=Asthma Control Questionnaire 7, AQLQ+12= Asthma Quality of Life Questionnaire for 12 years and older; ECG=electrocardiogram; FEV<sub>1</sub>= forced expiratory volume in 1 second; IP=investigational product; min=minute, PAQLQ=Pediatric Asthma Quality of Life Questionnaire; PDV= premature discontinuation visit **Note:** Time point for dosing is regarded as "0 minutes". When does collection time-points are concurrent, variables should be collected in the following order: Questionnaires, vital signs, ECG, clinical laboratory assessments, and spirometry.

- This is not a timed assessment. Sites should plan to perform these activities to allow for collection of timed spirometry.
- Questionnaires (ACQ-5, ACQ-7, AQLQ+12, and PAQLQ) are collected at all visits (except Visit 3 AQLQ+12, and PAQLQ).

  Vital signs should be started (approximately 5 to 0 minutes) ahead of the specified time point to ensure spirometry will be conducted as close to the specified time points as possible.
- Pre-dose vital signs (heart rate, blood pressure) will be collected twice, at least 5 minutes apart.

  Pre-dose ECG will be collected at Visit 2, Visit 6, and PDV only, or as clinically indicated.
- All clinical laboratory tests (hematology and chemistry) will be assessed approximately 60 minutes prior to dosing at Visit 6 in advance of first spirometry measurement. Laboratory tests may be performed at all other visits as clinically indicated.
- Every effort should be made to assess subjects' trough pre-dose and post-dose FEV1 at the same time throughout the study. Pre-dose FEV1 will be measured in the mornings between 06:00 and 10:00 AN, and within 1 hour of FEV<sub>1</sub> measured at Visit 2. From Visit 2 onwards, pre- and post-dose measurements will be with respect to administration of IP (Table 3).

At the start of each treatment visit, subjects must withhold all asthma medications, including Sponsor-provided Ventolin for at least 6 hours prior to start of test day procedures.

Dispense new IP to subjects for on-site dosing after trough pre-dose FEV1 measurement and for subsequent at-home use following the completion of all assessments. IP will be dosed before 10:00 AM following pre-dose FEV1 measurements at each visit At the start of each treatment visit, subjects must withhold all asthma medications, including Spansor-provided Ventolin for at least 6 hours prior testart of test day procedures.

Disponse new IP to subjects for on-site dosing after trough pre-dose FFV; measurement and for subsequent at-home use following the completion of all post-dose assessments. IP will be dosed before 10.00 AM following pre-dose FEV; measurements at each visit.

Out of the distribution of the dosed before the completion of all post-dose assessments. IP will be dosed before the completion of the dosed before the completion of t

## 4.1 Screening and enrollment period

Procedures will be performed according to study assessments and procedures presented in

Subjects meeting all entry criteria at the screening visit (Visit 1) will enter a 14- to 28-day screening (run-in) period. Subjects will discontinue their usual asthma medications at Visit of demographics, physical examination (including being medications review. Specification) demonstrated at either Visit 1 or Visit 1a; Visit 1a will be used for re-testing of needed; with only 1 reversibility re-test permitted prior to randomization [Visit 2]), vital signs (heart rate, blood pressure only), 12-lead ECG, AEs, serum pregnancy test, blood samples for hematology and clinical chemistry, FEV1 determination, Asthma Control Questionnaire-5 (ACQ-5), Asthma Control Questionnaire-7 (ACQ-7), dispensing/collecting eDiary, dispensing Ventolin, and administration of single-blind placebo MDI.

At Visit 1, placebo MDI and Sponsor-provided Ventolin prn to be used in response to asthma symptoms will be dispensed; during the screening (run-in) period, these will be the subject's only asthma medications. At Visit 2, compliance to placebo MDI dosing in screening (run-in) will be assessed by review eDiary completion as specified in the exclusion criteria. Ventolin usage will be assessed at Visit 2 and subjects using prohibitively high Ventolin usage as specified in the exclusion criteria will be screen-failed.

Demographic data and other characteristics will be recorded and will include the age and year of birth; gender, race, and/or ethnicity according to local regulations; alcohol consumption, and smoking history.

A standard medical medication, and surgical history will be obtained with review of the selection criteris with the subject.

# Randomization/treatment period

Procedures will be performed according to study assessments and procedures presented in

Table 1 and Table 2 for timed assessments.

Only Sponsor-provided IP and symptoms are a symptoms are a symptoms. Only Sponsor-provided IP administered QID and Ventolin prn to be used in response to asthma symptoms are allowed during the treatment period. IP should be taken in the morning upon waking, and then distributed equally throughout the day with the final dose taken before going to sleep. The evening before clinic visits, subjects should be advised to take the last dose at  $22:00 (10:00 \text{ PM}) \pm 2 \text{ hours}.$ 

At Visit 2 onwards, both IP and Sponsor-provided Ventolin should not be administered ≤6 hours prior to lung function testing (if Ventolin is needed within 6 hours of a study visit, either the entire visit must be rescheduled or just PFT assessment rescheduled).

At randomization (Visit 2), eligible subjects will enter a 12-week double-blind treatment period. The planned end-of-treatment will occur at Visit 6, the end of the 12-week treatment period.

## Dispensation of IP:

New IP will be dispensed to subjects at each visit where FEV<sub>1</sub> measurements are taken and the new IP should be used in advance of all post-dose measurements. To allow for proper preparation of IP, it is recommended that the seal around the study day treatment, look is opened 15 to 30 minutes prior to dosing and the instructions for administration of IP followed:

- After IP is primed and ready for use, provide assigned IP to subject
- Administer IP at the clinic
- Complete post-dose assessments

PT phicatio of any The study procedures carried out during this period will include: medical and surgical procedures, physical examination (includes weight a Visit 6 only), concomitant medications review, vital signs (heart rate, blood pressure only), 12-lead ECG at Visits 2 and 6, AEs, urine pregnancy test at Visits 2 and 4 (additionally, Visits 3 and 5 in the Czech Republic and also for the safety follow up visit in Argentina), serum pregnancy test at treatment discontinuation (Visit 6 or the PDV), blood samples for hemitology and clinical chemistry, spirometry, ACQ-5, ACQ-7, Asthma Quality of Life Question haire for 12 years and older (AQLQ+12)/Pediatric Asthma Quality of Life Questionnaire (PAQLQ), PEF, use of Ventolin therapy, asthma daytime/nighttime symptoms, night-time awakenings due to asthma symptom, dispensing/collecting eDiary, review compliance with Piary, dispensing and/or collection of IP, dispensing and/or collection of Ventolin, recording in eDiary of IP use, IP compliance, and randomization.

## Treatment discontinuation visit 4.3

Planned end of-treatment (EOT) will occur at Visit 6 (Week 12).

Procedures for planned EOT and PDV will assessments and procedures presented in Table 1.

The study procedures carried procedure Subjects who prematurely withdraw from study treatment (withdraw pre-week 12) will undergo a PDV. Procedures for planned EOT and PDV will be performed according to study

The study procedures carried out during the PDV visit will include: details of any surgical procedures will be recorded, physical examination (including weight), concomitant medications review, vital signs (heart rate, blood pressure only), 12-lead ECG, AEs, serum pregnancy test (at treatment discontinuation or PDV), blood samples for hematology and clinical chemistry, dispensation of IP (for spirometry only), dosing, spirometry, ACQ-5, ACQ-7,

AQLQ+12/PAQLQ, review of PEF, use of IP and Ventolin therapy, asthma daytime/night-time symptoms, night-time awakenings due to asthma symptoms, collecting eDiary, review compliance with eDiary, collection and final reconciliation of the IP and Ventolin, and IP

Conscheduled visit

Repeat assessments/visits, if needed, will be captured in unscheduled visits and the procedures uch application carried out during an unscheduled visit will be decided by the investigator.

4.5 Safety Follow-up period

Procedures will be performed according to study assessments and procedures procedures are discontinuation (Visit 6/FOCT). discontinuation (Visit 6/EOT or PDV).

The study procedures carried out during this period will include: recording of concomitant

medications and AEs.

5 STUDY ASSESSMENTS

The Rave WBDC system and the electronic patient reported outcome (ePRO; hereafter called eDiary) eDiary will be used for data collection and mery handling. The investigator will ensure that data are recorded on the eCRF and in accordance with the instructions provided.

The investigator ensures the accuracy completeness, and timeliness of the data recorded and of the provision of answers to data queries according to the Clinical Trial Agreement. The investigator will sign the completed CRF. A copy of the completed eCRF will be archived at the study site.

The laboratory safety assessments will be sent for analysis to a central laboratory.

The spirometry and ESG assessments will be performed at site using MasterScope equipment provided by eResearch Technology. The eDiary (AM3+) will be dispensed at screening which will also be used to collect PEF measurements, use of IP or Ventolin therapy, asthma unis, a tablet will be used to collect the AQLi transferred/reconciled with the eCRF data as summarized in Section 9.4.

Efficacy assessments

Efficacy assessments daytime/night-time symptoms, night-time awakenings due to asthma symptoms, ACQ-5, and ACQ-7 Pata. In addition to this, a tablet will be used to collect the AQLQ+12 data using the Stud Works software. This data will be recorded in the vendor's central database and

Efficacy assessments include spirometry, ACQ-7, AQLQ+12/PAQLQ, PEF, use of Ventolin therapy, asthma daytime/night-time symptoms, and night-time awakenings due to asthma symptoms.

## 5.1.1 Lung function measurement by spirometry

Lung function will be measured by spirometry at the study site using equipment provided by a central vendor. Spirometry will be performed by the investigator or authorized delegate

Subjects should not take Ventolin (or IP during 4).

Subjects should not take Ventolin (or IP during 4).

period but should also facilitate meeting the run-in FEV<sub>1</sub> and reversibility eligibility criteria.

Trough pre-dose and post-dose FEV<sub>1</sub> will be performed on a MasterScope provided for the study by the central reader at Visit 1 (screening), Visit 2 (baseline), and through Visit 6/PDV (endpoint measurements). For Visit 1/Visit 1a, pre- and post-dose measurements will be with respect to Sponsor-provided bronchodilator (Ventolin) and from Visit 2 onwards, will be with respect to IP.

It is important that all in-clinic dosing occurs progred 10:00 AM and that in-clinic dosing at Visits 3 through 6 is administered  $\pm 1$  hour in relation to the time of dosing at Visit 2.

Preferably, the same study personnel though test the subject's lung function throughout the study to reach optimal performance and to enhance reproducibility. The subject should rest at least 15 minutes prior to the test. For repeated measurements, eg, to assess best of at least 5, a pause of at least 1 minute between measurements is recommended.

The timing of FEV<sub>1</sub> assessment is presented in Table 3. Please note: the 5 minute post-IP dosing spirometry assessment. Visit 2 is crucial to accurately measure time of onset. The subject and site personnel should be adequately prepared for this assessment at the time of dosing.

The measurements are to be made with the subject seated in an upright position (preferably), or if not comfortable standing position is also acceptable. The same position should be used for all , measure artig the breathing thould be loosened.

Measurem spirometry measures during the entire study. The head must not be tilted during measurements. During the breathing maneuvers, the thorax should be able to move freely; hence tight clothing

Measurement procedures should be performed in accordance with the user manual for the study.

Timing of FEV<sub>1</sub> assessments

Visit 1: If a subject has not taken SABA or any bronchodilator ≤6 hours before lung function tests at Visit 1, they may proceed to pre-bronchodilator FEV<sub>1</sub> measurement and

reversibility eligibility assessments. If they have dosed with SABA or any bronchodilator ≤6 hours before study visit lung function tests, either the entire visit must be rescheduled or just PFT assessment rescheduled. Reversibility assessment will be performed in accordance with Section 5.1.1.1. Considerations for medications that may impact reversibility testing are stated in Section 7.8.2.

- Visit 2: Subjects should withhold administration of Sponsor-provided Ventolin or any bronchodilator for at least 6 hours before lung function tests at Visit 2. Trough pre-dose measurements should be taken at -60 and -30 minutes before administration of IP. Postdose measurements will commence at 5 minutes after administration of IP followed by measurements at all subsequent times as listed in Table 3. If a subject has taken Sponsor-provided Ventolin before Visit 2, either the entire visit must be rescheduted or just PFT assessment rescheduled.
- Visit 3 onwards: Subjects should withhold administration of Sponsor-provided Ventolin and IP for at least 6 hours before lung function tests at Visit 3 through 60h-clinic dosing will be administered prior to 10:00 AM and within 1 hour of the dosing at Visit 2. Trough pre-dose measurements should be taken at -60 and -30 minutes before administration of newly dispensed IP. Post-dose measurements will commence at minutes after administration of IP followed by measurements at all subsequent times as listed in Table 3. If a subject has taken IP or Sponsor-provided Ventolin before any on-treatment visit, either the entire visit must be rescheduled or just PFT assessment rescheduled.

Schedule of FEV<sub>1</sub> measurements at standard visits Table 3

| Timing of Spirometry Assessments | Assessment Window |
|---------------------------------------|-------------------|
| Pre- dose PFT -60 min | ±15 min |
| Pre- dose PFT -30 min | ±5 min |
| Post- dose PFT +5 min | ±2 min |
| Post- dose PFT +15 min | ±3 min |
| Post- dose PFT +30 min | ±5 min |
| Post- dose PFT +45 min X <sup>6</sup> | ±5 min |
| Post- dose PFT +60 mig | ±5 min |
| Post- dose PFT +120 min | ±10 min |
| Post- dose PFT + 180 min | ±10 min |
| Post- dose PF3 +240 min | ±10 min |
| Post- dose PFT +300 min | ±10 min |
| Post- do PFT +360 min | ±10 min |

Pre- and post- dose PFT measurements will be performed in relation to IP.

5.1.1.1 Reversibility test

To fulfill the reversibility. To fulfill the reversibility inclusion criterion, the increase in FEV<sub>1</sub> relative to baseline must be ≥15% approximately 30 minutes after inhalation of Sponsor-provided Ventolin.

Reversibility testing will be performed as follows:

Pre- and post- dose PFT measurements will be performed in relation to Ventolin at Visit 1, Visit 2 onward,

- 1. Perform pre-dose PFTs after at least 15 minutes of rest, and before administration of Ventolin.
- tension of such application 2. Subjects aged ≥12 years should administer 4 puffs of Ventolin. Subjects aged <12 years should administer 2 puffs of Ventolin.
- 3. Perform post-dose PFTs approximately 30 minutes after the administration of Ventolin.

## The reversibility is calculated as follows:

Reversibility=([Post FEV<sub>1</sub>-Pre FEV<sub>1</sub>]/Pre FEV<sub>1</sub>)X100

Pre-and post-dose FEV<sub>1</sub> measurements will be captured within the MasterScope. If the reversibility inclusion criterion is not met at Visit 1, the reversibility test may be repeated at Visit 1a prior to Visit 2 (randomization). Pre- and post-dose FEV<sub>1</sub> measurements are related to Sponsor-provided bronchodilator (Ventolin).

5.1.1.2 COVID-19 and Pulmonary Function Testing

In-clinic spirometry assessments should not be performed for objects exhibiting signs and symptoms for COVID-19. Any suspected prior or active cases should have a diagnostic test to confirm COVID-19 status. Any subjects with confirm COVID-19 should not perform spirometry assessments within 14 days of the station of symptoms and until the investigator considers the subject is no longer infectious. Device cleaning and hygiene guidance should be followed at all times.

5.1.2 Asthma Control Questionnaire-5

International guidelines for the treatment of asthma have identified that the primary clinical goal of asthma management is o optimize asthma control (minimization of symptoms, activity limitation, bronchoconstriction, and rescue  $\beta 2$  -agonist use) and thus reduce the risk of life-threatening exacerbations and long-term morbidity. The ACQ-5 (Appendix H, Asthma Control Questionnaire) was developed to meet these criteria. It measures both the adequacy of asthma control and change in asthma control, which occurs either spontaneously or as a result of treatment

The ACQ-5 will be administered using the eDiary during site visits as indicated in Table 1 Visits 1, 2, 3, 4, 5, 6, and PDV) and Table 2 for timed assessments at Visits 2, 4, 3, 5, 6, and PDV. The ACQ-5 self-administered adult version will be used for adults and adolescents aged 11 years and older. The Asthma Control Questionnaire-Interviewer-Administered [ACQ-IA] will be used for subjects aged <11 years; Section 5.1.4.

Subjects will be asked to complete the ACQ-5, consisting of 5 questions on symptom control; each of the questions will be scored on a 7-point scale (0=excellent asthma control; 6=extremely poor control). The questions take approximately 2 to 3 minutes to complete. Linguistically validated translations of the ACQ-5 into local languages will be used.

The ACQ-7 will be assessed at Visits 1, 2, 3, 4, 5, 6, and PDV and consists of the top scoring 5 symptoms from the ACQ-5 with 2 additional questions regarding FEV<sub>1</sub>% predicted value validated translations of the ACQ-7 into 1

## Asthma Control Questionnaire-Interviewer-Administered 5.1.4

The ACQ-IA version will be used for subjects aged <11 years and will be intervieweradministered (Appendix I, Asthma Control Questionnaire-Interviewer-Administered). Linguistically validated translations of the ACQ-IA into local languages will be used, with the results of the interviewer-administered version recorded into the eCRF.

## Asthma Quality of Life Questionnaire + 12/Pediatric Asthma Quality of Life Questionnaire 5.1.5 Life Questionnaire

# Asthma Quality of Life Question naise+12 5.1.5.1

The AQLQ+12 will be self-administered in all subjects aged ≥12 years using the eDiary during site visits as indicated in Table 1 and Table 2 for timed assessments at Visit 2 through Visit 6. Linguistically validated translations of the AQLQ+12 into local languages will be used.

The AQLQ was developed to measure the functional problems (physical, emotional, social, and occupational) that are most troublesome to adults with asthma Appendix F, Asthma Quality of Life +12 Questionnaire).

There are 32 questions in the AQLQ+12 and they are in 4 domains (symptoms, activity limitation, emotional function, and environmental stimuli). The activity domain contains 5 subject-species questions. This allows subjects to select 5 activities in which they are most limited and these activities will be assessed at each follow-up. Subjects are asked to think about how the Chave been during the previous 2 weeks and to respond to each of the 32 questions on a 7-point scale (7=not impaired at all; to 1=severely impaired). The overall AQLQ+12 score is the Hean of a second of this documents. mean of all 32 responses and the individual domain scores are the means of the items in those

## **Pediatric Asthma Quality of Life Questionnaire**

The PAQLQ will be self-administered during site visits as indicated in Table 1 and Table 2 for timed assessments at Visit 2 through Visit 6 in subjects aged 7 to 11 years. Responses to PAQLQ will be provided on paper and transcribed to the eCRF by site staff.

Subjects aged 4 to 6 years will complete the questionnaire with the help of a caregiver. The subject/caregiver will complete the PAQLQ on paper and responses will also be transcribed to the eCRF by site staff. As the PAQLQ is not validated for children <7 years of age, data for

Linguistically validated translations of the PAQLQ into local languages will be used. The PAQLQ has 23 questions in 3 domains (symptoms, activity limitation, and emotional function). The activity domain contains 3 subject-specific questions.

The PAQLQ, was developed to measure the functional problems (physical, emotional, and social) that are most troublesome to children with asthma (Appendix G, Pediatric Appendix Quality of Life Questionnaire).

social) that are most troublesome to children with asthma (Appendix G, Pediatric Appendix G, Pediatric Appendi

The eDiary will be utilized by all subjects enrolled in the study including children. Children, as necessary, will be assisted by a caregiver for the performance of assistments and navigation of the applicable questions.

5.1.6.1 Peak expiratory flow

Subjects will be trained at Visit 1. Throughout the study, subjects will record 3 PEF measures

on rising in the morning and before going to ted in the evening prior to taking any asthma therapy.

## eDiary investigational product use 5.1.6.2

Use of QID blinded IP will be colleged using the eDiary. Subjects will be asked in the evenings to enter into their eDiary (device, called AM3+), how many times they administered IP that day. The times of the administration and number of puffs will be recorded.

## eDiary Venton therapy use 5.1.6.3

Monitoring of Ventokin therapy in response to asthma symptoms use will be done only through the eDiary, where the number of Ventolin puffs taken in response to symptoms will be captured contact the investigator if their symptoms necessitate more than 8 puffs in a day.

The subject will use the above. twice daily (in the mornings and in the evenings). Sponsor-provided Ventolin will be dispensed

Subjects will be recommended not to take more than 8 puffs of Ventolin per day and advised to

The subject will use the eDiary for daily symptom reporting, entering symptoms twice daily.

The eDiary will be programmed to alert both the subject and study center when the below prespecified alert thresholds are crossed. Alerts will include:

- Decrease in morning peak flow  $\geq 20\%$  on at least 2 consecutive days compared with baseline, and/or
- Atension of such application An increase in rescue medication use of  $\geq 4$  puffs on at least 2 consecutive days compared with the average use during baseline, and/or
- >12 puffs of Ventolin in one day, and/or
- A night-time asthma symptom score of >baseline night-time score and  $\geq 2$  for at least 2 consecutive days, and/or
- A daytime asthma symptom score of 3 for at least 2 consecutive days
- >12 puffs of IP per day

The purpose of the alerts is to trigger a documented contact between the site and subject for further evaluation if deemed necessary by the investigator. The Sponsor will also receive programmed alerts to monitor subject follow-up. Alerts will include:

- Triggers in the eDiary will alert the subjects to signs of change of asthma and to contact their physician
- their physician

  A dedicated person from the Sponsor will review the ethary and compliance alerts (2 consecutive days of missing data) and contact the site
- Triggers in the eDiary will alert subjects in the eDiary will be ediary will alert subject possible sign of potential overdose
- , Qualified person from the site will contact the In case of eDiary or compliance aleres subject. For eDiary alerts, the subject asthma status should be evaluated, and it will be determined if a clinic visit is necessary

# An eDiary alert is not an astoma exacerbation per se.

Although the eDiary ale may initiate contact between the subject and the investigational site, the investigator or designee will always assess the subject's symptoms and determine whether to treat the subject for an exacerbation (Section 5.1.8).

Asthma symptoms should be captured in the eDiary by the subject every morning and evening.

# **Deterioration of asthma**

this study, deterioration of asthma is defined as 1 or more of the following items for ≥2 consecutive days:

- PEF: a decline of ≥20% from baseline
- Ventolin therapy use: >4 puffs/day and  $\geq 2 \times$  baseline
- Symptoms: night-time score that is >baseline and  $\geq 2$  OR a daytime score that is >baseline

and =3

Daytime is defined as the time period between the morning PEF assessment (upon rising in the morning) and the evening PEF assessment.

itation of extension of such application Night-time is defined as the time period between the evening PEF assessment (at bedtime) and the morning PEF assessment.

### 5.1.8 Asthma exacerbation definition

An asthma exacerbation is defined as deterioration of asthma which includes:

- Worsening of asthma signs/symptoms (Section 5.1.8.1)
- Increased use of 'as needed' reliever therapy
- Deterioration of lung function
- A medical intervention as described below (Section 5.1.8.3)

The worsening/onset of symptoms must include at least one of the following:

shortness of breath
wheezing
chest tightness
cough
sputum
night-time awakening due to asthma
activity limitation due to asthma
decreased PET These descriptions above are provided for definition, however, only savere asthma

- decreased PEF
- decreased FE

## Investigator justified asthma exacerbations 5.1.8.2

A vast majority of asthma exacerbations are associated with worsening of the symptoms or the symptoms

considered the overall clinical findings support the diagnosis of a severe asthma exacerbation (defined by required medical intervention as described in Section 5.1.8.3), but the symptomatic worsening does not meet the definition in Section 5.1.8.1 the investigator in justify the decision for defining the event as an exacerbation eCRF.

## 5.1.8.3 Severe asthma exacerbations

All protocol-defined severe asthma exacerbations need to fulfill the symptom criteria as defined in Section 5.1.8.1 and be supported by an eDiary alert or an investigator justification.

An asthma exacerbation will be considered **severe** if it results in at least 1 of the following:

- A temporary bolus/burst of SCS for at least 3 consecutive days to treat symptoms of asthmat worsening; a single depo-injectable dose of corticosteroids will be considered equivalent to a 3-day bolus/burst of SCS

  An emergency room or urgent care visit (1.7).
- in an emergency department or urgent care center) due to asthma that required \$\infty\$ the above)
- An in-patient hospitalization (defined as admission to an in-patient facility evaluation and treatment in a healthcare facility for ≥24 hours) due to asthma

## 5.1.8.4 Treatment for severe asthma exacerbations

The treatment for a **severe** asthma exacerbation is at least 3 consocutive days of SCS.

- The recommended treatment (GINA 2018) for a severe exacerbation is prednisolone (1 mg/kg/day up to 50 mg for adults and adolescence) once per day (preferably in the morning) for 5 to 7 days
- Tapering the prednisolone dose is not faced of the treatment has been given for <2 weeks (GINA 2018)

Treatment for <3 days does not constitute a severe asthma exacerbation, except if the subject is hospitalized due to asthma.

## Onset and duration of asthma exacerbations 5.1.8.5

For severe exacerbations, the duration is defined by the prescribed treatment.

For **severe** exacecoations:

- The stand date will be defined as the start date of prescribed treatment with a SCS
- The stop date will be defined as the last day of prescribed treatment with a SCS
- A single depot injectable dose of corticosteroids will be considered equivalent to a 3-day course of SCS. The corresponding stop date for this treatment will consequently be determined as the date of administration plus 2 days
- If multiple treatments are prescribed for the same exacerbation, the earliest start date and the latest stop date will be used
- For a severe asthma exacerbation requiring hospitalization with no documented corticosteroid treatment, hospitalization admission/discharge dates, or emergency visit date will be used as start/stop dates


## 5.1.8.6 Approach for capturing asthma exacerbations

## 5.1.8.6.1 Asthma exacerbation eCRF

If a severe asthma exacerbation requires hospitalization, the exacerbation should be reported as an SAE (Section 3.9) as well as on the Severe Asthma Exacerbation eCRF.

Severe asthma exacerbations will be considered study efficacy endpoints and will not be reported as AEs unless considered an SAE.

Safety assessment

reported as AEs unless considered an SAE.

5.2 Safety assessments

Safety assessments include clinical laboratory (hematology, chemistry, and pregnancy tests for females of childbearing potential) respectively 12.1 at 15.00 minutes. females of childbearing potential) parameters, 12-lead ECG readings, yital sign measurements, and collection of AEs.

5.2.1 Laboratory safety assessments

Blood samples for determination of clinical chemistry and hematology will be taken at the times indicated in Table 1 and Table 2 for timed assessments at Visit 2 through Visit 6.

Additional safety samples may be collected if chincally indicated at the discretion of the investigator.

Justry and hematology assessments will be performed under the street of characteristic visit 2 through the characteristic visit 2 through the character of the The clinical chemistry and hematology assessments will be performed using a centralized laboratory. Sample tubes and sample sizes may vary depending on laboratory method used and


Table 4 **Laboratory Safety Variables** 

| Hematology/Hemostasis (whole blood) | Clinical Chemistry (serum or plasma) |
|---|---|
| Red blood cells (erythrocytes) | Albumin |
| Hemoglobin | ALT |
| Hematocrit | ALP |
| Mean Corpuscular Hemoglobin | AST |
| Mean Corpuscular Hemoglobin Concentration | Bilirubin, total |
| Mean Corpuscular Volume | Calcium, total |
| White blood cells (leukocytes) | Chloride |
| Basophils (%) | Cholesterol, total |
| Basophils Abs | AST Bilirubin, total Calcium, total Chloride Cholesterol, total Creatinine Creatine kinase Gamma-glutamyl transportidase |
| Eosinophils (%) | Creatine kinase |
| Eosinophils Abs | |
| Lymphocytes (%) | Glucose (random) |
| Lymphocytes Abs | 0, |
| Monocytes (%) | Magnesium Phosphate |
| Monocytes Abs | |
| Neutrophils (%) | Protein, total |
| Neutrophils Abs | Sodium |
| Platelet count OR NOT | Triglycerides |
| Urine | Urea |
| Neutrophils (%) Neutrophils Abs Platelet count Urine Urine β-hCG pregnancy (at all other clinic visits, except Visit 1 and EOT or PDV) | Serum β-hCG pregnancy (Visit 1 and treatment discontinuation [EOT or PDV]) |

Abbreviations: Abs=absolute; ALP=alkaline phosphatase; ALT=alanine transaminase; AST=aspartate transaminase β-hCG=β-human chosonic gonadotropin; EOT=end-of-treatment; PDV premature discontinuation visit

If a subject shows an AST or ALT  $\geq$ 3× the upper limit of normal (ULN) and TBL  $\geq$ 2×ULN please refer to Section 3.9 and Appendix E, Hy's Law for further instructions.

# Resting 12-lead electrocardiogram

Twelve-lead ECGs will 'resting A 12 Lead ECG will be performed at the visits detailed in Table 1 and Table 2 for timed assessments at Visits 2, 6, and PDV. The timing and number of ECGs may be adjusted in

Twelve-lead ECGs will be obtained using a centralized laboratory after the subject has been resting semi supine for at least 10 minutes. All ECGs should be recorded with the subject in the same physical position. A standardized ECG machine should be used and the subject should be examined using the same machine throughout the study, where feasible.

After paper ECGs have been recorded, the investigator or designated physician will review each of the ECGs and may refer to a local cardiologist, if appropriate. A paper copy should be filed in the subject's medical records. If an abnormal ECG finding at screening/baseline is considered

Vital signs including resting pulse, and blood pressure, should be assessed at the visits detailed in Table 1 and Table 2 for timed assessments at Visit 2 and Visit 6. Measurements should taken in the sitting position after at least 10 minutes of rest.

Any clinically significant.

Any clinically significant changes in vital signs should be recorded as an AE if applicable.

5.2.4 Adverse event assessments

AEs will be collected from time of signature of informed consent/assent through to the follow-up period as described in Section 6

up period as described in Section 6.

5.3 Other assessments

5.3.1 Physical examination

A complete physical examination will be performed at screening (Visit 1), Visit 6, and PDV (if applicable) as detailed in Table 1. This will include an assessment of the following items: height in centimeters and BMI (both at Visit Von), weight, general appearance, respiratory system, cardiovascular system, abdomen, skin, bad and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeleta system (including spine and extremities), and neurological system.

# Concomitant medications 5.3.2

The collection and recording of all concomitant medications, including all pre-enrollment asthma therapies, will be performed at the visits detailed in Table 1. Permitted and restricted concomitant medications are described in Section 7.8.

All prescription drugs, herbal products, vitamins, minerals, and over-the-counter medications Subjects will taken within 3 months before screening (Visit 1) will be recorded as previous medications. All medications taken after screening and through the safety follow-up visit will be recorded as

Subjects will be maintained, after Visit 1, on IP and Ventolin to be used in response to asthma symptoms throughout the treatment period.

For restrictions relating to concomitant medications see Sections 3.1 and 3.2.

## 5.4 **Pharmacokinetics**

Not applicable.

## 5.5 **Pharmacodynamics**

Not applicable.

## 5.6 Genetics

Not applicable.

## 5.7 Biomarker analysis

Not applicable.

# istion of extension of such application SAFETY REPORTING AND MEDICAL MANAGEMENT 6

The investigator is responsible for ensuring that all staff involved in the study are familiar with the content of this section.

SAEs will be reported as per standard reporting guidance in sociated symptoms of asthma are considered as symptoms of disease under study and with not be recorded as AEs unless considered an SAE.

## Definition of adverse events 6.1

An AE is the development of any untoward medical occurrence in a subject or clinical study subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. A AE can therefore be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom (eg, nausea, chest pain), or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

The term AE is used to include both serious and non-serious AEs and can include a deterioration of a pre-existing medical occurrence. An AE may occur at any time, including the screening period, even if no IP has been administered.

# **Definitions of serious adverse event**

An SAE is an AE occurring during any study phase (ie, after the signing of the informed consent/assent through to the safety follow-up visit), that fulfills 1 or more of the following criteria:

- Results in death
- Is immediately life-threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization


- Results in persistent or significant disability or incapacity
- Is a congenital abnormality or birth defect
- extension of such application Is an important medical event that may jeopardize the subject or may require medical intervention to prevent 1 of the outcomes listed above

For further guidance on the definition of an SAE, see Appendix D, Additional safety information to the Clinical Study Protocol.

## 6.3 **Recording of adverse events**

## 6.3.1 Period for collection of adverse events

Adverse events and SAEs will be collected from time of signature of informed sonsent/assent, through the safety follow-up period.

## 6.3.2 Follow-up of unresolved adverse events

Any AEs that are unresolved at the subject's last assessment visit in the study are followed up by the investigator for as long as medically indicated, but without further recording in the eCRF. The Sponsor or a Safety and Pharmacovigilance Department representative retains the right to request additional information for any subject with ongoing AE(s)/SAE(s) at the end of the study (after the subject s final study visit) and capture that information in the eCRF, if judged necessary.

6.3.3 Variables

The following variables will be collected for each AE:

- AE (verbatim)

  The date when the AE started and stopped
- Maximum severity
- Seriousness
- Investigator ausality rating against the IP (yes or no)
- Action taken with regard to IP

• Date AE met criteria for SAE

• Date invest:

- Reason why the AE is considered serious
- Treatment given for the SAE
- Date of hospitalization 

57 of 142

- Date of discharge
- Probable cause of death
- Date of death
- Whether autopsy is performed
- Causality assessment in relation to study procedure(s)
- Causality assessment to other medication
- Description of AE

ansion of such application It is important to distinguish between serious and severe AEs. Severity is a measure of intensity whereas seriousness is defined by the criteria in Section 6.2. An AE of severe intensity need not necessarily be considered serious. For example, nausea that persists for several hours may be considered severe nausea, but not an SAE unless it meets the criteria shown in Section 6.2. On the other hand, a stroke that results in only a limited degree of disability may be considered a mild stroke but would be an SAE when it satisfies the criteria shown in Section 6.2.

The severity of the event should be assessed as mild, moderate, or severe.

6.3.4 Causality collection

The investigator and the Sponsor will assess causal relationship between IP and each AE, and answer 'yes' or 'no' to the question 'Do you consider that there is a reasonable possibility that the event may have been caused by the

For SAEs, causal relationship will also be assessed for other medication and study procedures. Note that for SAEs that could be associated with any study procedure the causal relationship is implied as 'yes'.

A guide to the interpretation of the causality question is found in Appendix D, Additional safety information of this Clinical Study Protocol.

## Adverse events based on signs and symptoms 6.3.5

All AEs spontaneously reported by the subject or care provider or reported in response to the open question from the study site staff: 'Have you/the child had any health problems since the previous visit/you were last asked?' or revealed by observation will be collected and recorded in the eCRF. When collecting AEs, the recording of diagnosis is preferred (when possible) over recording a list of signs and symptoms. However, if a diagnosis is known and there are other signs or symptoms that are not generally part of the diagnosis, the diagnosis and each sign or symptom will be recorded separately.

Asthma symptoms or signs, such as wheeze, cough, chest tightness, dyspnea, breathlessness, and phlegm, will be recorded as AEs only when:

- The sign or symptom is serious
- The subject discontinues IP due to the sign or symptom
- Such application The sign or symptom is new to the subject or not consistent with the subject's pre-existing asthma history (defined as within 1 year of Visit 1) as judged by the investigator

## 6.3.6 Adverse events based on examinations and tests

The results from the Clinical Study Protocol mandated laboratory tests, ECGs, vital signs, and other safety assessments will be summarized in the Clinical Study Report. Deterioration from baseline in these parameters should therefore only be reported as an AE if it fulfills way of the AE criteria or is the reason for discontinuation of treatment with the IP or is considered 'clinically significant'.

The criteria for determining whether the mandated laboratory tests, ECGs, vital signs, and other safety assessments are clinically significant and should be reported as AEs are generally:

- Test result is associated with accompanying symptoms or signs, and/or
- Test result requires additional diagnostic testing or medical/surgical intervention, and/or
- Test result leads to a change in study dosing of discontinuation from the study, significant additional concomitant drug treatment, or other oherapy, and/or
- Test result is considered to be an AE to the investigator or Sponsor.

If deterioration in a laboratory value, ECG, vital sign, or other safety assessment is associated with clinical signs and symptoms, the sign or symptom will be reported as an AE and the associated laboratory result/vital sign will be considered as additional information. Wherever possible, the reporting investigator uses the clinical, rather than the laboratory term (eg, anemia versus low hemoglobin value). In the absence of clinical signs or symptoms, clinically relevant deteriorations in non-mandated parameters should be reported as AE(s).

Any new or aggravated clinically relevant abnormal medical finding at a physical examination as compared with findings at the baseline assessment will be reported as an AE.

## Ą y's Law 6.3.7

Cases where a subject shows elevations in liver biochemistry may require further evaluation and occurrences of AST and/or ALT ≥3×ULN combined with TBL ≥2×ULN may require IP Aspension/discontinuation and study withdrawal, and may need to be reported as SAEs. Please refer to Section 3.9 and Appendix E, Hy's Law for further instruction on cases of increases in liver biochemistry and evaluation of Hy's Law.

## 6.3.8 **COVID-19 adverse events**

For subjects experiencing signs and symptoms indicating respiratory infection, confirmatory testing for COVID-19 is expected in line with national guidelines.


Non-serious confirmed COVID-19 AEs will be recorded within the clinical database but additional information may be collected within the safety database and/or narratives as required.

All SAEs in relation to COVID-19 shall be reported in line with the instructions for SAEON reporting described in Section 6.4.

Reporting of serious adverse events

All SAEs have to be reported.

All SAEs have to be reported.

All SAEs have to be reported.

reporting described in Section 6.4.

6.4 Reporting of serious adverse events

All SAEs have to be reported, whether or not considered causally related to the IP or to the study procedure(s). All SAEs will be recorded in the CDE study procedure(s). All SAEs will be recorded in the eCRF.

If any SAE occurs in the course of the study, then investigators of other site personnel should Safety and Pharmacovigilance Department within 1 day ie, immediately inform but no later than 24 hours of when he or she becomes aware of it.

Should the eCRF system become non-operational, walks shall be sent in paper form to:

Safety and Pharmacovi

Safety and Pharmacovigilance Department works with the investigator to ensure that all the necessary information is provided.

For fatal or life-threatening SAEs where important or relevant information is missing, active follow-up is undertaken immediately.

Investigator or other site personnel should inform the Safety and Pharmacovigilance Department of any follow-up information on a previously reported SAE ...think ca aware of it. within a calendar day ie, immediately, but no later than 24 hours of when he or she becomes

## **Overdose**

For the purpose of this study, an accidental or deliberate intake of blinded treatment of more than 12 puffs during one day is defined as an overdose and must be reported as such as described below.

All overdoses must be recorded on the Overdose/Medication Error eCRF. Any associated AEs should also be recorded as the AE diagnosis/symptoms on the relevant AE/SAE modules in the eCRF.

If an overdose occurs during the course of the study which has an associated SAE, then the investigator or other site personnel will inform the Safety and Pharmacovigilance Department immediately, or **no later than 24 hours** of when he or she becomes aware of the overdose. Safety and Pharmacovigilance Department works with the investigator to The ensure that all relevant information is provided to the Safety and Pharmacovigilance Department representative. For overdoses associated with an SAE, the standard SAE reporting timelines apply, see Section 6.4.

6.6 Pregnancy

All pregnancies and outcomes of the pregnancy should be reported to the and Pharmacovigilance Department representation. and Pharmacovigilance Department representative except the pregnancy is discovered before the study subject has received any IP.

6.6.1 Maternal exposure Maternal exposure If a subject becomes pregnant during the course of the study, IP should be discontinued immediately, 'Pregnancy' recorded as the reason for discontinuation on the eCRF, and the subject will be withdrawn from the stody. Pregnancy itself is not regarded as an AE unless there is a suspicion that the IP under study may have interfered with the effectiveness of a contraceptive medication. Congenital abnormalities/birth defeats and spontaneous miscarriages should be reported and handled as SAEs. Elective abortions without complications should not be handled as AEs. The outcome of all pregnancies (spontaneous miscarriage, elective termination, ectopic pregnancy, normal birth, or congenital amormality) should be followed up and documented even if the subject was discontinued from the study. If any pregnancy occurs in the course of the study, then the investigator or other site personnel Safety and Pharmacovigilance Department within 1 day ie, will inform the ammediately, but no later than 24 hours of when he or she becomes aware of it. Any conception occurring from the date of dosing through the safety follow-up visit should be reported. Safety and Pharmacovigilance Department will work with the investigator to ensure that all relevant information is provided.

The same timelines apply when outcome information is available.

## 6.6.2 Paternal exposure

sion of such application Pregnancy of a subject's partner is not considered to be an AE. However, any conception occurring from the date of dosing through the safety follow-up visit should be reported to the Safety and Pharmacovigilance Department representative and followed up for its

outcome.

## 6.7 **Medication error**

For the purposes of this clinical study, a medication error is an unintended failure or mistake in the treatment process for the Sponsor's IP that either causes harm to the subject or has the potential to cause harm to the subject.

A medication error is not lack of efficacy of the drug, but rather a humaror process related failure while the drug is in control of the study site staff or subject.

Medication error includes situations where an error:

- Occurred
- Was identified and intercepted before the subject received the drug
- Did not occur, but circumstances were recognized that could have led to an error

Examples of events to be reported in chinical studies as medication errors:

- Drug name confusion

  Dispensing error eg, medication prepared incorrectly, even if it was not actually given to the subject
- Drug not administration Drug not administration
- Drug not taken as indicated
- Drug now stored as instructed: eg, kept in the refrigerator when it should be at room temperature
- Wrong subject received the medication (excluding IWRS errors)

Wrong drug administered to subject (excluding IWRS errors)

Examples of events that **do not** require reporting as medication errors in clinical studies:

Errors related to or resulting from IWRS-including those which lead to 1 of the above listed events that would otherwise have been a medication error

- Accidental overdose (will be captured as an overdose)
- Subject failed to return unused medication or empty packaging
- Errors related to background medication, or standard of care medication in open-label

All medication errors must be recorded in the Overdose/Medication Error eCRF. Any city associated AEs should also be recorded as the AE diagnosis/symptoms on the relevant AE' modules in the eCRF.

If a medication error occurs during the he investigator or all

Pharmacovigilance Department immediately, or **no later than 24 hours** of when he or she becomes aware of the medication error.

Safety and Pharmacovigilance Department will work with the investigator to The ensure that all relevant information is provided to Safety and Pharmacovigilance Department representative. For medication errors associated with an SAE, the standard SAE reporting timelines apply, Section 6.4.

# Management of investigational product-related toxicities 6.8

In the absence of a specific antidote, pranagement of toxicities can be dealt with on the basis of the symptoms.

## INVESTIGATIONAL PRODUCT AND OTHER TREATMENTS 7

## Identity of investigational product(s) 7.1

BDA MDI is formed ated (Table 5) as both micronized budesonide and micronized albuterol co-suspended with spray-dried porous particles in a hydrofluoroalkane propellant. The co-suspension formulation ensures that subjects receive a consistent delivery of the drug from each actuation of the MDI.

Table 5 Investigational Product Strength and Dosage Form

| Investigational product name and dose | Product strength | Dosage Form/<br>Fill Count | Administration | Manufacturer |
|---|---|---|---|---|
| BDA MDI<br>80/180 μg | BDA MDI 40 µg budesonide and 90 µg albuterola per puff | MDI/120<br>actuations | Taken as 2 actuations | . 500 |
| BDA MDI<br>160/180 μg | BDA MDI<br>80 µg budesonide<br>and 90 µg<br>albuterol <sup>a</sup> per puff | MDI/120<br>actuations | Taken as 2 actuations | exemple of |
| BD MDI 160 μg | 80 μg budesonide<br>per puff | MDI/120 actuations | Taken as 2 actuations | |
| AS MDI 180 μg | AS MDI<br>90 μg albuterol<br>per puff <sup>a</sup> | MDI/120<br>actuations | Taken as 2 actuations | |
| Placebo MDI | 0 μg of active product <sup>b</sup> | MDI/120 actuations | Taken a02 actuations | |
| | Addition | al study medication | (Ventolia therapy) | |
| Ventolin HFA <sup>c</sup> | 108 μg albuterol<br>sulfate (90 μg<br>albuterol base) as<br>an aerosol<br>formulation | Albuterol (salbutamol) sulfate inhalation aeroso 200 puffs per capister | Ouring screening and (Section 5.1.1.1) as needed (generally 2 actuations per dose) during screening and treatment periods | |

Abbreviations: AS MDI=albuterol metered-dose inhaler; BD MDI=budesonide metered-dose inhaler; BDA MDI=budesonide/albuterol metered-dose in originary; HFA=hydrofluoroalkane.

Ventolin is a non-investigational medicinal product since it is taken as directed for reversibility testing (Visit 1 and repeat Visit 1a, if necessary) and as needed for symptoms during the screening period.

# Treatment groups include: BDA MDI 80/16 BDA N Dose and treatment regimens

BDA MDI 80/180 µg QID (given as 2 actuations of BDA MDI 40/90 µg per puff)

- BDA MDI 160/180 µg QID (given as 2 actuations of BDA MDI 80/90 µg per puff)
- BD MDI 160 µg QID (given as 2 actuations of BD MDI 80 µg per puff)
- AS MDI 180 µg QID (given as 2 actuations of AS MDI 90 µg per puff)
- Placebo MDI QID (given as 2 actuations)

<sup>&</sup>lt;sup>a</sup> Each puff contains 108 μg albute of sulfate corresponding to 90 μg albuterol base per actuation.

 $<sup>^{</sup>b}$  Each puff contains 183  $\mu g$  corous particles and 63  $\mu g$  of HFA-134a propellant made to be identical in appearance to BDA MDI, and AS MDI.

<sup>&</sup>lt;sup>c</sup> This table represents commercially available Ventolin formulation for the United States, each country participating in the Gudy will utilize commercially available Ventolin in that country, product strength may vary.

Randomization for adults and adolescents will be centralized and stratified by pre-study background therapy consisting of either ICS or non-ICS (subjects not previously treated with ICS), by ACQ-7 ( $\leq 1.5, >1.5$ ), and by age ( $\geq 12$  to 17,  $\geq 18$ ). Randomization for children aged 4

Handling and cleaning instructions for the MDI device will be available for the site to train subjects and also for the subjects to retain throughout the study (Appendix J, Meters Cleaning).

7.3 Labelling

Labelling

Labels will be prepared in accordance with Good Manufacturing Practice (GMP) and local regulatory guidelines. The labels will fulfill GMP Annex 13 requirements for labelling. Label text will be translated into local language.

The subject will receive a kit containing 2 MDI devices, individually wrapped in foil bags held within a carton. The MDI devices provided in this study and the packaging and labelling of the kits are visually identical to maintain the bling. A kee will be dispensed for every 15 days of treatment. Subjects will receive 2 kits at some

Each kit will contain the following brinded labels:

- Single panel canister label (English only)
- Single panel actuator label of multilanguage actuator booklet label
- MDI device shield label (single panel, English only)
- Foil bag label (single panel, English only) or multilanguage booklet label
- Single panel cacton label or multilanguage carton booklet label

The labels will include the following information:

- wame of Sponsor (Bond Avillion 2 Development LP Clinical Development Company: Avillion LLP)
- Investigational product dosage form, route of administration, and quantity of dosage units (blinded across all treatment groups)
- Storage conditions
- Study Trial Reference
- Medication ID number

- Directions for use
- The name of the investigator, where applicable (this will be added on the label manually or extension of such application when the IP is dispensed)
- The period of use eg, expiry date

The label will include the following standard statements:

- 'For clinical study use only' (or the required local statement)
- 'Keep out of reach of children'

## 7.4 Storage

Blinded supplies: BDA MDI 40/90 µg per puff, BDA MDI 80/90 µg per puff6BD MDI 80 µg per puff, AS MDI 90 μg per puff, and placebo should be stored below 25% (77°F) in a dry place. Excursions permitted up to 30°C (86°F).

Ventolin supplies: Store between 15°C and 25°C (59°F and 77°F). Store the inhaler with the mouthpiece down. For best results, the inhaler should be at room temperature before use. Do not use or store near heat or open flame. Exposure to temperatures above 120°F (49°C) may cause bursting. Never throw into a fire or incinerator. Temperature readings of the storage area (minimum/maximum) should be recorded one very working day at a minimum.

7.5 Compliance

The administration of all IPs will be captured in the subject's eDiary and not recorded in the eCRF, with the exception of the details of any interruptions for which the dates and reason for interruption will be recorded. The accountability will be recorded in the eCRF including the dose indicator readings for the returned kits. Data from the dose indicator will be compared with the subject's eDiary entriex and any discrepancies will be used to help in training the subject to accurately capture all IRadministration in the eDiary.

During the screening period, Ventolin usage will be reviewed to ensure the Study inclusion/exclusion criteria are adhered to. Ventolin will be dosed prn; therefore, compliance will not be applicable, other than the number of devices dispensed/returned and the usage being monitored.

# Accountability

The IPs provided for this study will be used only as directed in the Clinical Study Protocol.

All IPs will be returned to the approved study returns vendor for destruction after accountability and reconciliation is complete.

## 7.7 Metered-dose inhaler: handling and cleaning

Detailed handling instructions will be provided to the site in the form of a 'Site Manual' document, which will cover all aspects of the study with regards to IP. An 'Instructions For

Ine importance of the device cleaning and priming requirements should be emphasised to subjects. Priming of the IP MDI must occur. Device priming should not be conducted in theorem as spirometry assessments are being conducted.

7.8 Concomitant medications and a spirometry assessments are being conducted. same room as spirometry assessments are being conducted.

7.8 Concomitant medications and other treatments

7.8.1 Investigational product and Ventolin therapies

Only Sponsor-provided IP dosed QID and Sponsor-provided Ventolin therapy to be used in response to at these symmetric are all and the secondaries.

response to asthma symptoms are allowed during the study. No other asthma medications are allowed during the study.

Subjects on maintenance allergy immunotherapy (AIT) are allowed to continue their AIT; the new initiation of AIT during the study is not allowed

## Medications that may affect reversibility and FEV1 testing 7.8.2

Subjects are only eligible for enrollment on the DENALI study if they are taking SABA alone prn or with low-dose ICS; subjects presenting at Visit 1 being treated with any other asthma medication are ineligible. Therefore, the only restriction for eligible subjects' reversibility testing at Visit 1 (or 1A, if applicable) is the requirement not to take SABA (Visit 1) or Sponsor-provided Ventolin (Visic A) within 6 hours of lung function testing. At Visit 2 onwards, both IP and Sponsog provided Ventolin should not be administered within 6 hours prior to lung function testing

## Prohibited medications 7.8.3

Prohibited consemitant medications during the study include:

- Oral parenteral, or rectal corticosteroids (except if required to treat asthma exacerbation)
- Any other asthma medication except Sponsor-provided IP and Ventolin
  - Montelukast, for any indication
  - Inhaled disodium cromoglycate or inhaled nedocromil sodium
- 5-lipoxygenase inhibitors (ie, zileuton)
- Inhaled anticholinergies
- Phosphodiesterase inhibitors (ie, roflumilast)

- Omalizumab, benralizumab, mepolizumab, reslizumab, dupilumab or any other monoclonal or polyclonal antibody therapy for any reason (intra-ocular administration of monoclonal or polyclonal antibody therapy is allowed)
- extension of such application Beta2-adrenergic blockers including eye-drops (specific cardio-selective beta-blockers in low daily doses, eg, metoprolol in doses up to 100 mg/d, are allowed)
- Systemic treatment with potent cytochrome P450 3A4 inhibitors (eg, ketoconazole, itraconazole, and ritonavir)

## 8 STATISTICAL ANALYSES

## 8.1 Statistical considerations

All personnel involved with the analysis of the study will remain blinded until database lock

and identification of Clinical Study Protocol violators are identified.

Analyses will be performed by the Sponsor or its representatives.

The IDMC will have access to unblinded data in closed sessions with an unblinded statistician upon their request (see IDMC charter).

A comprehensive statistical analysis plan (SAP) will be represented prior to first subject randomized and any subsequent amendments will be documented with final arms. randomized and any subsequent amendments will be documented, with final amendments completed prior to the unblinding of the data.

8.1.1 Estimands

Two estimands are of interest in this study

The primary estimand of interest is the efficacy estimand, defined as the effect of the randomized treatment in all subjects assuming continuation of randomized treatment for the duration of the study, regardless of actual compliance. This estimand could be considered as a while-on-treatment strategy or a hypothetical strategy as defined in the draft International Conference on Harmonization (ICH) E9 Addendum.

The second estimand of interest is the attributable estimand, defined as the effect of treatment in subjects attributable to the randomized treatment. For this estimand, discontinuation of ... reatment for a re randomized treatment for reasons such as tolerability or lack of efficacy is considered a negative outcome. This estimand is a mixture of composite and hypothetical strategies as defined in the

# Sample size estimate

## **Initial assumptions and estimates**

A blinded sample size re-estimation was performed once 44% of subjects had completed Week 12. Based on the blinded estimate of variability, approximately 1000 subjects are required in order to demonstrate at least 90% power. Consequently, the total randomized adult and  68 of 142

adolescent subjects has been increased to 1000. This section details the initial assumptions of variability prior to calculating the blinded sample size re-estimation. Please refer to Section 8.2.2 for details on the sample size and power calculations following the blinded sample size re-estimation.

Prior to the blinded sample size re-estimation, randomization of approximately 120 subjects to each treatment group expected provide at least 93% probability to detect a 100 mL difference in the change from baseline in trough FEV<sub>1</sub> at Week 12 for comparison of BD MDI versus placebo MDI, BDA MDI versus placebo MDI, or BDA MDI versus AS MDI. This calculation was based on a standard deviation of 210 mL obtained from the placebo MDI group of Study PT008001 and an assumed dropout rate of 10% and 15% for active and placebo treatment group, respectively, prior to Week 12.

Prior to the blinded sample size re-estimation, it was assumed that the sample size of 120 subjects per treatment group would also provide >99% probability to detect a 130 mL difference in FEV<sub>1</sub> AUC<sub>0-6 hours</sub> over 12 weeks for comparison of BDA MDI versus BD MDI (effect sizes for AS MDI or BDA MDI versus placebo MDI should be considerably larger). This calculation assumed a 2% dropout prior to Week 1 and an effective standard deviation of 140 mL which was derived from the following: a per visit standard deviation of 200 mL (ProAir Respiclick Studies 301 and 304 and the AS MDI Dose-Ranging Study DC6930C00001), a correlation between visits of 65%, and projected subject completion of 4 out of 5 visits.

# 8.2.2 Blinded sample size re-extination

Following the blinded sample size re-estimation, randomization of approximately 200 subjects (≥18 years of age) to each treatment group will provide 90% probability to detect a 100 mL difference in the change from baseline in trough FEV₁ at Week 12 for comparison of BD MDI versus placebo MDI, BDA MDI versus placebo MDI, or BDA MDI versus AS MDI. This calculation is based on a standard deviation of 290 mL obtained from the blinded sample size re-estimation performed after 44% of subjects completed Week 12 and an estimated overall dropout rate of 11% prior to Week 12.

Following the Minded sample size re-estimation, the sample size of 200 subjects (≥18 years of age) per treatment group will also provide >99% probability to detect a 130 mL difference in FEV₁ Aloco over 12 weeks for comparison of BDA MDI versus BD MDI (effect sizes for AS MDI or BDA MDI versus placebo MDI should be considerably larger). This calculation assumes 2% dropout prior to Week 1 and an effective standard deviation of 290 mL obtained from the blinded sample size re-estimation performed after 44% of subjects completed Week 12.

Approximately 1000 adults (>10)

Approximately 1000 adults (≥18 years of age) and adolescent subjects (12 - 17 years of age, where approved) with asthma will be randomized 1:1:1:1:1 to 1 of 5 treatment groups (approximately 200 subjects per group: BDA MDI 80/180 μg QID, BDA MDI 160/180 μg QID, BD MDI 160 μg QID, AS MDI 180 μg QID, or placebo MDI). In addition, where approved, up

to 30 child subjects (aged 4 to 11 years) with asthma will be enrolled but will not receive high dose ICS and will be randomized 1:1:1 to receive low-dose BDA MDI 80/180 µg QID, AS MDI 180 µg QID, or placebo MDI. Approximately 2000 subjects will need to be screened, assuming

A second blinded sample size re-estimation will be performed once approximately 65% of the revised sample size has completed 12 weeks and prior to the last subject being randomized. This will allow the re-assessment of variability in a larger sample and at a point where any impact from COVID-19 with respect to lung function variability quantified more accurately. quantified more accurately. Final total enrollment in the study will be confirmed following the second blinded sample size re-calculation in order to ensure 90% power.

Any further potential increase in sample size will be capped at 1300, a 30% increase above the revised 1000 subjects.

8.3 Definitions of analysis sets

8.3.1 Full analysis set

The full analysis set is defined as all subjects who are replication.

The full analysis set is defined as all subjects who are randomized to treatment and take any amount of IP. Subjects will be analyzed according to the treatment they were assigned at randomization.

All efficacy analyses will be conducted on the full analysis set.

The efficacy and attributable estimated will include all data obtained before subjects discontinue randomized treatment.

## Safety analysis set 8.3.2

The safety analysis set a defined as all subjects receiving any amount of the IP. Subjects will be classified on the basis of treatment they actually received. If a subject receives >1 IP, he or she will be summarized according to the treatment the subject received the most. All safety summaries will be based on the safety analysis set.

Important protocol deviations will be listed and summarized by randomized treatment group. A

All subjects who failed any inclusion/exclusion criteria will failed criteria. This info All subjects who failed any inclusion/exclusion criteria will be listed along with details of the failed criteria. This information will also be summarized in terms of the number and percentage of subjects failing any of the inclusion/exclusion criteria and will be based on the full analysis set.

## 8.5 **Outcome measures for analyses**

## Primary efficacy analysis 8.5.1

The primary analysis will include all data obtained before subjects discontinue randomized treatment and will use the full analysis set, in accordance with the primary estimand (Section 8.1.1).

## 8.5.1.1 **Dual-primary efficacy endpoints**

The primary efficacy analysis comprises of 2 dual-primary endpoints of change from baseline in FEV<sub>1</sub> AUC<sub>0-6 hours</sub> over 12 weeks and change from baseline in trough FEV<sub>1</sub> at Week 12. Baseline FEV<sub>1</sub> will be taken as the average of the 60- and 30-minute pre-dose spirometry measures at randomization (Visit 2).

8.5.1.1.1 Derivation for FEV<sub>1</sub> AUC<sub>0-6 hours</sub>
FEV<sub>1</sub> AUC<sub>0-6 hours</sub> will be calculated for the changes from the baseline (randomization visit) using the trapezoidal rule and will be normalized by dividing by the time (in hours) from dosing

8.5.1.1.2 Derivation for trough FEV<sub>1</sub>

Trough FEV<sub>1</sub> will be taken as the average of the 60- and 30-minute pre-dose spirometry measures prior to dosing of IP.

In subjects with only 1 pre-dose assessment for trough, the value will be calculated from the single measurement.

single measurement.

## Secondary efficacy analyses 8.5.2

The secondary analyses will include all data obtained before subjects discontinue randomized treatment and will use the full analysis set, in accordance with the primary estimand (Section 8.1.1).

## Derivation for time to onset (15% increase in FEV<sub>1</sub>) on Day 1 and duration of 8.5.2.1 effect on Day 1

Time to onse (minutes) on Day 1 will be calculated as the time from dosing on Day 1 (randomization day; Visit 2) to the first instance within 30 minutes in which a percentage change from baseline in FEV<sub>1</sub> greater or equal to 15% is observed:

Sime of first 15% increase in percentage change from baseline in  $FEV_1$  – Time of dosing on Day 1 (randomization, Visit 2)

The duration of effect for each subject will be defined as the time from onset of at least a 15% increase in FEV1 to the offset of the 15% increase in FEV1 relative to baseline. If the offset of response was not achieved during the assessment period, the last available time of assessment will be used as the offset. If a subject had a second onset of response subsequent to achievement of offset, their data for that subsequent period will be excluded from the duration of response calculation.

The minimal important difference (MID) in ACQ-7 score is estimated to be 0.5 (Juniper 2005). On the basis of the MID, responders at Week 12 are defined as subjects achieving a decline from baseline of at least 0.5: On the basis of the MID, responders at Week 12 are defined as subjects achieving a decline from baseline of at least 0.5:

• Responder: (Week 12 – baseline) ≤-0.5

• Non-responder: (Week 12 – baseline) >-0.5

Subjects who discontinue treatment for any reason before Week 12 will be classified as non-

responders. Baseline is defined as the most recent non-missing score before the first dose of randomized IP.

Additionally, an exploratory endpoint will be considered to sixess the changes from baseline ACQ-7 overall score at Week 12 as the following 3 devel factor:

- Improvement: (Week 12 baseline)
- No Change: -0.5 < (Week 12 1)
- Worsening: (Week 12 baseline № 0.5

Subjects who discontinue treatment for any reason before Week 12 will be classified as nonresponders.

The interviewer-administered version will be implemented for children aged 4 to 10 years. As the ACQ-7 is not validated for children <6 years old, data for subjects who are 4 or 5 years of age will be excluded from the analyses of ACQ-7 endpoints.

## Exploratory efficacy analyses 8.5.3

Athrent and v (Section 8.1.1).

This docume 8.5.3.1 The exploratory analyses will include all data obtained before subjects discontinue randomized treatment and will use the full analysis set, in accordance with the primary estimand

## **Derivation of severe exacerbation endpoints**

For the production of summary statistics, the raw annualized severe asthma exacerbation rate will be calculated according to the following formula:

Annualized severe exacerbation rate= $\sum$  number of severe exacerbations\*365.25/ $\sum$  follow-up, where the summations are over all subjects within a treatment group.  72 of 142
For subjects who do not prematurely discontinue, the *follow-up* is calculated as:

Date of latest follow-up-date of randomization (Visit 2) + 1.

Otherwise, follow-up is calculated as the discontinuation date of randomized treatment:

Date of randomized treatment discontinuation-date of randomization (Visit 2) + 1.

### 8.5.3.2 **Derivation of deterioration of asthma variables**

of such application The deterioration of asthma rate will be calculated in a similar way as the raw annualized severe asthma exacerbation rate (Section 8.5.3.1).

8.5.3.3 Derivation of peak FEV1

Peak change from baseline in FEV1 will be calculated using the largest FEX value measured following dosing of IP.

8.5.3.4 Derivation of peak expiratory flow

The best of at least 3 PEF measurements will be recorded by the subject in the marring and

The best of at least 3 PEF measurements will be recorded by the subject in the morning and before going to bed in the evening prior to taking any asthma therapy. PEF will be analyzed separately for the morning and evening.

# Derivation of Asthma Control Questionnaire-5 variables 8.5.3.5

Derivations for responder status for ACO 5 will be performed as described in Section 8.5.3.2. At least 4 out of the 5 symptom items are needed to provide an overall ACQ-5 score.

## Derivation of Asthma Quality of Life Questionnaire +12 and Pediatric Asthma 8.5.3.6 Quality of Life Questionnaire variables

AQLQ consists of 32 questions in 4 domains and PAQLQ consists of 23 questions in 3 domains. Both are assessed on separate 7-point Likert scales from 1 to 7, with higher values indicating better health celated quality of life.

For overall health related quality of life and for each of the domains, the MID has been determined to be a change in score of 0.5 (Juniper 1994). On the basis of the MID, responders at Week 12 and defined as subjects achieving an increase from baseline of at least 0.5:

Kesponder: (Week 12 – baseline) ≥0.5

Non-responder: (Week 12 – baseline) < 0.5

Subjects who discontinue treatment before Week 12 for any reason will be classified as nonresponders. Baseline is defined as the most recent non-missing score before the first dose of randomized IP.

### 8.5.3.7 **Derivation of Ventolin therapy variables**

Ventolin therapy will be analyzed through the average number of administrations (puffs) per day.

Total daily number of puffs will be further characterized within 4-weekly time intervals of throughout the randomized treatment period. Further details will be provided in the SAP.

Baseline number of puffs per day will be based on the last 10 before the first dose of randomized IP

### 8.5.3.8 Derivation of other eDiary variables

# **Symptom-free days**

A symptom-free day is defined as the fulfillment of both of the following criteria:

- A day and night with no asthma symptoms (e, sthma symptom score=0)
- A night with no awakenings due to as thing symptoms

# Asthma control days

An asthma control day is defined as the fulfillment of all of the following criteria:

- A day and night with no aschma symptoms (ie, asthma symptom score=0)
- A night with no awakenings due to asthma symptoms
- A day and night with no use of prn Ventolin therapy

### Methods for statistical analyses 8.6

All tests will be 2-sided and at 5% level of significance unless otherwise stated.

addition to the a where appropriate.

8.6.1 In addition to the analyses described below, all variables will be summarized descriptively

# Analysis of the dual-primary variable

The first and second dual-primary variables, change from baseline in FEV<sub>1</sub> AUC<sub>0-6 hours</sub>, and change from baseline in trough FEV<sub>1</sub> will each be analyzed using a repeated measures (RM) linear model to compare treatment groups. The model will include baseline FEV<sub>1</sub>, percentage reversibility to Ventolin, and age as continuous covariates, and visit, treatment, the treatmentby-visit interaction, and prior ICS use (Yes/No) as categorical covariates. Baseline will be defined as the average of the pre-dose assessments collected on randomization (Visit 2).

P-values and point estimates with two-sided 95% confidence intervals will be calculated for each pairwise treatment contrast. More details will be provided in the SAP.

The planned treatment comparisons for the primary analysis will 18 step sequence as specified below. Coccurs All

occurs. All comparisons are of superiority. Formally, the null and alternative hypotheses for each comparison are:

 $H_0$ :Difference between treatment =0,

HA: Difference between treatment

Change from baseline in FEV<sub>1</sub> AUC<sub>0-6 hours</sub> over 12

- 1. AS MDI 180 μg QID versus placebo MDI
- 2. BDA MDI 160/180 μg QID versus
- 3. BDA MDI 160/180 μg QID versas BD MDI 160 μg

Change from baseline in trough FEV1 at Week 12:

- 4. BD MDI 160 μg QID versus placebo MDI QID
- 5. BDA MDI 160/\$20 μg QID versus placebo MDI QID
- 6. BDA MD 160/180  $\mu g$  QID versus AS MDI 180  $\mu g$  QID

Change from baseline in trough FEV<sub>1</sub> at Week 12:

7. BDA MDI 80/180 μg QID

8. PP Statistical testing for BDA 80/180 μg will proceed in a similar manner as for BDA 160/180 μg,

- 7. BDA MDI 80/180 µg QID versus placebo MDI QID
- 8. BDA MDI 80/180 μg QID versus AS MDI 180 μg QID

The Type I error will be controlled sequentially by testing in the above order. If a comparison is significant (alpha=0.05, two-sided), testing will proceed to the next comparison.

The above tests in steps 1 to 8 will exclude children (age 4 to 11 years). The analysis will be repeated to include children, but will be considered a supportive analysis of the dual-primary endpoint. In the supportive analysis including all ages, the comparison of BDA MDI 160/180 µg versus AS MDI 180 µg will exclude the child subjects aged 4 to 11 years as they will not be randomized to BDA MDI 160/180 µg. However, the comparison of BDA MDI 80/180 µg versus AS MDI 180 µg and BDA MDI 80/180 µg versus placebo MDI will include subjects from all age groups.

The comparisons of BDA MDI  $80/180~\mu g$  QID versus placebo MDI QID and BDA MDI  $80/180~\mu g$  QID versus BD MDI  $160~\mu g$  QID for FEV<sub>1</sub> AUC<sub>0-6 hours</sub> over 12 weeks are not included in the Type I error control procedure as they redundantly evaluate the contribution of abuterol to the combination, which is already captured in Steps 2 and 3. However, these comparisons will be reported for completeness.

All subjects who are randomized and are part of the full analysis set will be analyzed according to the strata they were allocated to in IVRS/IWRS in this primary analysis. A sensitivity analysis will be conducted based on subjects' actual strata to assess the impact of miss-stratification on the model results.

# 8.6.2 Analysis of the secondary efficacy ariables

For all secondary analyses the same treatment control arisons as for the primary analysis will be conducted (Section 8.6.1).

# 8.6.2.1 Median time to onset (15% increase in FEV<sub>1</sub>) and duration of effect

The median time to onset (defined as 3% increase in FEV<sub>1</sub>) over the pre-treatment value at randomization (Visit 2) will be corepared among treatment groups using a Wilcoxon rank sum test. Confidence intervals for the median treatment difference will be calculated using the Hodges-Lehmann method.

Descriptive statistics for duration of response will be reported by treatment group.

Only the subjects who achieve the 15% increase in FEV<sub>1</sub> within 30 minutes post-dose will be included in these calculations.

# 8.6.2.2 Asthma Control Questionnaire-7

The frimary analyses of ACQ-7 will be conducted in subjects that are uncontrolled at baseline  $ACQ-7 \ge 1.5$ ) as these are the subjects capable of demonstrating a clinically meaningful response with treatment.

The responder variable described in Section 8.5.2.2 at Week 12 will be analyzed using a logistic regression model with treatment and previous ICS use (Yes/No) as categorical covariates, and baseline ACQ-7 score, baseline post-dose percent predicted FEV<sub>1</sub> and age as continuous

covariates. From the logistic regression model treatment effects will be estimated by odds ratios and its corresponding 95% confidence interval along with p-values.

The treatment effect for change from baseline in ACQ-7 will be estimated using a mixed model. RM (MMRM) analysis. All data up to Week 12 will be included in the model, with terms for baseline post-dose percent predicts 1 Feet warriers. variance-covariance matrix will be assumed to be unstructured. If the procedure does not converge, then a heterogeneous TOEPH will be used instead. This model will be used to give an overall assessment of the treatment effect as well as 95% confidence intervals.

Change from baseline will also be described descriptively for all study visits.

The safety analyses will include all data obtained before subjects discontinue randomized treatment and will use the safety analysis set.

8.6.3.1 Adverse events

Adverse events will be summarized before subjects discontinue randomized treatment and will use the safety analysis set.

Adverse events will be summarized by treatment group, system organ class and preferred term assigned to the event by the Medical Dictionary for Regulatory Activities. AEs will also be listed for each subject.

### 8.6.3.2 Vital signs

Change from baseline throughout the study will be assessed for vital signs variables collected on the eCRF.

Baseline is defined as the most recent non-missing measurement before the first dose of randomized IPS

# 8.6.3.3 Clinical chemistry and hematology

Clinical chemistry and hematology parameters will be summarized by treatment group and Visit and will also be listed by subject.

Baseline is defined as the most recent non-missing measurement before the first dose of randomized IP.

### 8.6.3.4 Electrocardiogram

ECG parameters will be summarized by treatment group and Visit and will also be listed by subject.


Baseline is defined as the most recent non-missing measurement before the first dose of randomized IP.

Analysis of exploratory variables

The treatment comparisons in the secondary analyses given below are compared in the same way as the primary analysis.

8.6.4.1 Severe exacerbations

The raw annualized exacerbation rate will be lerivation described in Section 1.

Deterioration of asthma

Annualized deterioration of asthma will be summarized in the same way as the annualized severe asthma exacerbation rate (Section 8.6.4.1)

8.6.4.3 Peak FEV1

Peak FEV1 at Day 1 (Visit 2) and Day Prince of the same way as the annualized rough FEV1 and FFV Peak FEV<sub>1</sub> at Day 1 (Visit 2) and Day (Visit 3) will be analyzed using the same method as for trough  $FEV_1$  and  $FEV_1$  AUC<sub>0-6 hours</sub>. Baseline will be defined as the average of the pre-dose assessments collected on Day 1.

# Peak expiratory flow 8.6.4.4

The mean value of change from baseline in PEF data during the randomized treatment period will be analyzed by analysis of covariance with treatment, ACQ-7 at randomization ( $\leq 1.5 > 1.5$ ), and prior ICS use (Yes No) as factors, and age and baseline PEF score as continuous covariates. The summary measure for the comparison of treatments will be the estimated mean difference, presented with the corresponding 95% confidence interval.

Additionally, an RM analysis will be conducted and will be partitioned into 4-weekly time intervals across the randomized treatment period. The analysis model will additionally include time point and treatment\*time point as factors.

### 8.6.4.5 Asthma Control Questionnaire-5 variables

The responder variable for ACQ-5 at Week 12 will be analyzed using a logistic regression model in the same way as ACQ-7 (Section 8.6.2.2).

The treatment effect for change from baseline in ACQ-5 will be estimated using an MMRM analysis in the same way as ACQ-7 (Section 8.6.2.2).


78 of 142

The 3-factor categorization of ACQ-7 (Improvement; No change; Worsening) will be considered in an exploratory analysis using a logistic regression model adjusted for the same covariates as for the binary response of ACQ-7 (Section 8.6.2.2).

The domain scores as well as the overall scores are calculated from the unweighted arithmetic means of the individual question scores. The treatment effect for change from baseline in AQLQ+12 and PAQLQ overall scores up to Week 12 will be estimate. ACQ-5, using an MMRM analysis.

Change from baseline will also be described descriptively for all study visits for each of the domains and the overall scores domains and the overall scores.

In all the scenarios above, baseline is defined as the most recent non-missing measurement before the first dose of randomized IP.

As the PAQLQ is not validated for children <7 years of age, data for subjects who are aged 4 to 6 years will be excluded from the analyses of PAQLQ endpoints.

8.6.4.7 Ventolin therapy

Change from baseline in Ventolin therapy use compared with the mean value of available data during the study. The data will be analyzed using analysis of covariance with treatment, ACQ-7 at randomization (≤1.5/>1.5), and prigrifCS use (Yes/No) as factors, and age and baseline daily number of puffs as continuous covariates. The summary measure for the comparison of treatments will be the estimated mean difference, presented with the corresponding 95% confidence interval.

Additionally, an RM analysis will be conducted on the change from baseline Ventolin therapy partitioned into 4-weekly time intervals across the randomized treatment period. The analysis model will additionally include time point and treatment\*time point as factors.

# 8.6.4.8 Other eDiary variables

Asthma daytime/night-time symptoms and night-time awakenings due to asthma will be compared with the mean value of available data during the study. The data will be analyzed Sing analysis of covariance with treatment, ACQ-7 at randomization ( $\leq 1.5/>1.5$ ), and prior ICS use (Yes/No) as factors, and age and baseline as continuous covariates. The summary measure for the comparison of treatments will be the estimated mean difference, presented with the corresponding 95% confidence interval.

Additionally, an RM analysis will be conducted on the aforementioned eDiary endpoints, partitioned into 4-weekly time intervals across the randomized treatment period. The analysis model will additionally include time point and treatment\*time point as factors.

Subgroup analysis

The assessment of treatment effect will also be investigated in the stratification variables and other clinically important subgroups and will be defined in more detail in the SAP.

8.6.6 Interim analysis

No interim analyses will be conducted.

all subjects have completed the treatment period and until after the database has been locked.

8.6.7 Sensitivity analysis

8.6.7.1 Tipping point analysis

Multiple imputations tipping point analysis under the massing not at random assumption (MNAR) will be conducted. For subjects in the BDQ MDI groups, and subjects in AS MDI and BD MDI when comparing to placebo MDIChis method will impute missing values post-study discontinuation for lack of asthma control assuming they were more likely to have a worse outcome than as implied under the missing at random assumption (MAR). The tipping point analysis will incrementally penalize the missing data under the missing not at random assumption until a non-statistically significant comparison is observed.

The tipping point approach described above will be repeated and all missing data over the randomized treatment period will be imputed under the MNAR assumption. Further details will be provided in the SAR

## Attributable estimand 8.6.7.2

Analysis of the attributable estimand will be conducted in the full analysis set, but data that are missing to treatment discontinuation will be imputed based on the 95th or the 5th percentile of the eference group's distribution if the reason is reasonably attributable to tolerability or lack of efficacy. The 95th percentile would apply to an endpoint for which a higher value is a worse Outcome, while the 5th percentile would apply to an endpoint for which a higher value is a better outcome. More detail about the computation of the attributable estimand will be provided in the SAP.

# 8.6.7.3 COVID-19 pandemic impacts

As the trial is ongoing during the coronavirus disease (COVID-19) pandemic, it will be necessary to evaluate any potential intercurrent events due to COVID-19 and quantify their impact on the efficacy and safety profile of the study.

At a minimum, the number of missed visits, premature withdrawals, and efficacy assessments not done will be summarized descriptively by treatment group and overall across treatment groups. Where appropriate, the subject level data for missed visits and assessments will listed along with the corresponding link to COVID-19, as recorded in the eCRF. It is not anticipated that missing data and premature withdrawals due to COVID-19 will be related to randomized treatment. Therefore, missing data due to COVID-19 will be assumed missing at random in accordance with the efficacy estimand. If further sensitivity analyses are deemed necessary following a blinded review of missing efficacy due to COVID-19, further details will be provided in the statistical analysis plan, prior database lock and unblinding.

Similarly, at a minimum, the number of missed scheduled safety assessments due to COVID-19 will be summarized descriptively by treatment group and across treatment groups. Subjects with suspected or confirmed diagnosis of COVID-19, and/or COVID-19 related AEs and SAEs will be summarized descriptively. Subject level listings of missed safety assessments and COVID-19 related (S)AEs will be listed.

# 9 STUDY AND DATA MANAGEMENT

# 9.1 Training of study site staff

Before the first subject is entered into the study, a designated representative will review and discuss the requirements of the Chaical Study Protocol and related documents with the investigational staff and also train them in any study specific procedures and the Rave WBDC system(s) utilized.

The investigator will ensure that appropriate training relevant to the study is given to all of these staff, and that any new information relevant to the performance of this study is forwarded to the staff involved.

The investigator will maintain a record of all individuals involved in the study (medical, nursing, and other staff).

# Monitoring of the study

During the study, the Sponsor or a designated representative will have regular contacts with the study site, including visits to:

- Provide information and support to the investigator(s)
- Confirm that facilities remain acceptable

- Confirm that the investigational team is adhering to the Clinical Study Protocol, that data are being accurately and timely recorded in the eCRFs, that biological samples are handled in accordance with the Laboratory Manual, and that IP accountability checks are being
- including verification of informed consent/assent of participating subjects. This will required direct access to all original records for each subject (eg, clinic charts)

  Ensure all SAEs and AEs have been captured and remains subject safety while on attal.
- Verify the correct storage, handling, dispensation, and return of all IP
- Ensure withdrawal of informed consent/assent to the use of the subject biological samples is reported and biological samples are identified and disposed of/destroyed accordingly, and the action is documented, and reported to the subject

The designated representative will be available between visits of the investigator(s) or other staff at the center needs information and advice about the conduct of the study.

### 9.2.1 Source data

Source documents provide evidence for the existence of the subject and substantiate the integrity of the data collected. Source coursents are filed at the investigator's site.

Data entered in the eCRF that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records. Also, current medical records must be available.

Definition of what constitutes source data can be found in the Source Data Agreement, agreed with each investigator before site initiation.

### 9.2.2 Study agreements

The investigator/participating center should comply with all the terms, conditions, and obligations of the Clinical Study Protocol, or equivalent, for this study.

Clinical Trial Agreements with the investigator/participating center should be in place before any study-related procedures can take place, or subjects are enrolled.

### 9.2.3 **Archiving of study documents**

The investigator follows the principles outlined in the Clinical Trial Agreement.


### 9.3 Study timetable and end-of-study

The end-of-study is defined as 'the last visit of the last subject undergoing the study'.

asion of such application The study may be terminated at individual centers if the study procedures are not being performed according to Good Clinical Practice (GCP), or if recruitment is slow. The Sponsor may also terminate the entire study prematurely if concerns for safety arise within this study or in any other study with BDA MDI.

### 9.4 Data management

Data management will be performed by the Data Management Team at according to the Data Management Plan.

The data collected through third party sources will be obtained and reconciled against study data. Data from third parties will be transferred in accordance with data wansfer specifications and reconciled in accordance with the Data Management Plan.

AEs and medical/surgical history will be classified according to the terminology of the latest version of the Medical Dictionary for Regulatory Activities at the time of database lock. Medications will be classified according to the World Health Organization Drug Dictionary. All coding will be performed by the Medical Coding Team at

Data queries will be raised for inconsistent, impossible, or missing data. All entries to the study database will be available in an audit wall

The data will be validated as defined in the Data Management Plan. Quality control procedures will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. The Data Management Plan will also clarify the roles and responsibilities of the various functions and Bersonnel involved in the data management process.

# Serious adverse event@econciliation

SAE reconciliation reports are produced and reconciled with the applicable Safety and Pharmacovigilance Department safety database and/or the investigational site.

# Management of external data

Data Management will set up import agreements with third party data sources, to ensure external data is integrated in line with applicable data standards.

external data

Final database lock

Database loc'

L Database lock will occur once 'the last visit of the last subject participating in the study has been completed' all data have been coded, validated, signed, and locked, and clean file has been declared.

### 10 ETHICAL AND REGULATORY REQUIREMENTS

### 10.1 **Ethical conduct of the study**

Subject data protection

The informed consent/assent form will incorporate (or, in some cases, be accompanied and a separate document incorporating) wording that complies with relevant data protection privacy legislation.

Subjects will be assigned a unique identification of the protection of the pr

that are transferred to the Sponsor will contain the identifier only; subject names or any information which would make the subject identifiable will not be transferred. Subjects must be informed that his/her personal study-related data will be used by the Sponsor in accordance with local data protection law. The level of disclosure must also be explained to the subject. Subjects must also be informed that his/her medical records may be examined by study monitors, clinical quality assurance auditors, or other authorized personne appointed by the Sponsor, by appropriate EC members, and by inspectors from regulatory authorities.

# Ethics and regulatory review 10.3

An EC should approve the final Clinical Study Protocol, including the final version of the informed consent/assent form and any other written information and/or materials to be provided to the subjects. The investigator will ensure the distribution of these documents to the applicable EC and to the study site staff.

The opinion of the EC should be given in writing. The investigator should submit the written approval to the Sponsor or designated representative before enrollment of any subject into the

The EC should approve all advertising used to recruit subjects for the study.

The Sponsor or designated representative should approve any modifications to the informed consent/assent form that are needed to meet local requirements.

If required by local regulations, the Clinical Study Protocol should be re-approved by the EC annually.

Before enrollment of any subject into the study, the final Clinical Study Protocol, including the final version of the informed consent/assent form, is approved by the national regulatory authority or a notification to the national regulatory authority is done, according to local regulations.

The Sponsor or designated representative handles the distribution of any of these documents to the national regulatory authorities.

The Sponsor or designated representative will provide regulatory authorities, ECs, and investigators with safety updates/reports according to local requirements.

### 10.4 Informed consent/assent

The investigator(s) at each center will:

- ion of such application Ensure each subject and/or parent/legal representative (as applicable) is given full and adequate oral and written information about the nature, purpose, possible risks and benefit of the study
- Ensure each subject and/or parent/legal representative is notified that they discontinue from the study at any time
- Ensure that each subject and/or parent/legal representative is given the opportunity to ask questions and allowed time to consider the information provided
- Ensure each subject and/or parent/legal representative provides signed and dated informed consent/assent before conducting any procedure specifically for the study
- Ensure the original, signed informed consent assent form(s) is/are stored in the investigator's study file
- Ensure a copy of the signed informed consent/assent form is given to the subject
- Ensure that any incentives for subjects who participate in the study as well as any provisions for subjects harmed as a consequence of study participation are described in the informed consent/assent form that is approved by an EC

# Changes to the clinical study protocol and informed consent/assent 10.5

Study procedures will not be changed without the mutual agreement of the international coordinating in estigator and the Sponsor.

If there are any substantial changes to the Clinical Study Protocol, then these changes will be documented in a new version of the study protocol.

The new version of the Clinical Study Protocol is to be approved by the relevant EC and if applicable, also the national regulatory authority, before implementation. Local requirements are to be followed for new versions of Clinical Study Protocols.

The Sponsor will distribute any new versions of the Clinical Study Protocol to each investigator(s) for distribution to EC see Section 10.3.

If a change to a Clinical Study Protocol requires a change to a center's informed consent/assent form, the Sponsor and the center's EC are to approve (or a notification to the national regulatory authority is submitted where applicable for) the revised informed consent/assent form before the

Authorized representatives of the Sponsor, a regulatory authority, or an EC may perform audits of inspections at the center, including source data verification. The purpose of an audit or inspection is to systematically and independently examine all of the documents to determine whether the analyzed and accurately reported according to the Clinical Study Protocol, GCP, Riddelines of the ICH, and any applicable regulatory requirements. The investigator will contact the Sponsor immediately if contacted by a regulatory agency about an inspection at the center.

SUMMARY OF CHANGES

The following table provides a brief summary of major changes at does not include all nonsubstantial changes (eg, formatting, minor clerical, and typographical corrections).

### Changes to protocol amendment 2 11.1

| <b>Section</b> | Changes to Protocol Amendment 2 (Version 3.0) |
|---|---|
| Clinical Protocol Synopsis | Updated the number of adult and adolescent subjects pardomized from 600 to 1000, the number of subjects within each treatment arm from 120 to 200, and the number of subjects screened from 1000 to 2000. Updated the estimated screen failure rate from 40% to 50%. |
| ent must not be used to support any s | Exploratory endpoint: Specified that the change from baseline in the Asthma Control Questionaire-5 (ACQ-5) and responder analysis is <i>at Week 12</i> . Target subject population: Clarified to include subjects |
| otbelises | ≥4 years of age, where approved, ≥18 years of age for all other countries. |
| At Must M | Clarified ages for adult (≥18 years of age) and adolescent subjects (aged 12-17 years, where approved). |
| 3 | Added Subjects will be recommended not to take more than 8 puffs of Ventolin per day and advised to contact the investigator if their symptoms necessitate more than 8 puffs of Ventolin in a day. |
| | Addition of initial assumptions for calculations of sample size and information about the blinded sample size-re- |

| Section Section | Changes to Protocol Amendment 2 (Version 3.0) |
|---|---|
| | estimation. Re-estimation was performed once 44% of subjects had completed Week 12. |
| | Updated to describe and justify a second blinded same size re-estimation once approximately 65% of the revised sample size completes 12 weeks of the study and before the last subject is randomized. |
| | Modified the cap in sample size to 1300, and specified this is a 30% increase above the revised number of 1600 subjects as opposed to the previously calculated cap of 800, a 33% increase above the planned number of 600 |
| | subjects. |
| 1 Introduction | 1.1 Background |
| | Added Albuterol is approved its many countries as salbutamol in multiple formulations for the treatment or prevention of bronchoconstriction. |
| | 1.3 Benefit/risk and ethical assessment |
| | Added justification to continue study enrollment and treatment during the COVID-19 pandemic. |
| | 2.4 Sprdy design |
| n di | Added recommendation to not exceed 8 puffs of Ventolin per day. |
| agort any mar | Figure 1: Updated to reflect new sample size estimates. |
| 2 Study Objectives SUPY | 2.4 Exploratory objectives |
| 2 Study Objectives support | Specified that the change from baseline in the Asthma Control Questionaire-5 (ACQ-5) and responder analysis is at Week 12 |
| 3 Subject selection, enrollment, | 3.1 Inclusion criteria |
| randomization, restrictions, | y Inclusion criteria 2 updated to add <i>In the Czech Republic</i> , |
| termination | Germany, Serbia, Slovakia, and Ukraine only subjects ≥18 years will be included. |
| | Inclusion criteria 5 updated the predicted normal value of pre-bronchodilator FEV <sub>1</sub> for subjects age 4-7 to $\geq 50\%$ (from $\geq 50$ to $< 90\%$ ) and to add Subjects 4 to 17 years of age who previously failed inclusion criteria 5 due to the |

# Section **Changes to Protocol Amendment 2 (Version 3.0)** upper $FEV_1$ limit will be permitted to re-screen once and will be required to meet all eligibility criteria upon rescreening. Inclusion criteria 7 updated: Subjects 4 to 11 years will be eligible if they provide 2 acceptable / repeatable measurements. Inclusion criteria 15 revised to define the practice of complete abstinence, to remove *highly* when describing methods of effective birth control methods, and modified to clarify appropriate methods of double-barrier birth control. The definition of menopausal women was updated to remove the reference to $\geq 50$ years of age. Inclusion criteria 16 modified to emove the word *highly* when referring to effective methods of double-barrier contraception. 3.2 Exclusion Priter Exclusion eritema 4 updated to include dupilumab Chisio Ocriteria 24 updated to include Currently **(égnyint or** breastfeeding. This document must not be used to support any many Exclusion criteria 28 updated to previously been randomized from enrolled and to add For pediatrics, see inclusion criterion 4. 3.3 Subject enrollment and randomization Updated the number of adult and adolescent subjects randomized from 600 to 1000, the number of subjects within each treatment arm from 120 to 200, and the number of subjects screened from 1000 to 2000. Updated the estimated screen failure rate from 40% to 50%. 3.7 Methods for unblinding Clarified methods for unblinding and specified that decisions will be based on the investigator's clinical judgement. The requirement that the investigator should discuss with the Sponsor medical monitor or other appropriate personnel, when possible, was removed.

| Section Section | Changes to Protocol Amendment 2 (Version 3.0) |
|---|---|
| | 3.9 Treatment discontinuation by subject and/or |
| | Sponsor |
| | The following reason for IP discontinuation was added: <i>In</i> |
| | subjects who have elevated liver enzymes AST and/or |
| | $ALT \ge 3$ times the upper limit of normal (×ULN) and |
| | total bilirubin ≥2×ULN (ie, meeting the criteria of at |
| | least potential Hy's Law), IP will be suspended until the |
| | liver test values return to the normal range. If the ST, |
| | ALT, or total bilirubin reach these elevated levels again, |
| | after recommencement of IP, the subject will be |
| | discontinued from IP and withdrawn from the study. |
| | 3.11 Screen failures |
| | The following exception for screen failures was added: |
| | Subjects who are screen failures will not be re-screened |
| | with the exception of children and adolescents who |
| | screen-failed because they did not meet the now obsolete |
| | 40 |
| | who previously fasted to meet the upper FEV1 % |
| | predicted threshold, but who met all other eligibility |
| | requirements, may re-screen once. Upon re-screening, |
| | upper FEV1 % predicted limit. Children and adolescents who previously faced to meet the upper FEV1 % predicted threshold, but who met all other eligibility requirements, may re-screen once. Upon re-screening, these subjects must meet all eligibility requirements in order to be randomized. Table 1: Added pregnancy testing to Visits 3 and 5, added Ventolin administration (recorded in MasterScope) to Screening, and removed IP administration (recorded in MasterScope) at Screening. Footnote h: Updated from Visits 2 and 4 to all other visits for pregnancy testing. Footnote i: updated upper threshold values for FEV₁ to ≥50% from ≥50-<90% in subjects aged 4-17 years. 4.2 Randomization/treatment period Added urine pregnancy testing at Visits 3 and 5 in the Czech Republic and at the safety follow up visit in Argentina. Clarified that serum pregnancy tests are required at Visit 6 or the premature discontinuation visit (PDV). |
| Section 4 Study plan and timing of | Table 1: Added <i>pregnancy testing</i> to Visits 3 and 5, |
| procedures | added Ventolin administration (recorded in |
| na | MasterScope) to Screening, and removed IP |
| 31 | administration (recorded in MasterScope) at Screening. |
| A MILL | <b>Footnote h:</b> Updated from <i>Visits 2 and 4</i> to <i>all other visits</i> |
| 2001 | for pregnancy testing. |
| ent, | <b>Footnote i:</b> updated upper threshold values for FEV <sub>1</sub> to |
| (10) | $\geq$ 50% from $\geq$ 50-<90% in subjects aged 4-17 years. |
| ZEO | |
| e No | 4.2 Randomization/treatment period |
| 200 | A 11 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
| X NV | Added urine pregnancy testing at Visits 3 and 5 in the |
| aus | Czech Republic and at the safety follow up visit in |
| KL' | Argentina. Clarified that serum pregnancy tests are |
| | required at Visit 6 <i>or the premature discontinuation visit</i> (PDV). |
| 5 Study Assessments | Administrative changes |
| | 5.1.1.1 Reversibility test |
| | Clarified that pre-dose PFTs are to be done after <i>at least</i> |
| 1 | 15 minutes of rest and before administration of Ventolin. |

| Section | Changes to Protocol Amendment 2 (Version 3.0) |
|---|---|
| | 5.1.1.2 COVID-19 and Pulmonary Function Testing |
| | New section added to specify that spirometry should not be done if subjects are showing signs and symptoms of |
| | COVID-19 and to indicate that participants with suspected COVID-19 should receive a test to confirm diagnosis. |
| | COVID-19 and to indicate that participants with suspected COVID-19 should receive a test to confirm diagnosis. 5.1.2 Asthma Control Questionnaire-5 |
| | Sentence revised to Linguistically validated translations of |
| | the ACQ-5 into local languages will be used (removed with results transcribed into the eCRF). |
| | 5.1.3 Asthma Control Questionnaire-7 |
| | Sentence revised to Linguistically validated translations of the ACQ-7 into local languages will be used (removed |
| | with results transcribed into the eCRF). |
| | 5.1.6.1 Peak expiratory flow |
| | with results transcribed into the eCRF). 5.1.6.1 Peak expiritory flow Modified to record 3 PEF measures from the best of at least 3. 5.1.6.3 eDiary Ventolin therapy use |
| | 5.1.6.3 eDiary Ventolin therapy use |
| a any ma | Added recommendation that subjects should not take more than 8 puffs of Ventolin per day and to contact the investigator if more than 8 puffs are needed. |
| SUPPOT | 5.1.8.5 Treatment for severe asthma exacerbations |
| At must not be used to support any man | Clarified that treatment for less than 3 days doesn't constitute a severe asthma exacerbation except if the subject is hospitalized due to asthma. |
| nust not | Table 4 Laboratory safety variables |
| rt n' | Updated urine pregnancy test timing, added PDV to list of abbreviations, and added a reference to section 3.9. |
| 6 Safety reporting and medical management | 6.3.7 Hy's Law |
| management | Updated that occurrences of AST and/or $ALT \ge 3 \times ULN$ combined with $TBL \ge 2 \times ULN$ may require $IP$ |
| | suspension/discontinuation and study withdrawal and |

| <u>Section</u> | Changes to Protocol Amendment 2 (Version 3.0) |
|---|---|
| | may need to be reported as SAEs. A reference to section 3.9 was also added. |
| | 6.3.8 COVID-19 adverse events |
| | Added to provide instructions on how to handle AEs related to the COVID-19 pandemic. |
| 7 Investigational product and other treatments | 7.2 Dose treatment regimens Updated that subjects should not take more than 8 puffs |
| | Updated that subjects should not take more than a puffs of Ventolin per day. 7.5 Compliance |
| | Updated that Ventolin usage will be monitored during the study. |
| | 7.8.1 Investigational product and Ventolin therapies |
| | Added Subjects on maintenance allergy immunotherapy (AIT) are allowed to continue their AIT; the new initiation of APT during the study is not allowed. |
| | 7.8.3 Promibited medications |
| ) | Starified the use of oral, parenteral, or rectal corticosteroids to include (except if required to treat |
| * any me | asthma exacerbation). |
| Support | Added Montelukast, for any indication |
| int must not be used to support any main | <b>Dupilumab</b> was added to the list of prohibited monoclonal or polyclonal antibodies and the use of <b>intra-ocular</b> monoclonal or polyclonal antibody therapy was clarified to be allowed. |
| | Clarified the use of beta2-adrenergic blockers including eye-drops specific cardio-selective beta-blockers in low daily doses, eg, metoprolol in doses up to 100 mg/d, are allowed. |
| 8 Statistical analysis | 8.2 Sample size estimate |

| <b>Section</b> | Changes to Protocol Amendment 2 (Version 3.0) |
|---|---|
| | Added Section 8.2.1 to describe the initial assumptions for |
| | sample size estimates and <b>Section 8.2.2</b> to describe the |
| | process for blinded sample size re-estimation. This re- |
| | estimation resulted in updates to the number of adult and |
| | adolescent subjects randomized from 600 to 1000, the |
| | number of subjects within each treatment arm from 120 to |
| | 200, and the number of subjects screened from 1000 to |
| | <b>2000</b> . The screen failure rate was updated from 40% to |
| | 50%. The potential increase in sample size cap was |
| | increased from 800 to 1300. |
| | Described processes for a second blinded sample size re- |
| | estimation. |
| | idi |
| | 8.5.1.1 Dual-primary efficacy endpoints |
| | Specified that baseline FEV will be taken as the average |
| | of the 60- and 30-minute gre-dose spirometry measures at |
| | randomization and notion or before randomization. |
| | 8.5.2.2 Derivation of Asthma Control Questionnaire-7 |
| | 8.5.2.2 Derivation of Asthma Control Questionnaire-7 variables Added an exploratory endpoint for the 3 factor endpoint |
| | Added are exploratory endpoint for the 3 factor endpoint |
| | koategootzation (Improved, No change, Worsening) from |
| | haseline to Week 12 |
| 3 | |
| Inal | 8.5.3.4 Derivation of peak expiratory flow |
| , 2003 | The best of at least 5 PEF measurements was updated to at |
| aport | least 3 PEF measurements. |
| nt must not be used to support any man | 8.6.1 Analysis of the dual-primary variable |
| is section of the sec | Clarified that primary comparisons <i>will exclude the</i> |
| , e ), e | children (ages 4-11 years) and specified that the analysis |
| -0.0 | will be repeated to include children, but will be |
| A CO | considered a supportive analysis of the dual-primary |
| A MILES | endpoint. |
| <b>3</b> ) | Added supportive analysis of participants randomized |
| | according to actual strata they were allocated to. |
| | 8.6.4.5 Asthma Control Questionnaire-5 variables |
| | Added exploratory analysis of the 3-factor categorization endpoint for ACQ-7. |

| Section Section | Changes to Protocol Amendment 2 (Version 3.0) |
|---|---|
| | 8.6.7.3 COVID-19 pandemic impacts |
| | Added to describe statistical methods that will be used to evaluate the impact of the COVID-19 pandemic on efficacy and safety variables. |
| 12 List of References | Added reference to the American Academy of Allergy Asthma and Immunology for information regarding COVID-19 and Asthma. |
| Appendix E, Hy's Law | Indicated when subjects with elevated liver enzymes will be suspended from or discontinued from IP. |
| | Updated definitions of potential Hy's Law and Hy's Law. |
| Appendix L, COVID-19 emergency | Added processes to ensure subject safety during the |
| measures permitted to ensure | COVID-19 pandemic. Instructions for management of |
| subject safety | subjects with or suspected COMD-19 infection, delayed |
| | visits, remote visits, subject discontinuation, shipment of |
| | study drug to subjects, laboratory testing, and spirometry |
| | testing are provided. |

# 11.2 Changes to protocol amenament 1 (Version 2.0)

| Section | Changes to Protocol Amendment 1 (Version 2.0) |
|---|---|
| Clinical Study Protocol Synopsis | Administrative change. |
| What | Clarification provided on the target subject population. |
| gupport ari. | Changes to Protocol Amendment 1 (Version 2.0) Administrative change. Clarification provided on the target subject population. Clarification on Sponsor-provided IP dose frequency (QID). |
| 4.0 Study plan and timing of procedures use | Administrative changes. |
| procedures | Table 1: Addition of and adjustments to |
| OTTO | table/footnote(s) to confirm that new IP will be |
| Jet! | dispensed and used for FEV <sub>1</sub> measurements and that at |
| in the state of th | Visit 6 and PDV, IP will be dispensed for the purposes |
| | of completing FEV <sub>1</sub> measurements but will not be taken home by the subjects. |
| | Table 2: Table title updated to Timed assessments at |
| | Visit 2 through Visit 6 and Premature Discontinuation |
| | Visit. |

| | Adjustments to the table to clarify drug dispensing and dose timing. |
|---|---|
| | 4.2 Randomization/treatment period |
| | Clarification and instructions regarding proper IP preparation, dispensing, and dosing for post-dose assessments (ie, new IP in relation to FEV <sub>1</sub> ) at each interest clinic dosing visit. |
| | Addition of new recommendation for opening the seal around the study day treatment box. |
| | around the study day treatment box. 4.3 Treatment discontinuation |
| | Addition of dispensation of IP (for spirometry only) and dosing to procedures carried out during PDV visit. |
| 5.0 Study assessments | 5.1.1 Lung function measurement by spirometry |
| At must not be used to support any man | Administrative changes including clarification that IP should be dosed before 10:00 AM in all in-clinic dosing visite. S1.1.1 Reversibility test Clarification that pre- and post-dose FEV <sub>1</sub> measurements are in relation to Sponsor-provided bronchodilator (Ventolin). |
| SUPPORT | 5.1.6 eDiary |
| 30,40,50 | Administrative changes. |
| , pe use | 5.2.3 Vital signs measurements |
| at must not | Removal of <i>supine</i> as position for measuring blood pressure. |
| | 7.8 Concomitant medications and other treatments |
| other treatments | Addition of <i>medications</i> to the title. |
| | 7.8.1 Investigational product and Ventolin therapies |
| L | |

| Clarification on Sponsor-provided IP dose frequency (dosed QID). | |
|---|---|
| 7.8.3 Prohibited medications | Ä |
| Correction of naming for cytochrome P <b>450</b> 3A4 inhibitors. | an application |

# 12

- LIST OF REFERENCES

  1. American Academy of Allergy Asthma and Immunology (AAAAI). QOVID-19 and Asthma: What Patients Need to Know. 04 Jun 2020. Accessed 19 Jun 2020. https://www.aaaai.org/conditions-and-treatments/library/asthmachbrary/

  2. Bond Avillion 2 Development LP, 2018 Immunology (AAAAI). QOVID-19 and Asthmachbrary/

  2. Bond Avillion 2 Development LP, 2018 Immunology (AAAAI). QOVID-19 and Asthmachbrary/

  2. Bond Avillion 2 Development LP, 2018 Immunology (AAAAI). QOVID-19 and Asthmachbrary/

  3. Bond Avillion 2 Development LP, 2018 Immunology (AAAAI). QOVID-19 and Asthmachbrary/

  3. Bond Avillion 2 Development Avillion 2 Development Avillion 2 Development Avillion 2 Development Avillion 2 Develo Inhalation Suspension (BD MDI, PT008); Alburerol Sulfate Pressurized Inhalation Suspension (AS MDI, PT007).
- 3. Cooper PR, Panettieri RA. Steroids completely reverse albuterol-induced β2-adrenergic receptor tolerance in human small airways J Allergy Clin Immunol. 2008;122(4):734-740.
- 4. Corren J. Summary information for chaled corticosteroid and long-acting β2-adrenergic agonist combination product use in patients in the united states who have asthma or chronic obstructive pulmonary disease Clin Ther. 2007;29:823-843.
- 5. Global Initiative for Asthona. Global strategy for asthma management and prevention. 2018. Available from: http://winasthma.org/2018-gina-report-global-strategy-for- asthmamanagement-and-wevention/.
- 6. Juniper EF, Quyatt GH, Willan A, Griffith LE. Determining a minimal important change in a disease specific quality of life questionnaire. J Clin Epidemiol. 1994;47(1):81-87.
- 7. Junioer EF, Svensson K, Mörk AC, Ståhl E. Measurement properties and interpretation of Free shortened versions of the asthma control questionnaire. Respir Med. 2005;99(5):553-558.
- 8. Kerwin E, Barnes N, Gibbs M, et al. Fluticasone furoate/vilanterol once daily improves night-time awakenings in asthma patients with night symptoms; post-hoc analyses of three randomized controlled trials. J Asthma. 2017; Epub ahead of print. DOI: 10.1080/02770903.2017.1362429.
- 9. Kavuru M, Melamed J, Gross G, Laforce C, House K, Prillaman B, et al. Salmeterol and fluticasone propionate combined in a new powder inhalation device for the treatment of  95 of 142

- asthma: a randomized, double-blind, placebo-controlled trial. J Allergy Clin Immunol. 2000;105(6 Pt 1):1108-1116.
- 10. Mendes ES, Horvath G, Campos M, Wanner A. Rapid corticosteroid effect on
- 11. Mendes ES, Cadet L, Arana J, Wanner A. Acute effect of an inhaled glucocorticosteroid goch albuterol-induced bronchodilation in patients with moderately severe asthma. Chest. 2015;147(4):1037-1042. 12. Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, et al. Standardisation of spirometry. Eur Respir J. 2005;26(2):319-338.
- budesonide and formoterol in one pressurised metered-dose inhales h adults and adolescents with moderate to severe asthma. Drugs. 2006;66:2263-2254.
- 14. O'Byrne PM, Bisgaard H, Godard PP, Pistolesi M, Palmqyist M, Zhu Y, et al. Budesonide/formoterol combination therapy as both maintenance and reliever medication in asthma. Am J Respir Crit Care Med. 2005
- 15. O'Byrne PM. Acute asthma intervention: resignes from the STAY study. J Allergy Clin Immunol. 2007;119(6):1332-1336.
- 16. Rabe KF, Atienza T, Magyar P, Karsson P, Jorup C, Lalloo UG. Effect of budesonide in combination with formoterol for reliever therapy in asthma exacerbations: a randomized controlled, double-blind study, Eancet. 2006;368(9537):744-753.
- 17. Tattersfield AE, Postma S, Barnes PJ, Svensson K, Bauer CA, O'Byrne PM, et al. Exacerbations of asthma: a descriptive study of 425 severe exacerbations. The FACET International Study Group. Am J Respir Crit Care Med. 1999;160(2):594-599.

This document must not be used to

The daduled that the lead to support on the land to th

# APPENDIX B, PRIMARY INVESTIGATOR SIGNATURE PAGE

| I agree to conduct the study in accordance with the co | urrent protocol. |
|---|---|
| Principal Investigator's Name (print) | — of such ap |
| Principal Investigator's Signature | Date of et |
| Principal Investigator's Name (print) Principal Investigator's Signature Please keep the signed original form in your study files a monitor. COPT and the standard and the st | and return a copy to your local study |
| et not be used to support any man | |

# APPENDIX C, GLOBAL INITIATIVE FOR ASTHMA (GINA, 2018)

The table below is not a table of equivalence, but of estimated clinical comparability. Coses may be country-specific application. Some seems of the country see Categories of low, medium, and high doses are based on published information and available doses are arbitrary, but for most ICSs are those that, with prolonged use, are associated with increased risk of systemic side effects.

Subjects enrolling in this study may be taking low-dose ICS, the below table shows GINA guidance in relation to low-dose ICS in relation to inclusion criterion 4.

Low, Medium, and High Doses of Inhaled Corticosteroids

| Adults and a | dolescents (12 years an | ıd older) | |
|---|---|---|---|
| 000000000000000000000000000000000000000 | Daily desage (μg) | | |
| DRUG | <u> </u> | | HIGH |
| Beclometasone dipropionate (CFC) <sup>a</sup> | 300-508 | >500-1000 | >1000 |
| Beclometasone dipropionate (HFA) | C 100-200 | >200-400 | >400 |
| Budesonide (DPI) | 200-400 | >400-800 | >800 |
| Ciclesonide (HFA) | 80-160 | >160-320 | >320 |
| Beclometasone dipropionate (CFC) <sup>a</sup> Beclometasone dipropionate (HFA) Budesonide (DPI) Ciclesonide (HFA) Fluticasone furoate (DPI) Fluticasone propionate (HFA) Mometasone furoate Triamcinolone Retonide | 100 | NA | 200 |
| Fluticasone propionate (DPI) | 100-250 | >250-500 | >500 |
| Fluticasone propionate (HFA) | 100-250 | >250-500 | >500 |
| Mometasone furcate | 110-220 | >220-440 | >440 |
| Triamcinolone Retonide | 400-1000 | >1000-2000 | >2000 |
| , <sup>1</sup> / <sub>2</sub> ( | Children 6-11 years | | |
| Beclometasorie dipropionate (CFC) <sup>a</sup> | 100-200 | >200-400 | >400 |
| Beclova tasone dipropionate (HFA) | 50-100 | >100-200 | >200 |
| Budesonide (DPI) Budesonide (nebules) Ciclesonide | 100-200 | >200-400 | >400 |
| Budesonide (nebules) | 250-500 | >500-1000 | >1000 |
| Ciclesonide | 80 | >80-160 | >160 |
| Fluticasone furoate (DPI) | NA | NA | NA |
| Fluticasone propionate (DPI) | 100-200 | >200-400 | >400 |
| Fluticasone propionate (HFA) | 100-200 | >200-500 | >500 |
| Mometasone furoate | 110 | ≥220 <b>-</b> <440 | ≥440 |

| Triamcinolone acetonide | 400-800 | >800-1200 | >1200 |
|-------------------------|---------|-----------|-------|
|-------------------------|---------|-----------|-------|

# Low Daily Doses of Inhaled Corticosteroids for Children 5 Years and Younger

| Low Daily Doses of Inhaled Corticost | teroids for Children 5 Years and Younger |
|---|---|
| DRUG | Low daily dosage (µg) (age group with adequate safety and effective data) |
| Beclometasone dipropionate (HFA) | 100 (ages ≥5 years) |
| Budesonide nebulized | 500 (ages ≥1 year) o |
| Fluticasone propionate (HFA) | 100 (ages ≥4 years) |
| Mometasone furoate | 110 (ages ≥ wears) |
| Budesonide pMDI + spacer | Not sufficiently stanted in this age group |
| Ciclesonide | Not sufficiently studied in this age group |
| Triamcinolone acetonide | Not sufficiently studied in this age group |
| Abbreviations: HFA=hydrofluoroalkane propel | o authorn |

Beclometasone dipropionate CFC is included for comparison with other literature.

# APPENDIX D, ADDITIONAL SAFETY INFORMATION

# Further guidance on the definition of a serious adverse event

# Life-threatening

'Life-threatening' means that the subject was at immediate risk of death from the AE as it occurred or it is suspected that use or continued use of the product would result in the subject's death. 'Life-threatening' does not mean that an AE occurred in a more severe form it might have caused death (eg, hepatitis that resolved without hepatic failure).

Hospitalization

Outpatient treatment in an emergency room is not in itself an SAE, although the reasons for it may be (eg, bronchospasm, laryngeal edema). Hospital admissions and/or surgical operations planned before or during a study are not considered AEs if the illness or disease existed before the subject was enrolled in the study, provided that it did not deteriorate in an unexpected way during the study.

Important medical event or medical intervention

Medical and scientific judgement of situations and Medical and scientific judgement should be exercised in deciding whether a case is serious in situations where important medical containing on the immediately life-threatening or result in death, hospitalization, disability, or incopacity, but may jeopardize the subject or may require medical intervention to prevent 1 or more outcomes listed in the definition of serious. These should usually be considered as crious.

Simply stopping the suspect drug does not mean that it is an important medical event; medical judgement must be used Examples of important medical events include but are not limited to:

- Angioedema not severe enough to require intubation but requiring intravenous hydrocortisone treatment.
- Heatotoxicity caused by paracetamol (acetaminophen) overdose requiring treatment With N-acetylcysteine.

Intensive treatment in an emergency room or at-home for allergic bronchospasm.

- Blood dyscrasias (eg, neutropenia or anemia requiring blood transfusion, etc.) or convulsions that do not result in hospitalization.
- Development of drug dependency or drug abuse.

# A guide to interpreting the causality question

When making an assessment of causality, consider the following factors when deciding if there is a 'reasonable possibility' that an AE may have been caused by the drug:

- Time Course. Exposure to suspect drug. Has the subject actually received the suspect drug? Did the AE occur in a reasonable temporal relationship to the administration of the suspect drug?
- Consistency with known drug profile. Was the AE consistent with the previous knowledge of the suspect drug (pharmacology and toxicology) or drugs of the same pharmacological class? Or could the AE be anticipated from its pharmacological properties?
- De-challenge experience. Did the AE resolve or improve on stopping or reducing the dose of the suspect drug?
- No alternative cause. The AE cannot be reasonably explained by another cause such as the underlying disease, other drugs, and other host or environmental factors.
- Re-challenge experience. Did the AE reoccurrif the suspected drug was reintroduced after having been stopped? The Sponsor wouldn't normally recommend or support a re-challenge.
- Laboratory tests. A specific laboratory investigation (if performed) has confirmed the relationship.

In difficult cases, other factors could be considered such as:

- Is this a recognized feature of overdose of the drug?
- Is there a known mechanism?

Causality of 'reated' is made if after a review of the relevant data there is evidence for a 'reasonable possibility' of a causal relationship for the individual case. The expression 'reasonable possibility' of a causal relationship is meant to convey, in general, that there are facts (evidence) or arguments to suggest a causal relationship.

The causality assessment is performed on the basis of the available data, including enough information to make an informed judgement. With limited or insufficient information in the case, it is likely that the event(s) will be assessed as 'not related'.

Causal relationship in cases where the disease under study has deteriorated because of lack of effect should be classified as no reasonable possibility.


# APPENDIX E, HY'S LAW

# Introduction

This Appendix describes the process to be followed to identify and appropriately report cases of Hy's Law. It is not intended to be a comprehensive guide to the management of elevated liver biochemistries.

During the course of the study, the investigator will remain vigilant for increases in liver biochemistry. In subjects who have elevated liver enzymes AST and/or ALT ≥ 3×ULN and total bilirubin  $\geq 2 \times ULN$ , IP will be suspended until the liver test values return to the normal range. If the AST, ALT, or total bilirubin reach these elevated levels again, after recommencement of IP, the subject will be discontinued from IP and withdraws from the study. The investigator is responsible for determining whether a subject meets potential Hy's Law criteria at any point during the study.

The investigator participates, with the Sponsor's clinical project representatives, in review and assessment of cases meeting potential Hy's Law (PHL) criteria agree whether Hy's Law (HL) criteria are met. Hy's Law criteria are met if there is no alternative explanation for the elevations in liver biochemistry other than drug induced Wer injury caused by the IP.

The investigator is responsible for recording data pertaining to potential HL/HL cases and for reporting AEs and SAEs according to the outcome of the review and assessment in line with standard safety reporting processes.

Definitions

Potential Hy's Law

Aspartate aminotransferase and or alanine transaminase ≥3× ULN combined with TBL

≥2×ULN at any point during the study after the start of IP irrespective of an increase in alkaline phosphatase.

# Hy's Law

AST and/or  $\overrightarrow{AST} \ge 3 \times ULN$  combined with TBL  $\ge 2 \times ULN$ , where no other reason, other than the IP, can be found to explain the combination of increases, eg, elevated alkaline phosphatase

This documental HL and HL, the elevation in transaminases must precede or be coincident with the elevations in transaminases and TBL must occur.

Identification of potential Hv's Law 27

To identify cases of PHL it is important to perform a comprehensive review of laboratory data for any subject who meets any of the following identification criteria in isolation or in combination:

- ALT ≥3×ULN
- AST >3×ULN
- TBL >2×ULN

When a subject meets any of the identification criteria, in isolation or in combination, the central laboratory will immediately send an alert to the investigator and the medical monitor assigned to the project.

The investigator will also remain vigilant for any local laboratory reports where the identification criteria are met; where this is the case, the investigator will:

- Notify the medical monitor assigned to the project.
- Request a repeat of the test (new blood draw) by the central laboratory.
- Contact the medical monitor to discuss the elevated local laboratory values and whether these constitute an AE. Where an AE is entered due to elevations of local laboratory values, the AE will be queried in the eCRF and elevated local laboratory values, units and ranges will be entered to the query response.
- When the identification criteria are met from central or local laboratory results, the investigator will without delay:
  - Determine whether the subject meets PHL criteria by reviewing laboratory reports from all previous visits (including both central and local laboratory results).
- The investigator will, without delay, review each new laboratory report and if the identification criteria are met, will:
  - Notify the medical monitor assigned to the project.
  - Determine whether the subject meets PHL criteria by reviewing laboratory reports from all previous visits.
  - Promptly enter the laboratory data into the laboratory eCRF.

# Follow-up

# Potential Hy's Law criteria not met

If the subject does not meet PHL criteria the investigator will:

Inform the medical monitor assigned to the project that the subject has not met PHL criteria.

Perform follow-up on subsequent laboratory results according to the guidance provided in the Clinical Study Protocol.

# Potential Hy's Law criteria met

If the subject does meet PHL criteria, the investigator will:

Determine whether PHL criteria were met at any study visit before starting IP (Actions required when potential Hy's Law criteria are met before and after starting IP)

Notify the medical monitor assigned to the project who will then inform the central study team

The medical monitor assigned to the project will discuss the issue with the investigator to provide guidance and agree an approach for the study subjects' follow-up and the continuous review of data. Subsequent to this contact the investigator will:

Monitor the subject until liver biochemistry parameters and appropriate clinical symptoms and signs return to normal or baseline levels, or as long as medically indicated

Investigate the cause of the event and perform diagnostic investigations as discussed with the medical monitor assigned to the project. For studies using a central laboratory add: This includes deciding which the tests available in the HL laboratory kit should be used.

Complete the 3 Liver eCRF modules as information becomes available

If at any time (in consultation with the medical monitor assigned to the project) the PHL case meets serious criteria, report it as an SAE using standard reporting procedures.

# Review and assessment of potential Hy's Law cases

No later than 3 weeks after the biochemistry abnormality was initially detected, the medical monitor assigned to the project contacts the investigator to review available data and agree on whether there is an alternative explanation for meeting PHL criteria other than drug induced liver injury caused by the IP. The medical monitor assigned to the project and global safety physician will also be involved in this review with other subject matter experts, as appropriate.

According to the outcome of the review and assessment, the investigator will follow the instructions below.

If there is an agreed alternative explanation for the ALT or AST and TBL elevations, a determination of whether the alternative explanation is an AE will be made and subsequently whether the AE meets the criteria for an SAE:

If the alternative explanation is **not** an AE, record the alternative explanation on the appropriate eCRF

If the alternative explanation is an AE/SAE, record the AE/SAE in the eCRF accordingly and follow the Sponsor's standard processes

If it is agreed that there is **no** explanation that would explain the ALT or AST and TBL elevations other than the IP:

Report an SAE (report term 'Hy's Law') according to the Sponsor's standard processes.

- The 'Medically Important' serious criterion should be used if no other serious criteria apply.
- As there is no alternative explanation for the HL case, a causality assessment of 'related' should be assigned.

If, there is an unavoidable delay, of over 3 weeks, in obtaining the information necessary to assess whether or not the case meets the criteria for HL, then it is assumed that there is no alternative explanation until such time as an informed decision can be made:

Report an SAE (report term 'potential Hy's Law') applying serious criteria and causality assessment as per above

Continue follow-up and review according to agreed plan. Once the necessary supplementary information is obtained, repeat the review and assessment to determine whether HL criteria are met. Update the SAE report according to the outcome of the review amending the reported term if an alternative explanation for the liver biochemistry elevations is determined.

# Actions required when potential Hy's Law criteria are met before and after starting IP

This section is applicable to subjects who meet PHL criteria on study treatment having previously met PHL criteria at a study visit before starting IP.

At the first on study treatment occurrence of PHL criteria being met the investigator will:

Determine if there has been a significant change in the subjects' condition compared with the last visit where PHL criteria were met

- If there is no significant change no action is required.
- If there is a significant change, notify the Sponsor representative, who will inform the central study team, then follow the subsequent process described in Potential Hy's Law criteria met of this Appendix.

A 'significant' change in the subject's condition refers to a clinically relevant change in any of the individual liver biochemistry parameters (ALT, AST, or TBL) in isolation or in combination, or a clinically relevant change in associated symptoms. The determination of whether there has been a significant change will be at the discretion of the investigator; this may be in consultation with the medical monitor assigned to the project if there is any uncertainty.

# Actions required for repeat episodes of potential Hy's Law

This section is applicable when a subject meets PHL criteria on study treatment and has already met PHL criteria at a previous on study treatment visit.

The requirement to conduct follow-up, review, and assessment of a repeat occurrence(s) of PHL is based on the nature of the alternative cause identified for the previous occurrence.

The investigator should determine the cause for the previous occurrence of PHL criteria being met and answer the following question:

Was the alternative cause for the previous occurrence of PHL criteria being met found to be the disease under study or did the subject meet PHL criteria before starting study treatment and at their first on study treatment visit as described in Actions required when potential Hy's Law criteria are met before and after starting IP.

If No: follow the process described in Potential Hy's Law criteria met of this Appendix.

If Yes:

Determine if there has been a significant change in the subject's condition compared with when PHL criteria were previously met

If there is no significant change, no action is required

If there is a significant change:

A 'significant' change in the subject's condition refers to a clinically relevant change in any of the individual liver biochemistry parameters (ALT, AST, or TBL) in isolation or in combination, or a clinically relevant change in associated symptoms. The determination of whether there has been a significant change will be at the discretion of the investigator; this may be in consultation with the medical monitor assigned to the project if there is any uncertainty.
# APPENDIX K, SPIROMETRY ASSESSMENT CRITERIA

## **Acceptable Versus Usable Tests**

## Acceptable Tests must meet the following Criteria:

- 1. Acceptable start of exhalation with brisk upstroke, no hesitation or false start, and back extrapolation volume <5% of forced vital capacity (FVC) or 0.150 L, whichever is the greater (see example in Figure 1)
- 2. No cough during the first second
- 3. No valsalva maneuver
- 4. No leak
- 5. No obstruction of mouthpiece
- 6. No extra breaths
- 7. Plateau achieved: ie, the volume-time curve shows no change in volume (<0.025 L) for ≥1 second, and the subject has tried to exhale for at least 6 seconds

An acceptable test meets all 7 criteria listed. This is to be considered the "gold standard".

Usable spirometry tracings are those that only meet criteria 1 and 2. When this occurs, repeat testing up to 8 attempts for pre-dose and 5 attempts for post-dose assessments, in an effort to obtain 3 acceptable spirograms. If only usable tests are obtained, report results based on the 3 best usable trials with observed limitations.

Figure 1 Example of a Usable Spirogram



EV=back extrapolation volume

The expanded version of the early part of a subject's volume-time spirogram, illustrating back extrapolation through the steepest part of the curve, where flow is PEF rate, to determine the new "time zero". Forced vital capacity -4.291 L; EV - 0.123 L (2.9% FVC): back extrapolation line through peak expiratory flow.

# **Between-Maneuver Reproducibility Criteria**

#### **Pre-dose Assessments**

After 3 acceptable spirograms have been obtained, apply the following tests:

- The 2 largest values of FVC must be within 0.150 L of each other
- The 2 largest values of FEV<sub>1</sub> must be within 0.150 L of each other

If these criteria are met, the spirometry testing for that time point may conclude, however, if possible, please continue collecting additional spirograms to a maximum of 8 pre-dose and 5 post-dose attempts. The highest FEV<sub>1</sub> and the highest FVC obtained at each testing time point (even if from different reproducible tracings), will be collected.

If acceptability criteria are not met, continue testing until they are met, or the subject cannot/should not continue (maximum of 8 attempts).

#### **Post-dose Assessments**

- After 2 acceptable spirograms have been obtained, apply the following tests:
- The 2 largest values of FVC are within 0.150 L of each other and/or
- The 2 largest values of FEV<sub>1</sub> are within 0.150 L of each other

If these criteria are met, the spirometry testing for that time point may conclude. The highest  $FEV_1$  and the highest FVC obtained at each testing time point (even if from different reproducible tracings), will be collected.

If acceptability/reproducibility criteria are not met, continue testing until they are met, or the subject cannot/ should not continue (maximum of 5 attempts).

# APPENDIX L, COVID-19 EMERGENCY MEASURES PERMITTED TO ENSURE SUBJECT SAFETY

The following activities were implemented in order to ensure subject safety during the global lockdown due to the COVID-19 pandemic. While global lockdown restrictions are currently being released, the pandemic continues and in certain territories cases remain on the rise. Therefore, necessary emergency measures accepted during the initial global lockdown will be permitted to protect subject safety in the event that infection rates return to levels requiring the return of government or local restrictions on movement of people and goods.

Any procedure performed outside the protocol specified requirements will be documented as a protocol deviation.

### **Visit Management:**

# **Delayed Visits**

- Out of window visits should be considered if it is necessary to safeguard the health of the subject and site staff or enables an on-site subject visit.
- If a return to lockdown is announced or the site is on lockdown and cannot process a visit, if possible, visits should be rescheduled to earlier/later as required to safeguard subjects and site staff.
- Randomization: If a subject is in screening and cannot complete the randomisation visit within 28 days due to local COVID-19 lockdown restrictions, the screening period may be extended to a maximum of 9 weeks. In the event of an extension to the screening period >28 days due to COVID, the following safety measurements should be repeated in advance of randomisation: safety laboratory assessments, ECG, vital signs, concomitant medications, and medical/surgical history.
- Visit 6/Week 24: All efforts should be made to complete the associated assessments in the clinic, even if this is visit is delayed. If necessary, while waiting for the time to complete this visit, an unscheduled call and drug dispensing should be done to ensure the subject has sufficient IP during this time.

| Remote Visits | • | Where subjects have COVID-19 infection or infectious, the site is on lock down, local restrictions prohibit attendance, or similar, a telephone visit should be completed. All assessments performed should be documented in the same way they would if the visit would have happened on-site. Before performance of a remote visit, verbal consent must be |
|---|---|---|
| | | obtained and documented in the subject's medical notes to ensure that the subject understands the implications of continuing in the study when face to face visits are temporarily not possible due to COVID 19 restrictions. Where possible, the Principal Investigator should ask the subject to confirm their agreement in writing either by email or via a letter. Where multiple in-clinic visits will be missed, written consent of the subject will be required. |
| | • | If a remote visit is completed and it is considered appropriate<br>and safe to continue study drug, this could be dispatched direct<br>to the subject by courier. |
| | • | Randomization visits cannot be conducted remotely and therefore subjects in screening who do not wish to attend an on-site visit should be screen-failed as 'withdrawal of consent'. |
| Subject<br>Discontinuation | • | Where repeated visits are likely to be missed, the site should discuss with the subject and consider ongoing treatment options. Where a subject does not wish to attend further clinic visits, a PDV visit should be scheduled. |
| Shipment of Drug<br>from Site to Subjects | • | Subjects should provide verbal consent via a telephone call to use their personal details to complete the site to subject shipment request. Consent must be documented in the subject medical records and preferably confirmed in writing via an email or other written means (eg, via post) via a phone call initially and followed up by written consent at the earliest possibility. |
| Safety Labs | • | Where central analysis is not possible, local testing is permitted. Lab normal ranges would need to be made available. |

| | • In the event that routine safety lab tests are missed due to temporary inability of subject to get to site due to COVID-19, an unscheduled lab should be done at their next clinic visit if possible. |
|---|---|
| Spirometry | • The investigator should request confirmation from the subjects to confirm that they are not aware of having been exposed to COVID-19 that they are not currently infected or infectious, and should exercise their medical judgement with respect to this information prior to conducting spirometry assessments. Sites should continue to follow hygiene and cleaning guidance within the manuals to minimize possible cross-contamination. |
| Subjects with Confirmed COVID- 19 Infection | <ul> <li>If a subject has confirmed COVID-19 this is to be reported as an AE/SAE, but is not per se a reason to withdraw the subject.</li> <li>The investigator should determine whether the subject's IP should continue, be interrupted, or stopped in accordance with the Clinical Study Protocol.</li> <li>The investigator should continue to reassess the benefit-risk of continued study involvement for a study subject infected with COVID-19. In-clinic visits for this subject should only recommence once the infection has resolved and the subject is no longer considered to be infectious.</li> <li>For new subjects previously identified as COVID-19 positive, a re-test must be performed after resolution of symptoms (if present). The subject can only be considered for enrollment 4 weeks after having a negative result.</li> </ul> |